# STATISTICAL ANALYSIS PLAN AMENDMENT 3

Study: MG0003

**Product: Rozanolixizumab** 

A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY EVALUATING EFFICACY AND SAFETY OF ROZANOLIXIZUMAB IN ADULT PATIENTS WITH GENERALIZED MYASTHENIA GRAVIS

SAP/Amendment Number
Final SAP
SAP Amendment 1
SAP Amendment 2
SAP Amendment 2
SAP Amendment 3 This document cannot a phication a sphication a sphicatio 10 November 2021

#### **Confidentiality Statement**

#### Confidential

This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.


# **TABLE OF CONTENTS**

| LIST OF A | BBREVIATIONS | 7 |
|---|---|---|
| 1 INTR | ODUCTION | 11 |
| 2 PROT | OCOL SUMMARY | 11 |
| 2.1 Stu | dy objectives | 11 |
| 2.1.1 | Primary objective | 11 |
| 2.1.2 | Secondary objective | 11 |
| 2.1.3 | Other objectives | 11 |
| 2.2 Stu | dy endpoints | 11 |
| 2.2.1 | dy endpoints Efficacy endpoints 1 Primary efficacy endpoint 2 Secondary efficacy endpoints 3 Other efficacy endpoints Pharmacokinetic/pharmacodynamic endpoints 1 Pharmacokinetic endpoint 2 Pharmacodynamic endpoints Safety endpoints 1 Secondary safety endpoints 2 Other safety endpoints Anti-drug antibody endpoints Immunological endpoints Other and exploratory endpoints dy design and conduct | 11 |
| 2.2.1 | .1 Primary efficacy endpoint | 11 |
| 2.2.1 | .2 Secondary efficacy endpoints | 12 |
| 2.2.1 | .3 Other efficacy endpoints | 12 |
| 2.2.2 | Pharmacokinetic/pharmacodynamic endpoints | 13 |
| 2.2.2 | .1 Pharmacokinetic endpoint | 13 |
| 2.2.2 | .2 Pharmacodynamic endpoints | 13 |
| 2.2.3 | Safety endpoints | 13 |
| 2.2.3 | .1 Secondary safety endpoints | 13 |
| 2.2.3 | .2 Other safety endpoints | 13 |
| 2.2.4 | Anti-drug antibody endpoints | 14 |
| 2.2.5 | Immunological endpoints | 14 |
| 2.2.6 | Other and exploratory endpoints | 14 |
| 2.3 Stu | dy design and conduct | 14 |
| | ermination of sample size | |
| | A ANALYSIS CONSIDERATIONS | |
| | neral presentation of summaries and analyses | |
| 3.2 Ger | neral study level definitions | |
| 3.2.1 | | |
| 3.2.1 | | |
| 3.2.2 | Study periods | 20 |
| 3.2.3 | Mapping of assessments performed at Premature End of Treatment Visit | 20 |
| 3.2.2<br>3.2.3<br>3.3 Def | inition of Baseline values | 21 |
| 3.4 Pro | tocol deviations | 21 |
| 3.5 Ana | alysis sets | 21 |
| 3.5.1 | Enrolled Set | 21 |
| 3.5.2 | Randomized Set | |
| 3.5.3 | Safety Set | 21 |
| 3 5 4 | Pharmacokinetic Per-Protocol Set | 21 |

| 3.5 | 5.5 Full Analysis Set | .21 |
|-----|-----------------------------------------------------|------|
| 3.6 | Treatment assignment and treatment groups | .22 |
| 3.7 | Center pooling strategy | .22 |
| 3.8 | Coding dictionaries | .22 |
| 3.9 | Changes to protocol-defined analyses | .22 |
| 4 5 | STATISTICAL/ANALYTICAL ISSUES | .23 |
| 4.1 | Adjustments for covariates | .23 |
| 4.2 | | .24 |
| 4.2 | | . 24 |
| 4.2 | Dates and times. Missing data due to COVID-19. | .25 |
| 4.2 | 2.3 Missing data due to COVID-19 | .26 |
| 4.3 | Handling of repeated and unscheduled measurements | .27 |
| 4.4 | Interim analyses and data monitoring | .27 |
| 4.4 | | .27 |
| | 4401 D. (10 11 1) | 20 |
| | 4.4.2.2 Data required for Interim analysis | . 29 |
| 4.5 | 171GILLOUILUI DUGGIOD | |
| 4.6 | Multiple comparisons/multiplicity | .30 |
| 4.7 | Use of an efficacy subset of study participants | |
| 4.8 | Active-control studies intended to show equivalence | .32 |
| 4.9 | Examination of subgroups | .32 |
| 4.9 | | |
| 4.9 | | |
| 4.9 | | |
| 5 5 | STUDY POPULATION CHARACTERISTICS | .33 |
| 5.1 | Participant disposition. | .33 |
| 5.2 | Protocol deviations | .34 |
| 6 I | DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS | .34 |
| 6.1 | Demographics | |
| 6.2 | Other Baseline characteristics | |
| 6.3 | Medical history and concomitant diseases | .36 |
| 6.4 | Prior and concomitant medications | |
| 6.4 | | |
| 6.4 | 8 | |
| 6.4 | | |
| | MEASUREMENTS OF TREATMENT COMPLIANCE | |
| 8 I | EFFICACY ANALYSES | |
| 8.1 | Handling of intercurrent events | .38 |

| 8.2 | St | Statistical analysis of the primary efficacy endpoint | 39 |
|---|---|---|---|
| 8.2 | 2.1 | Derivation of primary efficacy endpoint | 43 |
| 8.2 | 2.2 | Primary analysis of the primary efficacy endpoint | 43 |
| 8.2 | 2.3 | Sensitivity analyses of the primary efficacy endpoint | 45 |
| | 8.2 | 2.3.1 Sensitivity Analysis #1 | 45 |
| | 8.2 | 2.3.2 Sensitivity Analysis #2 | 45 |
| | 8.2 | 2.3.3 Sensitivity Analysis #3 | |
| | 8.2 | 2.3.4 Sensitivity Analysis #4 | 46 |
| 8.2 | 2.4 | Supplementary analyses of the primary efficacy endpoint | 46 |
| | 8.2 | 2.4.1 Supplementary Analysis #1 | |
| | 8.2 | 2.4.2 Supplementary Analysis #2 | 47 |
| 8.2 | 2.5 | Additional Analysis | 47 |
| 8.2 | 2.6 | 2.4.1 Supplementary Analysis #1 2.4.2 Supplementary Analysis #2 Additional Analysis Exploratory Analysis Statistical analysis of the secondary efficacy endpoints MG-ADL Responder Rate at Visit 10 (Day 43) | 47 |
| 8.3 | St | statistical analysis of the secondary efficacy endpoints | 47 |
| 8.3 | 3.1 | MG-ADL Responder Rate at Visit 10 (Day 43) | 52 |
| 8.3 | 3.2 | Change from Baseline to Day 43 (Visit 10) in MG-C score | 52 |
| 8.3 | 3.3 | Change from Baseline to Day 43 (Visit 10) in QMC score | 53 |
| 8.3 | 3.4 | Change from Baseline in PRO Muscle Weakness Fatigability score | |
| 8.3 | 3.5 | Change from Baseline in PRO Physical Fatigue score | 53 |
| 8.3 | 3.6 | Change from Baseline in PRO Bulbar Symptoms score | 54 |
| 8.4 | A | Analysis of other efficacy endpoints | |
| 8.4 | 4.1 | Use of rescue therapy due to worsening (IVIg, PEX) | 54 |
| 8.4 | 4.2 | Time to first rescue therapy | 54 |
| 8.4 | 4.3 | Time to MG-ADI response ( $\geq$ 2.0 points improvement from Baseline) | 55 |
| 8.4 | 4.4 | QMG score | 55 |
| 8.4 | 4.5 | QMG responder rate (≥3.0 points improvement from Baseline) | |
| 8.4 | 4.6 | MG-C score | |
| 8.4 | 4.7 | MGC responder rate (≥3.0 points improvement from Baseline) | |
| 8.4 | 4.8 | MG-ADL score | |
| | 4.9 | MG-ADL responder rate (≥2.0 points improvement from Baseline) | |
| - ( | 4.10 | | |
| | 4.11 | | |
| 8.4 | 4.12 | MG Symptoms PRO 'Bulbar Symptoms' | 58 |
| 8.4 | 4.13 | Patient Global Impressions of Severity | 58 |
| 8.4 | 4.14 | | |
| 8.4 | 4.15 | MGII overall scores, ocular sub-scores, and generalized domain score | s58 |
| 8.4 | 4.16 | | |
| 8.4 | 4.17 | ' EQ-5D-5L | 58 |

| 8.4.18 | 8 Minimal symptom expression | 59 |
|---|---|---|
| 9 PH | ARMACOKINETICS AND PHARMACODYNAMICS | 59 |
| 9.1 I | Pharmacokinetics | 59 |
| 9.2 I | Pharmacodynamics | 60 |
| 9.2.1 | MG-specific autoantibodies | 60 |
| 9.2.2 | Total serum IgG and IgG subclasses | .,61 |
| 9.3 | Anti-drug antibody status | 61 |
| 9.3.1 | ADA Data Consideration | 62 |
| 9.3.2 | ADA summaries | 64 |
| 9.4 I | mmunology | 66 |
| 9.4.1 | | 66 |
| 9.4.2 | Serum cytokines | 66 |
| 9.4.3 | Serum immunoglobulin concentrations | 66 |
| 9.4.4 | Anti-tetanus toxoid serum titers | 67 |
| 10 SA | FETY ANALYSES | 67 |
| 10.1 I | Extent of exposure | |
| 10.2 A | Adverse events | |
| 10.2.1 | Data considerations | |
| 10.2.2 | 2 AE summaries | 69 |
| 10.2.3 | Adverse Events of Focus | 70 |
| 10.2.4 | | 71 |
| 10.3 | Clinical laboratory evaluations. | |
| 10.3.1 | | |
| 10.4 V | Vital signs, physical findings, and other observations related to safety | |
| 10.4.1 | | 74 |
| 10.4.2 | 2 Electrocardiograms. | 74 |
| 10.4.3 | | |
| | 0.4.3.1 Physical examination | |
| | 0.4.3.2 Suicidal risk monitoring | |
| | Assessment and management of Tuberculosis (TB) | |
| | HER ANALYSES | |
| | Specific analyses for Pharmaceuticals and Medical Devices Agency (PMDA) | |
| 1 | Headache questionnaire | |
| 12 RE | FERENCES | 79 |
| 13 AP | PENDICES | 80 |
| 13.1 | QMG Scale | 80 |
| 13.2 N | MG-C score | 81 |
| 13.3 N | MG-Activities of Daily Living | . 82 |

#### LIST OF ABBREVIATIONS

**AChR** Acetylcholine Receptor **ADA** Anti-Drug Antibody

AE Adverse Event

**AEOF** Adverse Event of Focus

arkeiing authorization athereof. **AESI** Adverse Event of Special Interest **AESM** Adverse Event of Special Monitoring

**ALP** Alkaline Phosphatase

**ALQ** Above the Limit of Quantification

**ALT** Alanine Aminotransferase **ANCOVA** Analysis of Covariance

**AST** Aspartate Aminotransferase

**ATC** Anatomical Therapeutic Chemica

Below the Limit of Quantification BLO

**BMI Body Mass Index** BP **Blood Pressure** 

**BUN** Blood Urea Nitrogen Change from Baseline CfB CI Confidence Interval **CRF** Case Report Form

**CSR** Clinical Study Report

C-SSRS Columbia Suicide Severity Rating Scale

**CTCAE** Common Terminology Criteria for Adverse Events

CVCoefficient of Variation **DEM Data Evaluation Meeting** 

**ECG** Electrocardiogram

Estimated Glomerular Filtration Rate

EQ Visual Analogue Scale

EQ-5D-5L Euro-Quality of Life 5-Dimensions, 5 Levels

ES **Enrolled Set** 

**FAS** Full Analysis Set

**FDA** Food and Drug Administration Geometric Coefficient of Variation geoCV

Geometric Mean geoMean

| | GGT | Gamma Glutamyltransferase |
|---|---|---|
| | HbA1c | Glycosylated Hemoglobin |
| | hCG | Human Chorionic Gonadotropin |
| | HLGT | High Level Group Term |
| | HLT | High Level Term |
| | IA | Interim Analysis |
| | ICH | International Council for Harmonisation |
| | IDMC | Independent Data Monitoring Committee |
| | ICE | Intercurrent Event |
| | Ig | Immunoglobulin |
| | IgA | Immunoglobulin A |
| | IgE | Immunoglobulin E |
| | IgG | Immunoglobulin G |
| | IgM | Immunoglobulin M |
| | IMP | High Level Group Term High Level Term Interim Analysis International Council for Harmonisation Independent Data Monitoring Committee Intercurrent Event Immunoglobulin Immunoglobulin A Immunoglobulin G Immunoglobulin M Investigational Medicinal Product |
| | INR | International Normalized Ratio |
| | IPD | Important Protocol Deviation |
| | IVIg | Intravenous Immunoglobulin G |
| | IWRS | Interactive Web Response System |
| | LDH | Lactate Dehydrogenase |
| | LLOQ | Lower Limit of Quantification |
| | LLT | Lower Level Term |
| | LSMD | Least Squares Mean Difference |
| | MA MAR MedDRA MG MG-ADL MG-C | Markedly Abnormal |
| | MAR | Missing at Random |
| | MedDRA | Medical Dictionary for Regulatory Activities |
| | MG | Myasthenia Gravis |
| | MG-ADL | Myasthenia Gravis -Activities of Daily Living |
| 8 | MG-C | Myasthenia Gravis- Composite |
| | MGFA | Myasthenia Gravis Foundation of America |
| | MGII | Myasthenia Gravis Impairment Index |
| | MG-QOL15r | Myasthenia Gravis MG Quality of Life 15 Item Scale<br>Revised |
| | MI | Multiple Imputation |
| | MMRM | Mixed Model for Repeated Measures |

| MNAR | Missing not at Random |
|---|---|
| MSE | Minimum Symptom Expression |
| MSR | Minimum Significant Ratio |
| MuSK | Muscle Specific Kinase |
| n | Number of Participants |
| NAb | Neutralizing Antibody |
| NRI | Nonresponse Imputation |
| OLE | Open-Label Extension |
| PD | Pharmacodynamic |
| pDILI | Potential Drug Induced Liver Injury |
| PEOT | Number of Participants Neutralizing Antibody Nonresponse Imputation Open-Label Extension Pharmacodynamic Potential Drug Induced Liver Injury Premature End of Treatment Plasma Exchange Patient Global Impressions of Change |
| PEX | Plasma Exchange |
| PGI-C | Patient Global Impressions of Change |
| PGI-S | Patient Global Impressions of Severity |
| PK | Pharmacokinetic |
| PK-PPS | Pharmacokinetic Per-Protocol Set |
| PLS | Population-Level Summary |
| PMDA | Pharmaceuticals and Medical Devices Agency |
| PRO | Patient-Reported Outcome |
| PT | Preferred Term |
| PTT | Partial Thromboplastin Time |
| QMG | Quantitative Myasthenia Gravis |
| RBC | Red Blood Cell Count |
| RLZ | Rozanolixizumab |
| RBC RLZ RPACT RS SAP SC SD SGOT | R Package for Adaptive Clinical Trials |
| RS | Randomized Set |
| SAP | Statistical Analysis Plan |
| sc | Subcutaneous |
| SD O | Standard Deviation |
| SGOT | Serum Glutamic-Oxaloacetic Transaminase |
| SGPT | Serum Glutamic-Pyruvic Transaminase |
| SMQ | Standardised MedDRA Query |
| SOC | System Organ Class |
| SS | Safety Set |


#### 1 INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to provide all information that is necessary to perform the statistical analyses of study MG0003, including interim and final analyses. It also defines the summary tables, figures and listings (TFLs) to be included in the final Clinical Study Report (CSR) according to the protocol.

This SAP is based upon, and assumes familiarity with, the following documents:

- Protocol Amendment 4: 23 February 2021
- IDMC Charter: 19 January 2021

If a future protocol amendment necessitates a substantial change to the statistical analysis of the study data, this SAP may be amended accordingly. Changes to the analysis from the protocol are documented in Section 3.9. The content of this SAP is compatible with the International Council for Harmonisation (ICH)/Food and Drug Administration (FDA) E9 Guidance documents.

#### 2 PROTOCOL SUMMARY

# 2.1 Study objectives

#### 2.1.1 Primary objective

To demonstrate the clinical efficacy of rozanolixizumab in patients with generalized myasthenia gravis (MG).

# 2.1.2 Secondary objective

To assess safety and tolerability of rozanolixizumab in MG patients.

#### 2.1.3 Other objectives

- To assess pharmacokinetic (PK) characteristics of rozanolixizumab
- To assess the pharmacodynamics (PD) effects of rozanolixizumab on IgG, disease-specific autoantibodies
- To evaluate the emergence and incidence of anti-drug antibody (ADA) and impact on PK and PD
- To evaluate the effects of rozanolixizumab on the concentration of total protein, IgM, IgA, and IgE, serum and plasma complement levels and serum cytokines
- To assess the effect of rozanolixizumab on tetanus IgG antibodies
- To assess the effect of rozanolixizumab on exploratory biomarkers and protein expression, and explore the relationship between protein, and metabolite biomarkers and cause, progression, and appropriate treatment of MG

#### 2.2 Study endpoints

# 2.2.1 Efficacy endpoints

# 2.2.1.1 Primary efficacy endpoint

• Change from Baseline to Day 43 (Visit 10) in MG-activities of daily living (ADL) score

## 2.2.1.2 Secondary efficacy endpoints

- MG-ADL responder (≥2.0 points improvement from Baseline) at Day 43 (Visit 10)
- Change from Baseline to Day 43 (Visit 10) in MG-Composite (MG-C) score
- Change from Baseline to Day 43 (Visit 10) in quantitative myasthenia gravis (QMG) score
- Change from Baseline to Day 43 (Visit 10) in the MG Symptoms patient-reported outcome (PRO) 'Muscle Weakness Fatigability' score
- Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Physical Fatigue' score
- Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Bulbar Symptoms' score

# 2.2.1.3 Other efficacy endpoints

- Use of rescue therapy due to worsening (IVIg, PEX)
- Time to first rescue therapy
- Time to MG-ADL response (≥2.0 points improvement from Baseline)
- Change from Baseline in QMG at each scheduled assessment during Treatment and Observation Periods
- QMG responder (≥3.0 points improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in MG-C score at each scheduled assessment during Treatment and Observation Periods
- MG-C responder (≥3.0 points improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
- MG-ADL responder (≥2.0 points improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in the MG Symptoms PRO 'Muscle Weakness Fatigability' score at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in the MG Symptoms PRO 'Physical Fatigue' score at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in the MG Symptoms PRO 'Bulbar Symptoms' score at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in the MG Symptoms PRO 'Respiratory Symptoms' score at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in the MG Symptoms PRO 'Ocular Symptoms' score at each scheduled assessment during Treatment and Observation Periods
- Patient Global Impressions of Severity (PGI-S) at each scheduled assessment during the Treatment and Observation Periods

- Patient Global Impressions of Change (PGI-C) at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in MG-ADL (excluding ocular items) at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in QMG (excluding ocular items) at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline in MG-C score (excluding ocular items) at each scheduled assessment during Treatment and Observation Periods
- Change from Baseline to Day 43 in MG Quality of Life 15 Item scale revised (MG-QOL15r)
- Change from Baseline to Day 43 in Euro-Quality of Life 5-Dimensions, 5 levels (EQ-5D-5L)
- Minimal Symptom Expression (MG-ADL score of 0 or 1) at any time up to and including Day 43 (Visit 10)
- Change from Baseline in MG Impairment Index (MGII) scores at each scheduled assessment during Treatment Period
- Change from Baseline in MGII ocular sub-scores at each scheduled assessment during Treatment Period
- Change from Baseline in MGII generalized domain sub-scores at each scheduled assessment during Treatment Period

# 2.2.2 Pharmacokinetic/pharmacodynamic endpoints

#### 2.2.2.1 Pharmacokinetic endpoint

• Plasma concentration of rozanolixizumab at each scheduled assessment during the Treatment and Observation Periods.

# 2.2.2.2 Pharmacodynamic endpoints

- Change (absolute and percentage) from Baseline in MG-specific autoantibodies at each scheduled assessment during the Treatment and Observation Periods
- Change (absolute and percentage) from Baseline in serum total IgG and IgG subclasses concentrations at each scheduled assessment during the Treatment and Observation Periods

# 2.2.3 Safety endpoints

# 2.2.3.1 Secondary safety endpoints

- Occurrence of treatment-emergent adverse events (TEAEs)
- TEAEs leading to withdrawal of investigational medicinal product (IMP)

# 2.2.3.2 Other safety endpoints

- Occurrence of adverse events of special monitoring (AESM)
- Vital sign changes from Baseline (systolic and diastolic blood pressure (BP) and pulse rate at each scheduled assessment during the Treatment and Observation Periods)

- 12-lead electrocardiogram (ECG) change from Baseline at each scheduled assessment during the Treatment and Observation Periods
- Laboratory change from Baseline at each scheduled assessment during the Treatment and Observation Periods (hematology, clinical chemistry, and urinalysis)
- Suicidality as measured by the Columbia Suicide Severity Rating Scale (C-SSRS)

#### 2.2.4 Anti-drug antibody endpoints

ADA status at each scheduled assessment during the Treatment and Observation Periods

#### 2.2.5 Immunological endpoints

- Change from Baseline in serum complement levels (C3 and C4) and plasma complement levels (C3a and C5a) at each scheduled assessment during the Treatment and Observation Periods
- Change from Baseline in serum cytokines at each scheduled assessment during the Treatment Period
- Change from Baseline in serum immunoglobulin concentrations (total IgA, IgE, and IgM) at each scheduled assessment during the Treatment and Observation Periods
- Change from Baseline in anti-tetanus toxoid serum fiters at each scheduled assessment during Treatment and Observation Period

#### 2.2.6 Other and exploratory endpoints

- Exploratory biomarkers may be measured to evaluate the effect of rozanolixizumab
- Proteins, and metabolites changes that may be measured to understand the cause, progression, and appropriate treatment of MG

A specific SAP will be written to describe the analysis methods for those endpoints, as the results will not be summarized in the CSR. The nature and format of these analyses will be detailed in this SAP.

# 2.3 Study design and conduct

This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, 3-arm, repeat dose study evaluating the efficacy and safety of two doses of rozanolixizumab and matching placebo in patients with generalized MG who experience moderate to severe symptoms (Myasthenia Gravis Foundation of America [MGFA II-IVa]) and are being considered for additional treatment such as IVIg or PEX.

Fixed unit doses across body weight tiers and study arms will be employed:

Treatment Arm 1 (rozanolixizumab) – equivalent to approximately

- Bodyweight <50kg: dose to be administered
- Bodyweight ≥50kg and <70kg: dose to be administered
- Bodyweight ≥70kg and <100kg: dose to be administered
- Bodyweight ≥100kg; dose to be administered

Treatment Arm 2 (rozanolixizumab) – equivalent to approximately

- Bodyweight <50kg: dose to be administered
- Bodyweight ≥50kg and <70kg: dose to be administered
- Bodyweight ≥70kg and <100kg: dose to be administered
- Bodyweight ≥100kg; dose to be administered

The placebo arm will be 0.9% sodium chloride aqueous solution (physiological saline, preservative free) for subcutaneous (sc) administration.

Approximately up to 388 study participants will be screened at about 135 sites from North America, Europe and Asia to achieve the minimum targeted number of 150 to a maximum of 240 evaluable study participants.

Participants have the opportunity to rollover into an open-label extension (OLE) study, as described below. The OLE study, MG0004 (chronic treatment) will be replaced by MG0007, which consists of chronic treatment based on MG worsening. Upon study site approval of MG0007, as well as fulfilment of regulatory requirements, study participants will have the opportunity to rollover directly into MG0007. In the event a study participant has already started MG0004, a minimum treatment duration of 6 visits (if IMP treatment is held for low IgG, study participants missed dose(s) can be counted as part of the total 6 visits for completion of MG0004 and meet eligibility requirements for MG0007) must be completed prior to moving into MG0007. Once the site is active for MG0007, no further participants will enroll in MG0004 and the study will be closed at the site once all eligible study participants have discontinued MG0004 and had the opportunity to rollover into MG0007.

The maximum duration of MG0003 study per study participants will be up to 18 weeks, consisting of a Screening Period (1 to 28 days to account for central laboratory turn-around time), a Treatment Period (6 weeks), and a blinded Observation Period (8 weeks).

- 1. All study participants who complete the 6-week Treatment Period may roll over into an 8-week Observation Period.
- 2. All eligible study participants who complete the Observation Period will be invited to be rerandomized into an OLE study to either active dose arm 1 or 2.
- 3. Study participants who experience disease worsening during the 6-week Treatment Period (e.g., an increase of 2 points on the MG-ADL or 3 points on the QMG scale between two consecutive visits) may be considered for rescue therapy (IVIg or PEX) at the discretion of the Investigator.
- 4. Study participants who need rescue therapy during the 6-week Treatment Period will receive IVIg or PEX and complete any subsequent visit(s). No further infusions of rozanolixizumab will be administered after initiation of rescue therapy. Once the participant completes Visit 10, he or she will move into the 8-week Observation Period.
- 5. Study participants who complete the Treatment Period and require initiation of rescue therapy after they start the 8-week Observation Period, may either opt to receive IVIg or PEX or complete the EOS visit and immediately roll over into an OLE study where the participant

- will receive rozanolixizumab. Participants who opt to receive IVIg or PEX will complete any remaining visits in the Observation Period and will not be invited to join an OLE study.
- 6. Study participants who did not complete the 6-week Treatment Period because they needed rescue therapy and require initiation of a second course of rescue therapy while in the 8-week Observation Period can roll over to an OLE study if a minimum of 2 weeks have lapsed since completion of the last IVIg or PEX session. The EOS visit must be completed before enrolling into an OLE study. Alternatively, they can be treated with IVIg or PEX. Study participants who opt to receive IVIg or PEX will complete any remaining visits in the Observation Period and will not be invited to join an OLE study.
- 7. Study participants who discontinue study medication for any reason other than requiring rescue therapy will not be eligible for enrollment into an OLE study.

A schematic diagram of the study is provided in Figure 2-1.

**FIGURE 2-1: STUDY SCHEMATIC** 



IVIg=intravenous immunoglobulin G; PEX=plasma exchange; Rozimab=rozanolixizumab

## 2.4 Determination of sample size

As detailed in Section 4.4, this study will consist of 2 stages, with a formal interim analysis at the end of Stage 1.

Based on historical data, the mean difference in adjusted changes from Baseline of MG-ADL at Day 43, between rozanolixizumab and placebo, is assumed to be 1.5 to 2.0 and the standard deviation is assumed to be 3.5 to 4. A difference of >1.5 could be judged to be clinically meaningful.

It is proposed that the interim analysis will be conducted when approximately 90 eligible study participants have been treated and are evaluable for the primary endpoint, i.e., approximately 30 study participants per dose group in Stage 1. If the study is not stopped for futility after Stage 1, the sample size will be increased, subject to a maximum cap, to provide an overall conditional power target of 90% based on the observed effect size in Stage 1. For each dose that is not futile, the comparison-wise conditional power will be calculated which is the probability of, given the observed data, to achieve a significant result for the completed trial if only the considered treatment is selected. If two doses are selected, then the conditional power associated with the higher treatment effect will be used to determine the stage 2 sample size. Conditional power will be calculated as described in formula 7.2 of Wassmer and Brannath (2016). Similarly, the stage 2 sample size required to achieve a target conditional power of 90% will be calculated using a formula derived from formula 7.4 of Wassmer and Brannath (2016) as follows:

SD = pooled standard deviation from the stage 1 statistical model using all dose groups TP = target conditional power = 0.9

CRP = Conditional rejection probability at stage 1 for the dose group being considered Delta = assumed true treatment effect for second stage data

If two doses are considered for stage 2 then the above formula will be applied with the conditional error divided by two, to account for multiplicity. Depending upon the selection of one, or two, of the doses after Stage 1, a further 60 to up to a maximum of 150 eligible study participants will be randomized in Stage 2 of the study. Thus, the total sample size of the study could range between 150 and 240 study participants if the study is not futile at Stage 1.

The power of the study using the above adaptive design and expected sample sizes with a sample size cap of 80 per arm and various scenarios of true treatment effect and standard deviation were determined from a stimulation study using the statistical software ADDPLAN MC, the results of which are summarized in Table 2-1.

The simulation results also indicate that across the various scenarios the average sample size for the study ranges between 169 and 203 study participants. The power for scenarios 5 to 7 and 12 to 14, that is, when the high dose has an effect compared to placebo of 2 points, are at least 80%, indicating that the sample size re-assessment process helps maintain reasonable power when only one dose has a clinically meaningful effect of 2 and the data variability is greater than anticipated (standard deviation[SD]=4).

The chances of stopping the study for futility i.e. both doses individually futile, when at least one dose has a clinically meaningful true effect of 2 or more versus placebo, is less than 3%.

These results support the strategy of entering 30 eligible study participants per dose group in Stage 1 and between 30 to 50 study participants per dose group in Stage 2. Note that ADDPLAN MC implements the sample size increase rule 'per arm' rather than 'per stage', so that if only one dose is selected for Stage 2, then the maximum sample size for this stage is 100, whereas if two

doses are selected than the maximum Stage 2 sample size is 150. Therefore, if an overall study sample size cap of 240 (i.e., 150 in Stage 2) were implemented, irrespective of whether one or two doses are selected, then we would expect power for each scenario to be slightly increased compared to those contained in Table 2-1.

Table 2-1: Simulation results from ADDPLAN MC (x100,000 simulations per scenario) with a capped maximum sample size of 80 per arm using a Bonferroni intersection test

| | Treati<br>Effe | | | | | Interim | | Average |
|---|---|---|---|---|---|---|---|---|
| Scenario | Dose 1 | Dose 2 | Standard<br>Deviation | Power | Proportion<br>Futility | Proportion Selecting Low Dose | Proportion Selecting High Dose | Sample Size |
| 1 | 0.0 | 0.0 | | 0.020 | 0.335 | 0.474 | 0.474 | 169.0 |
| 2 | 1.0 | 1.0 | | 0.400 | 0.049 | 0.781 | 0.782 | 203.3 |
| 3 | 1.0 | 1.5 | | 0.632 | 0.023 | 0.657 | 0.914 | 199.1 |
| 4 | 1.5 | 1.5 | 3.5 | 0.750 | 0.011 | 0.838 | 0.841 | 199.8 |
| 5 | 1.0 | 2.0 | | 0.864 | 0.008 | 0.474 | 0.975 | 186.4 |
| 6 | 1.5 | 2.0 | _ | 0.892 | 0.004 | 0.697 | 0.942 | 191.7 |
| 7 | 2.0 | 2.0 | | 0.943 | 0.002 | 0.859 | 0.860 | 189.9 |
| 8 | 0.0 | 0.0 | | 0.020 | 0.335 | 0.467 | 0.463 | 168.1 |
| 9 | 1.0 | 1.0 | | 0.315 | 0.066 | 0.734 | 0733 | 199.9 |
| 10 | 1.0 | 1.5 | 00 | 0.515 | 0.037 | 0.621 | 0.875 | 198.2 |
| 11 | 1.5 | 1.5 | 4.0 | 0.632 | 0.021 | 0.795 | 0.797 | 199.4 |
| 12 | 1.0 | 2.0 | U.S | 0.755 | 0.016 | 0.468 | 0.953 | 189.5 |
| 13 | 1.5 | 2.0 | 20 | 0.792 | 0.010 | 0.663 | 0.912 | 193.7 |
| 14 | 2.0 | 2.0 | 7 2 | 0.871 | 0.005 | 0.823 | 0.822 | 192.3 |

# 3 DATA ANALYSIS CONSIDERATIONS

# 3.1 General presentation of summaries and analyses

Statistical analysis and generation of tables, figures, participant data listings, and statistical output will be performed using SAS® Version 9.3 or higher. All tables and listings will use Courier New font size 9.

Descriptive statistics will be displayed to provide an overview of the study results. For continuous variables, descriptive statistics will include number of participants with available measurements (n), mean, SD, median, minimum, and maximum.

For categorical variables, the number and percentage of participants in each category will be presented. Unless otherwise noted, the denominator for percentages will be based on the number of participants included in the respective analysis set. Participants with missing data can generally be accounted for using the following approaches:

- For summaries of demographics and Baseline characteristics: summarize percentages based on all participants in the analysis set and include a "Missing" category (corresponding to participants with missing data for the variable being summarized) as the last row in the list of categories being summarized.
- For summaries of efficacy and safety variables, unless otherwise specified: summarize percentages based only on those participants with observed data for the variable being summarized. As the denominator may be different from the number of participants in the analysis set being considered, the denominator should be displayed in the table. The general format for displaying this will be "n/Nsub (%)."

Unless otherwise noted, all percentages will be displayed to one decimal place. No percentage will be displayed for zero counts, and no decimal will be presented when the percentage is 100%.

For the purpose of the tabulations the lower and upper confidence limits for the percentages will be truncated at 0 and 100% respectively.

Statistical tests of efficacy variables will be presented as p-values rounded to three decimal places. P-values less than 0.001 will be presented as "<0.001" and p-values greater than 0.999 will be presented as ">0.999". Statistical comparisons will be two-sided and will be performed at the 0.05 level of significance unless specified otherwise. The significance levels used as part of the multiple testing procedure are detailed in Section 4.6.

For PK concentrations, summary statistics will include geometric mean, geometric coefficient of variation (geoCV), 95% confidence intervals (CIs) for geometric mean, arithmetic mean, SD, median, minimum, and maximum. All summaries of PK variables will be based on the observed values. No imputation will be used.

Decimal places for descriptive statistics will always apply the following rules:

- "n" will be an integer;
- Mean, SD, and median will use one additional decimal place compared to the original data;
- CV [%] will be presented with one decimal place;
- Minimum and maximum will have the same number of decimal places as the original value.

If no participants have data at a given time point, for example, then only n=0 will be presented. However, if n<3, present the n, minimum and maximum only. If n=3, n, mean, median, minimum and maximum will be presented only. The other descriptive statistics will be left blank.

Derived variables in general will display the mean, SD and median to 1 more decimal place than the variables used in the derivation. If the number of decimal places reported in the raw data is varied, then use either the maximum raw number of reported decimal places or 3, whichever is the lowest, as a guide for the descriptive statistics.

# 3.2 General study level definitions

### 3.2.1 Analysis time points

All data will be analyzed based on the visits identified per the Schedule of Activities in protocol. Mapping to analysis visit windows is not applied, except for premature end of treatment (PEOT) visits (specified in Section 3.2.3).

#### 3.2.1.1 Relative day

Relative day for an event will be derived with the date of the first sc infusion of IMP as reference.

Relative days for an event of measurement occurring before the date of first sc infusion will be prefixed with '-' and are calculated as follows:

```
Relative Day = [(Event Date - Date of First Infusion)]
```

The relative day for an event or measurement occurring on or after the reference date to the date of the last infusion is calculated as follows:

```
Relative Day = [(Event Date - Date of First Infusion) + 1]
```

For events or measurements occurring after the date of the last sc infusion, relative day will be prefixed with '+' in the data listings and will be calculated as follows:

```
Relative Day = + [(Event Date – Date of Last Infusion)]
```

There is no relative Day 0. Relative day is not calculated for partial dates in cases where relative day is shown in a participant data listing. In such cases, relative day should be presented as '--' in the participant data listings.

### 3.2.2 Study periods

The maximum duration of the study per participant will be approximately 18 weeks, consisting of the following 3 periods:

- Screening Period: 1 to 28 days
- Treatment Period: 6 weeks
- Observation Period: 8 weeks

The end of the study is defined as the date of the last visit of the last participant in the study.

The following definitions for starting and entering the study periods will be applied:

- Treatment Period starts with the first day of IMP and ends after Day 43/PEOT assessments. All participants in the Safety Set will be considered to have started the Treatment Period. A participant is considered to have completed the Treatment Period if assessments from Treatment Period Day 43 are completed.
- Observation Period starts one day after the end of the Treatment Period and ends after the final assessments on the last visit. Participants with assessment on any Observation Period day are considered to have started the Observation Period. Participants who have a completed status in the study termination case report form are considered to have completed the Treatment and Observation Periods.

# 3.2.3 Mapping of assessments performed at Premature End of Treatment Visit

PEOT assessments will be assigned to the next scheduled site visit (following the last scheduled visit that the study participant completed prior to PEOT) where each assessment is evaluated as

per protocol. This approach means that there is a chance that PEOT data will be mapped to different visits according to the schedule of assessments.

#### 3.3 Definition of Baseline values

Baseline will be the last available value prior to or on the same date (and time if time is collected for the individual assessment) of the first infusion of IMP in the Treatment Period, or if missing, the Screening value. Scheduled or unscheduled measurements can be used as the Baseline value. If a Baseline measurement is not available but an unscheduled measurement occurs after the planned baseline measurement time point but before dosing, then the unscheduled measurement will be used. MG-specific autoantibodies MuSK and AChR Baseline is detailed in Section 9.2.1, and ADA Baseline is detailed in Section 9.3.1.

#### 3.4 Protocol deviations

Important protocol deviations (IPDs) are deviations from the protocol which potentially could have a meaningful impact on study conduct or on the primary efficacy, key safety, or PK/PD outcomes (if applicable) for an individual study participant. The criteria for identifying important protocol deviations will be defined within the appropriate protocol-specific document. Important protocol deviations will be reviewed as part of the ongoing data cleaning process and data evaluation. All IPDs will be identified and documented prior to unblinding and will be utilized to decide, which data will exclude study participants from the Pharmacokinetic Per-Protocol Set (PK-PPS).

#### 3.5 Analysis sets

#### 3.5.1 Enrolled Set

The Enrolled Set (ES) will consist of all study participants who have signed the informed consent.

#### 3.5.2 Randomized Set

The Randomized Set (RS) will consist of all study participants who were randomized, using the treatment assigned instead of the actual treatment received.

#### 3.5.3 Safety Set

The Safety Set (SS) will consist of all randomized study participants who received at least one dose of IMP and analyzed according to the actual treatment the participants received.

# 3.5.4 Pharmacokinetic Per-Protocol Set

The PK-PPS will consist of a subset of the SS, consisting of those study participants who received at least 1 dose of rozanolixizumab, had at least 1 quanifiable concentration of rozanolixizumab, and no important protocol deviations affecting the PK variable, as confirmed during a pre-analysis review of the data prior to database lock. Post-Baseline deviations will not necessarily lead to total exclusion of a study participant from the PK-PPS but may lead to exclusion of specific data.

#### 3.5.5 Full Analysis Set

The Full Analysis Set (FAS) will consist of all study participants in the RS, who have a Baseline and least 1 post-Baseline MG-ADL measurement.

# 3.6 Treatment assignment and treatment groups

If after unblinding it is determined that study participants at any time receive incorrect treatment from their randomized assignment, then for safety and PK/PD analyses these study participants will be reallocated to the appropriate treatment group. For example, if study participants randomized to placebo received rozanolixizumab, then for the safety and PK/PD analyses, these study participants will be reallocated to rozanolixizumab. If a study participant received both doses of rozanolixizumab at different time points, then the study participant will be allocated to the higher dose (i.e. group) group in the safety and PK/PD analysis. Study participants randomized to rozanolixizumab will only be reallocated to the placebo treatment group if they never received rozanolixizumab.

Efficacy data will be summarized by randomized treatment group as shown below:

- Placebo
- Rozanolixizumab equivalent, displayed as RLZ
- Rozanolixizumab equivalent, displayed as RLZ

# 3.7 Center pooling strategy

It is planned to recruit study participants in North America, Europe, and Asia in this study, with possible extension to other regions and countries. The data from all sites will be pooled for analyses. Geographic regions and countries are categorized as following,

- Asia (excluding Japan): Taiwan
- Europe: Belgium, Czech Republic, Germany, Denmark, Spain, France, United Kingdom, Georgia, Hungary, Italy, Poland, Russian Federation, Serbia
- North America: Canada, United States
- Japan: Japan

# 3.8 Coding dictionaries

Adverse events (AEs) and medical histories will be coded using version 24.0 or later of the Medical Dictionary for Regulatory Activities (MedDRA®).

Medications will be coded according to B3 version Mar 2021 or later of the World Health Organization Drug Dictionary (WHODD).

# 3.9 Changes to protocol-defined analyses

- Mixed model for repeated measures (MMRM) analysis of covariance (ANCOVA) is specified as the model used for the analysis of primary endpoint. In the SAP, MMRM is used as the model only.
- ADDPLAN MC is specified in the protocol for making determinations from the interim analysis. However, SAS or the R package for Adaptive Clinical Trials (RPACT) will be used instead. For the purposes of this analysis, these packages will provide the same functions as ADDPLAN MC.

- The treatment group by week interaction term is specified to be used in the model of analysis of primary efficacy endpoint. In the SAP, treatment group by day interaction will be used instead.
- The Full Analysis Set (FAS) will consist of all study participants in the RS, who have a baseline and at least one post-Baseline MG-ADL measurement. The protocol incorrectly states this as SS.
- Stratification factors used in statistical modeling, such as muscle specific kinase [MuSK(+/-)] and acetylcholine receptor [AChR(+/-)] are defined in the SAP as two binary variables, instead of one binary variable [MuSK(+) or AChR(+)] this is to account for study participants who may be double-positive.
- Estimands and Intercurrent event handling strategies have been updated based on regulatory feedback.
- Minimal Symptom Expression (MG-ADL score of 0 or 1) at any time up to and include both treatment and observation phase, where the protocol only states to include up to Day 43 (Visit10).
- Potential Hy's Law has been updated to Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 3x Upper Limit of Normal (ULN) and total Bilirubin (TBL) > 2x ULN, and Alkaline Phosphatase (ALP) < 2x ULN.
- Calculation of Low-density lipoprotein (LDL) will follow Friedewald equation, where LDL in mmol/L= TC HDL TRIG/2.22; LDL in mg/dL= LDL=TC-HDL-TRIG/5 (if all values are in mg/dL). This formula is applicable only if Triglycerides is less than or equal to 400 mg/dL (4.52 mmol/L).
- MG-C responders are defined as at least a 3-point improvement (decrease) from Baseline instead of 5-point improvement.
- Patient Global Impressions of Severity (PGI-S) at each scheduled assessment during the Treatment and Observation Periods instead of change from Baseline of PGI-S.

# 4 STATISTICAL/ANALYTICAL ISSUES

# 4.1 Adjustments for covariates

The efficacy analyses will be adjusted for the following covariates:

- Baseline MG-ADL score,
- Region (North America, Europe, and Asia [excluding Japan], Japan),
- Stratification factors MG-specific autoantibodies, including muscle specific kinase [MuSK(+/-)] and acetylcholine receptor [AChR(+/-)], both as binary variables.

In statistical modeling, the stratification factors MuSK(+/-) and AChR(+/-) will be based on the values from MG-specific autoantibody assessment at Baseline. In case Baseline MG-specific autoantibody result is missing (and not resolved after data queries), a post-Baseline measurement may be used. If this is not available, then the historical result will be used in the model; if the historical result is missing as well, the stratification factor from IWRS randomization file will be used to determine values used in the model (i.e., if the stratification is MuSK in IWRS, then

MuSK(+/-) will be imputed as positive, otherwise negative; similarly, if stratification factor is AChR in IWRS, then AChR(+/-) will be imputed as positive, otherwise negative).

# 4.2 Handling of dropouts or missing data

# 4.2.1 Efficacy data

The rules for handling missing data of individual items in the calculation of the QMG, MG-C, MG-ADL, MG Symptom PRO, MGII, and MG-QOL15r scores at a certain visit are described in Section 13.1, Section 13.2, Section 13.3, Section 13.4, Section 13.5 and Section 13.6, respectively.

Imputation methods for missing overall scores (including missing data due to intercurrent events Section 8.1) for the analyses of primary and secondary endpoints are listed as below. The estimand corresponding to these analyses are described in Section 8.

| Efficacy<br>Endpoints | Statistical<br>Analysis Type | Statistical Analysis Methods | Imputation Methods |
|---|---|---|---|
| Primary | Primary | MMRM A AND A | Imputation: maximum likelihood estimation |
| | Sensitivity 1 | MMRM | Imputation: maximum likelihood estimation |
| | Sensitivity 2 | MMRM | Imputation: J2R |
| | Sensitivity 3 | MMRM | Imputation: maximum likelihood estimation |
| | Sensitivity 4 | MMRM | Imputation: maximum likelihood estimation |
| | Supplemental 1 | Trimmed Mean using ANCOVA | Imputation: worst score |
| eni | Supplemental 2 | MMRM | Imputation: maximum likelihood estimation |
| Secondary<br>(continuous) | Secondary | MMRM | Imputation: maximum likelihood estimation |
| O. T. | Sensitivity | MMRM | Imputation: J2R |
| | Supplemental | Trimmed Mean using ANCOVA | Imputation: worst score |
| Secondary<br>(binary) | Secondary | Logistic model | Imputation: NRI |


MMRM=mixed model for repeated measures; ANCOVA= analysis of covariance; J2R=Jump to reference; NRI= nonresponse imputation

For other binary efficacy endpoints (e.g. QMG responder), missing data will be imputed using nonresponse imputation (NRI). That is, study participants with missing data at the timepoint of interest, and all timepoints after use of rescue medication will be treated as non-responders.

For ordinal endpoints (EQ-5D-5L, PGI-S, PGI-C), the observed case method will be applied. No further imputation is used.

#### 4.2.2 Dates and times

Partially or completely missing dates may be imputed for the following reasons:

- Classification of AEs as TEAEs;
- Classification of medications as past, prior, or concomitant medications:
- Durations of AEs;

Imputed dates will not be shown in listings. All dates will be displayed as reported in the database.

The following rules will be applied for partially or completely missing start dates:

- If year, month and day are all missing then assign the date of first dose of IMP. If an imputed start date is after the specified end date, then assign January 01 of the year of the end date, or the date of screening if this is later (if the latter imputation results in an end date that is earlier than the start date, then use January 01).
- If month and day are missing, and year is:
  - the same as the year of the first dose of IMP then assign the month-day of first dose of IMP. If the imputed start date is after the specified end date, then assign January 01, or the month-day of screening date if this is later (if the latter imputation results in an end date that is earlier than the start date, then assign January 01);
  - not the same as the year of the first dose of IMP then assign January 01.
- If only day is missing, and month-year is:
  - the same as the month-year of the first dose of IMP then assign the day of first dose of IMP. If the imputed start date is after the specified end date, then assign first day of the month, or the day of screening date if this is later (if the latter imputation results in an end date that is earlier than the start date, then assign first day of the month);
  - not the same as the month-year of the first dose of IMP then assign the first day of the month.

The following rules will be applied for partial stop dates:

- If only the month and year are specified, then use the last day of the month;
- If only the year is specified, then use December 31 of the known year;
- If the stop date is completely unknown, then use discharge date or data cut-off date.

Note: Discharge date refers to the date of the end of study visit for completed study participants or the date of discontinuation for study participants that were withdrawn. For any AEs with known start date after the date of discontinuation, the date of last contact will be used as the discharge date. For study participants still ongoing in the study at the time of the data cut-off, and for whom no discharge date is available, the date of the data cut-off will be used instead of the discharge date.

Any medication with a start date on the first dosing date and time unknown, will be assumed to be concomitant.

Imputed AE dates will be used for the calculation of duration of AEs as described in Table 4–1

Table 4–1: Calculation rules for duration of AEs

| Data<br>availability | Onset date | Outcome date | Calculation rules |
|---|---|---|---|
| Complete data | D1 | D2 | Duration = D2 - D1 + 1 day |
| Start date partially or completely missing | | D2 | Duration $\leq D2 - D0 + 1$ day<br>Notes: D0 is imputed start date per above rules. |
| End date<br>partially or<br>completely<br>missing | D1 | - PUBLIC | For ongoing AE: Duration ≥ D3 - D1 day For resolved AE: Duration ≤ D3 - D1 day Notes: D3 is imputed end date per above rules. |
| Start and end<br>date partially or<br>completely<br>missing | - annot Y | ing sun | For ongoing AE: Duration $\geq D3 - D0$ day For resolved AE: Duration $\leq D3 - D0$ day Notes: D0 is imputed start date and D3 is imputed end date per above rules. |

# 4.2.3 Missing data due to COVID-19

Missing data is expected to be one of the major implications of the COVID-19 pandemic. The following approaches/strategies will be applied to assess the impact of COVID-19 pandemic in this study.

- Added an eCRF page "COVID-19 Impact", including impacted visits, impact categories and relationship to COVID-19 pandemic.
- Additional fields were added in protocol deviation specification documents to record protocol deviations relationship to COVID-19 pandemic.
- Included additional summary analyses based on the timing of COVID-19 impact (pre/during/post COVID-19 pandemic).

• Additional intercurrent events related to COVID-19 pandemic were included in the estimands for the evaluation of the primary and secondary efficacy endpoints.

#### 4.3 Handling of repeated and unscheduled measurements

All repeated and unscheduled measurements will be presented in the listings, where applicable. The following general rules will apply to all repeated and unscheduled measurements:

- For repeated or unscheduled measurements obtained prior to the first dose of IMP the latest reliable value (scheduled or unscheduled) will be used in the calculation of descriptive statistics (i.e., Screening and/or Baseline);
- For repeated or unscheduled measurements obtained at the designated Baseline visit and prior to the first dose of IMP, the latest reliable value (scheduled or unscheduled) will be defined as the Baseline;
- For repeated or unscheduled measurements obtained at any time point after the first dose of IMP, the scheduled values (if non-missing) will always be used in the calculation of changes from Baseline and for the descriptive statistics (i.e., in summaries by time point). If repeated scheduled values are obtained at any time point, the latest non-missing will be used.

See Section 10.3 for the rules applied to repeated lab results.

See Section 10.4.2 for the rules applied to ECG triplicate measurements.

# 4.4 Interim analyses and data monitoring

# 4.4.1 Timing of and basis for periodic data reviews and interim analysis

An independent Data Monitoring Committee (IDMC) will be formed to monitor the ongoing safety and efficacy of the study.

Approximately 3 periodic data reviews are planned to oversee the safety of the study:

- The first periodic data review will be performed when approximately 15 study participants have completed the 6-week Treatment Period;
- The second periodic data review will be conducted after approximately 60 study participants have completed the 6-week Treatment Period (ad hoc as needed);
- Third review dependent on the outcome of the interim analysis (see details below) will be conducted after approximately 150-180 study participants have completed the 6-week Treatment Period.

The timing of any further data reviews will be decided by the IDMC in conjunction with sponsor. Further details of the IDMC will be provided in an IDMC charter.

In addition to the periodic data reviews mentioned above, a formal interim analysis (IA) is planned for this study at the end of Stage 1, once approximately 90 (see Section 2.4 for sample size details) enrolled study participants (30 per arm) are evaluable for the primary endpoint (having completed up to Day 43). The IA is based on an a 2-stage adaptive design and powered on the primary efficacy endpoint: change from Baseline to Day 43 in MG-ADL.

For the periodic data reviews, all data available at the time of the data cut-off will be included. For the formal interim analysis, only data for the 90 study participants at Stage 1 that have

completed the primary endpoint will be included in the analysis. Listings and descriptive statistics for both the periodic data reviews and the interim analysis may include data beyond the specified cut-off visit for study participants who were enrolled earlier. This will also include data for screen failures.

The database will not be locked for each periodic data review or for the interim analysis. Study enrollment will not be halted during the periodic data reviews or interim analysis. A snapshot of the data will be taken at the required cut-off timepoint.

The data should be as clean as possible for the periodic data reviews and interim analysis, but it is not required to have resolved all queries prior to each database snapshot.

Protocol deviations will be considered for the interim analysis; thus, it will be required to schedule a data evaluation meeting (DEM) prior to the interim analysis. Protocol deviations will not be considered for the periodic data reviews.

At IA, stage 1 data will be presented to and reviewed by the IDMC and the following decisions will be made:

1. Early stopping for futility: if there is no evidence of either dose of rozanolixizumab being effective compared to placebo.

Notes: the non-binding futility stopping rule will require that the nominal Stage 1 p-value of each dose to be greater than 0.5 (1-sided). This corresponds to both estimated treatment effects being in the wrong direction, i.e., inferiority.

2. Move to the next stage:

Before moving to the next stage, the following will be considered:

- 2.1 Dose Selection: If the study is not stopped for futility (not established), then the "best dose" of rozanolixizumab (and the other active dose if the mean response is not worse than 1 point than the selected "best dose") will be selected for Stage 2 of the study.
  - This approach allows selection of the dose with the largest effect defined in terms of the observed mean responses and any doses with a mean response no worse than the best dose by 1 point providing that they are not dropped due to futility, i.e., to be retained nominal 1-sided p-value must be less than 0.5. However, this may not be the sole criterion for selecting the dose, since, additionally, the IDMC will take account other factors, including safety, for the assessment of overall benefit-risk, which will be detailed in the IDMC charter.
- 2.2 Sample size re-estimation: it will be conducted during the IA, as mentioned in Section 2.4.

Note: Early Stopping for Efficacy will not be considered during the IA hence no alpha spending function will be implemented.

#### 4.4.2 Data required for periodic data reviews and interim analyses

The analyses and data required for review are described in this SAP and include all data specified in the IDMC Charter.

#### 4.4.2.1 Data required for periodic data reviews

Required safety and efficacy data to be used to support the periodic data review will include the ne) rate following:

- Adverse events
- **ECGs**
- Vital signs
- Medical and procedure history
- Prior and concomitant medications
- **Demographics**
- Safety labs (hematology, chemistry, urinalysis)
- Total IgG
- Pregnancy
- C-SSRS
- MG-ADL observed results and change from Baseline
- MG-ADL responder (≥2.0 points improvement from Baseline) rates
- MG-C score observed results and change from Baseline
- OMG score observed results and change from Baseline

These data will be summarized using descriptive statistics. Data will also be provided in listings.

#### Data required for interim analysis 4.4.2.2

Descriptive summaries to be used to support the interim analysis for futility will include the following:

- **Demographics**
- Baseline characteristics
- **ECGs**
- Vital signs
- Important PD
- Analysis of MG-ADL change from Baseline at Day 43
- MG-ADL observed results and change from Baseline
- MG-ADL responder (≥2.0 points improvement from Baseline) rates
- MG-C score observed results and change from Baseline
- QMG score observed results and change from Baseline
- Adverse events

- Safety labs (MA values in hematology, chemistry)
- Total IgG

Any changes to this list will be documented in IDMC meeting minutes.

These data will be summarized using descriptive statistics. Data will also be provided in listings: For the futility analysis, dose selection, and sample size re-estimation for Stage 2, a treatment acy endr comparison will be conducted using the primary endpoint (MG-ADL) as described in Section 8.2.2.

#### 4.5 **Multicenter studies**

Individual center results will not be displayed.

#### 4.6 Multiple comparisons/multiplicity

The statistical analysis of the primary efficacy and selected secondary efficacy endpoints will account for multiplicity and control the familywise type I error rate at a 2-sided alpha level of 0.05 by using a parallel gatekeeping testing procedure with a truncated Hochberg test for each of the 6 type I error families (corresponding to the primary endpoint and the five secondary endpoints).

The hypotheses are mapped into 2 sets so that hypotheses within each set correspond to the same rozanolixizumab dose.

Serial restrictions are applied so that the endpoints can only be tested for each dose, if all previous endpoints for that dose are significant.

For family 1, (the primary endpoint hypotheses corresponding to the pairwise comparisons of each dose versus placebo) the Hochberg truncation parameter is set to 0 which is equivalent to using the Bonferroni approach, where the type I error will be split equally between dose level rozanolixizumab so that each dose level will be tested at a 2-sided alpha level of 0.025. Whereas, for families 2-5 the Hochberg truncation parameter is set to 0.2, and for the final family the truncation parameter is 1, so that the standard Hochberg test is used.

The scenarios for the sequential procedure are described below and begins with the evaluation of the primary efficacy endpoint.

**Scenario 1**: One of the two doses of rozanolixizumab is statistically significant for the primary endpoint:

- 1. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in MG-C score at a 2sided alpha level of 0.025. If significant in favor of rozanolixizumab, then proceed to step 2. Otherwise, the testing procedure is concluded.
- 2. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in QMG score at a 2sided alpha level of 0.025. If significant in favor of rozanolixizumab, then proceed to step 3. Otherwise, the testing procedure is concluded.
- 3. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in MG Symptoms PRO 'Muscle Weakness Fatigability' score at a 2-sided alpha level of 0.025. If significant in favor of rozanolixizumab, then proceed to step 4. Otherwise, the testing procedure is concluded.

- 4. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in MG Symptoms PRO 'Physical Fatigue' score at a 2-sided alpha level of 0.025. If significant in favor of rozanolixizumab, then proceed to step 5. Otherwise, the testing procedure is concluded.
- 5. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in MG Symptoms PRO 'Bulbar Symptoms' score at a 2-sided alpha level of 0.025.

Scenario 2: Both doses of rozanolixizumab are statistically significant for the primary endpoint:

- 1. Perform a truncated Hochberg test of rozanolixizumab vs placebo for change from Baseline to Day 43 in MG-C score at a 2-sided alpha level of 0.05:
  - a) Both doses are significant if the larger of the 2-sided p-values is less than or equal to 0.5(1+0.2)\*0.05=0.03. Then 2-sided alpha=0.05 is transferred to the next pairwise comparison (family).
  - b) If the previous step does not hold, then one dose is significant if the smaller 2-sided p-value <0.025. In which case, 2-sided alpha=0.5(1-0.2)\*0.05=0.02 is transferred to the next family.
  - c) Otherwise, the testing procedure is concluded.
- 2. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in QMG score:
  - a) If both doses are significant in the previous family, then perform a truncated Hochberg test at 2-sided alpha=0.05 as described in 1.
  - b) If only 1 dose is significant in the previous family, then perform a 2-sided test alpha=0.02 for the single dose which was significant in the previous family. If this dose is significant then transfer alpha=0.02 to the next family.
  - c) If no significant tests result from scenarios a or b above, then the testing procedure is concluded.
- 3. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in MG Symptoms PRO 'Muscle Weakness Fatigability' score:
  - a) If both doses are significant in the previous family, then perform a truncated Hochberg test at 2-sided alpha=0.05 as described in 1.
  - b) If only 1 dose is significant in the previous family, then perform a 2-sided test at alpha=0.02 for the single dose which was significant in the previous family.
  - c) If no significant tests result from scenarios a or b above, then the testing procedure is concluded.
- 4. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in MG Symptoms PRO 'Physical Fatigue' score:
  - a) If both doses are significant in the previous family, then perform a truncated Hochberg test at 2-sided alpha=0.05 as described in 1.
  - b) If only 1 dose is significant in the previous family, then perform a 2-sided test at alpha=0.02 for the single dose which was significant in the previous family

- c) If no significant tests result from scenarios a or b above, then the testing procedure is concluded
- 5. Test rozanolixizumab vs placebo for change from Baseline to Day 43 in MG Symptoms PRO 'Bulbar Symptoms' score:
  - a) If both doses are significant in the previous family, then perform a standard Hochberg test at 2-sided alpha=0.05. Both doses are significant if the larger of the 2-sided p-values less than 0.5(1+1)\*0.05=0.05. If not, then one dose is significant if the smaller p-value less than 0.025.
  - b) If only 1 dose is significant in the previous family, then perform a 2-sided test at alpha=0.02 for the single dose which was significant in the previous family
  - c) The testing procedure is concluded following steps 5a and 5b.

Note: all p-values used in the above procedure will be based upon the inverse-normal combination approach as described for the primary endpoint.

# 4.7 Use of an efficacy subset of study participants

A sensitivity analysis of the primary endpoint will be performed based on the FAS.

## 4.8 Active-control studies intended to show equivalence

Not applicable.

# 4.9 Examination of subgroups

#### 4.9.1 General subgroups

The primary and continuous secondary efficacy endpoints will be evaluated for subgroups of interest including:

- Age  $(18 < 65 \text{ years}, \ge 65 \text{ years})$
- Age  $(18 <65, 65 <85, \ge 85 \text{ years})$
- Sex (male, female)
- Region (North America, Europe, and Asia [excluding Japan], Japan)
- Stratification factors MG-specific autoantibodies, MuSK(+/-) and AChR(+/-)

Note: The stratification factors MuSK(+/-) and AChR(+/-) in the subgroup analysis will be based on the values from MG-specific autoantibody assessment taken at Baseline, using the same algorithm for missing values as specified in Section 4.1. Historical MuSK (+/non +) and historical AChR(+/non +) will also be examined in the subgroup analysis, in this case, Baseline MuSK(+/-) and Baseline AChR(+/-) will replaced by Historical MuSK (+/non +) and historical AChR (+/non +).

The MG-ADL scores and change from Baseline will be summarized in the five subgroups as above and additional subgroups as follow:

Duration of disease at Baseline (<median, ≥ median)</li>

- MGFA disease class at Baseline
- Thymectomy at Baseline (yes, no)
- Baseline MG-ADL category (<5,  $\ge$ 5).

The following subgroups of MG baseline medications will be derived in the analysis datasets and used for ad-hoc reporting purposes. See Section 6.4.3 for definition of MG baseline medications.

- Baseline Oral steroid (yes, no)
- Baseline Immunosuppressants other than oral steroid (yes, no)
- Baseline Cholinesterase inhibitor (yes, no)

All subgroup analyses will be descriptive; no statistical testing of treatment-by-subgroup interactions nor statistical testing of treatment effects within subgroups will be carried out. No subgroup analysis is planned for safety variables.

Forest plots will be provided to summarize subgroup analysis.

Subgroup analyses will only be performed for subgroups where there are at least 5 study participants in each subgroup level, otherwise it will not be performed.

# 4.9.2 Examination of COVID-19 subgroups

Summary tables will be produced for study participant disposition, demographics and other Baseline characteristics to account for the amount of data captured pre-, during and post- the COVID-19 pandemic. The cut-off dates for the subgroup levels will be defined prior to database lock. Details of the analyses will be specified in the following sections.

## 4.9.3 Examination of weight subgroups and administered doses

To support the goal of a fixed dosing strategy for Rozanolixizumab, additional subgroup analyses will be performed by administered dose group for each weight subgroup below:

- Weight ( $< 50 \text{kg}, 50 < 70 \text{ kg}, 70 < 100 \text{kg}, \ge 100 \text{kg}, \text{total}$ )
- Administered dose (Placebo, RLZ , R

# 5 STUDY POPULATION CHARACTERISTICS

# 5.1 Participant disposition

The following outputs will be created.

Summaries:

- Reasons for screen failures (as collected on the Study Termination Screen Failure Case Report Form [CRF] page) will be summarized using the ES for overall. Additionally, the reasons for screen failures will be summarized by pre-, during and post- the COVID-19 pandemic based on the screen failure date relative to the pandemic cut-off date.
- Disposition of study participants screened will be summarized using the ES for overall,
   by region and by site. In this summary, the site number, principal investigator name, first

participant in date, last participant out date, will be captured by randomized treatment and by each analysis set (RS, SS, FAS and PK-PPS).

- Disposition of analysis sets will be summarized by treatment groups, RLZ total and by analysis sets (RS, SS, FAS and PK-PPS) using the RS.
- Disposition and discontinuation reasons using the RS will contain the number and percentage of study participants who started, completed and permanently discontinued Treatment Period / Observation Period overall and by pre-, during and post- the COVID-19 pandemic based on the start, completed and discontinuation date relative to the pandemic cut-off date. The discontinuation reason in each period will also be summarized. Discontinuation due to COVID-19 pandemic and mandatory withdrawal due to need for rescue therapy and roll over to extension study will be listed as subcategory under "Other" reason.
- Discontinuation due to AEs using the RS will summarize the total number of study
  participants who discontinued the study due to AEs by treatment group, RLZ total and
  the categories: AE serious fatal, AE non-fatal and other AE non-serious fatal.
- Count of participants by visit using RS will summarize the number of participants at each visit by treatment group.
- Impact of COVID-19 for any reason using the RS will summarize number and percentage of study participants in each impact category by visit.

Listings of study participant disposition, study discontinuation and study participants who did not meet study eligibility criteria will be provided.

### 5.2 Protocol deviations

A summary of number and percentage of study participants with an important protocol deviation by relationship to COVID-19 pandemic and treatment group will be provided for the RS. Additionally, the summary will be repeated by pre-, during and post- the COVID-19 pandemic based on the deviations start date relative to the pandemic cut-off date.

A listing of important protocol deviations will be provided based on the RS.

# 6 DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS

# 6.1 Demographics

Demographic variables will be summarized on the RS, by categories mentioned below using descriptive statistics by treatment group, RLZ total and overall. The same summary will also be presented by stages.

## Categories for continuous variables (including n, mean, SD, Median, Min and Max):

- Age at the time of study entry (years) as captured on Demographics CRF
   Notes: Missing age will be calculated as year of informed consent signed year of birth
- Height (cm)
- Weight (kg)

• Body Mass Index (BMI) (kg/m<sup>2</sup>) calculated as:  $BMI = \frac{\text{Weight (kg)}}{(\text{Height (m)})^2}$ 

#### Categorical variables (using frequency counts and percentages):

- Age (18 to <65, 65 to <85,  $\ge 85$  years)
- Age ( $\leq$ 18, 19 to  $\leq$ 65,  $\geq$ 65 years)
- BMI ( $<30 \text{ kg/m}^2$ ,  $\ge 30 \text{ kg/m}^2$ )
- Bodyweight (<50kg, 50kg to <70 kg, 70kg to <100kg,  $\ge100$ kg)
- Bodyweight (<50kg,  $\ge50$ kg)
- Bodyweight (<70kg,  $\ge70$ kg)
- Sex (Male, Female)
- Race (American Indian or Alaska native, Asian, Black, Native Hawaiian or Other Pacific Islander, White, Other/Mixed)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Region (North America, Europe, Asia [excluding Japan], Japan)
- Country

Additional subgroup summary of above variables will be presented by pre-, during and post- the COVID-19 pandemic based on the enrolled date relative to the pandemic cut-off date.

For subgroup summary by weight subgroups and total for the administered dose and RLZ total, following variables will be analyzed:

- Age at the time of study entry (years) as captured on Demographics CRF
- Sex (Male, Female)
- Weight (kg)
- Region (North America, Europe, Asia [excluding Japan], Japan)

A by-participant listing of demographics will be provided using the RS. Childbearing potential and lifestyle will be listed using the ES separately.

# 6.2 Other Baseline characteristics

The following variables will be summarized by treatment group, RLZ total and overall for the RS. The same summary will also be presented by stages:

- MGFA disease class at Baseline
- MG medication as captured on Prior and Concomitant Medications CRF where indication is MG, details in Section 6.4.3
- Myasthenic crisis (yes/no) as captured on History of MG CRF
- Thymectomy (yes, no) as captured on Medical History CRF and Procedure History CRF.
- MG-specific autoantibody (MuSK+ / AChR+) as recorded into the IWRS at randomization

- Historical MuSK antibody status (positive, negative, unknown) as captured on Confirmatory (Historical) Diagnostic Tests for Primary Condition CRF
- Historical AChR antibody status (positive, negative, unknown) as captured on Confirmatory (Historical) Diagnostic Tests for Primary Condition CRF
- Baseline MuSK antibody status (positive, negative, unknown) as evaluated at Baseline visit
- Baseline AChR antibody status (positive, negative, unknown) as evaluated at Baseline visit
- Comparison between historical and Baseline MG-specific autoantibody (MuSK+ / AChR+)
- Baseline MG-ADL score
- Baseline MG-ADL category ( $<5, \ge 5$ )
- Baseline QMG score
- Baseline total IgG value
- Duration of disease (years)

Duration of disease (years) will be calculated as:

Disease Duration = 
$$\frac{\text{(Date of randomization-Date of Initial MG Diagnosis}^{1}+1)}{365.25}$$
.

<sup>1</sup>If the date of initial MG diagnosis is partial, it should be imputed to the most recent feasible date (i.e., last day of the month if only day is missing, or the last day of the year if day and month are missing). Note that if the date of randomization is missing then the duration of disease will be derived using the date of screening.

• Age at initial MG diagnosis (years)

Age at initial MG diagnosis will be calculated as:

Age at initial MG diagnosis = 
$$\frac{\text{(Date of Initial MG Diagnosis}^2 - \text{Date of Birth} + 1)}{365.25}$$

<sup>2</sup>If the date of initial MG diagnosis is partial, it should be imputed to the most recent feasible date (i.e., last day of the month if only day is missing, or the last day of the year if day and month are missing).

The summary will be repeated by pre-, during and post- the COVID-19 pandemic based on the enrolled date relative to the pandemic cut-off date.

Additionally, summary by weight subgroup and total for administered dose and RLZ total will be provided for above variables.

Aby-participant listing of Baseline characteristics will be provided.

# 6.3 Medical history and concomitant diseases

Previous and ongoing medical history will be summarized by treatment group, RLZ total and overall, system organ class (SOC), high level term (HLT) and preferred term (PT). Medical procedures are not coded.
Medical history will be listed for the RS. Besides, history of headaches, procedure history and family medical history for drug-induced liver injury (DILI) will be provided in separate byparticipant listings using the RS.

#### 6.4 Prior and concomitant medications

The number and percentage of study participants taking Past, Prior, Baseline, Concomitant or Concomitant Only medications will be summarized using the RS by Anatomical Therapeutic Chemical (ATC) class, presenting as Anatomical Main Group (ATC Level 1), Pharmacological Subgroup (ATC level 3), PT, treatment group and overall.

Additionally, all rescue medications mentioned in Protocol section 6.5.4 and identified if Rescue Medication is ticked as yes on CRF will be summarized using the RS.

Medications classified as past, prior, Baseline concomitant or concomitant only will be listed using the RS. A by-participant listing of concomitant procedures will also be listed using the RS. Originally reported dates will be used for listings.

#### 6.4.1 Categories of prior and concomitant medications

Medications will be classified as follow based on imputed start and stop dates & times as outlined in Section 4.2.2.

- Past medications will include any medications that started and stopped before the first administration of IMP.
- **Prior** medications will include any medications that started before the first administration of IMP.
- Baseline medications will include any medications that started prior to dosing and continued after (classified as prior and concomitant medications).
- Concomitant medications will include any medications that have been taken at least once after the first administration of IMP during the Treatment and/or Observation Period.
- Concomitant Only medications will include any medication that started after the first administration of IMP and continues during the Treatment and/or Observation Period.

Table 6–1: Concomitant Medications Classification

| Medication Started | Medication finished | Classification |
|---|---|---|
| Before 1st Dose IMP | Before 1 <sup>st</sup> Dose IMP | Past |
| Before 1st Dose IMP | Any time | Prior |
| Before 1st Dose IMP | After 1st Dose IMP | Baseline (= prior and concomitant) |
| Any time | After 1st Dose IMP | Concomitant |
| After 1st Dose IMP | After 1st Dose IMP | Concomitant Only |


#### 6.4.2 Assignment of medications to study period

The following rules will be used to assign a concomitant medication to a study period:

- **Treatment Period:** a medication will be assigned to the Treatment Period if it has been taken at least once between the first administration of IMP on Day 1, up to the minimum of Day 43 and 7 days after the last dose of IMP. This includes medications that started prior to the Treatment Period and those that continued into the Observation Period.
- **Observation Period:** a medication will be assigned to the Observation Period if it has been taken at least once from the day after Treatment Period to the EOS visit. This includes medications that started prior to the Observation Period.

Thus, a medication taken from the time of the first drug administration in the Treatment Period to the end of the study will be assigned to the Treatment Period and the Observation Period.

#### 6.4.3 Baseline MG medication definition

MG Baseline medication is defined as an indication related to MG and includes one of the following ATC codes:

- (Corticosteroids)
- (Immunosuppressants)
- (Parasympathomimetics)

# 7 MEASUREMENTS OF TREATMENT COMPLIANCE

Not applicable. The number of infusions will be recorded as detailed in Section 10.1.

### 8 EFFICACY ANALYSES

All efficacy analyses will be performed using the RS unless specified otherwise, including for the interim analysis.

### 8.1 Handling of intercurrent events

The main intercurrent events (ICEs) of interest are:

- ICE1 The use of rescue therapy prior to Day 43 (Visit 10)
- ICE2 Permanent treatment discontinuation (or withdrawal from study) due to TEAEs

Two additional types of ICEs will be included to account for data affected by the COVID-19 pandemic as follows:

- ICE3 Treatment discontinuation due to suspected/confirmed COVID-19 infection ("Confirmed COVID-19" or "Suspected COVID-19" as the relationship to COVID-19 in the COVID-19 Impact eCRF)
- ICE4 Treatment discontinuation due to non-COVID-19 infection related issues ("General circumstances around COVID-19 pandemic without infection" or "other" as the relationship to COVID-19 in the COVID-19 Impact eCRF)

The number and percentage of study participants with each intercurrent event will be summarized by treatment group and RLZ total.

The strategies to handle ICEs are summarized as below:

| Strategies | Description |
|---|---|
| Hypothetical & treatment policy strategy | If study participants experience ICE1, data at and after the point of the ICE for the purpose of analysis will be treated as missing and imputed under proposed method per Section 4.2.1. |
| | For participants experiencing ICE2-4, data in the Treatment Period from Baseline to Day 43 will be used regardless of whether any ICEs occurred, missing data will be imputed per Section 4.2.1. |
| | For participants who permanently discontinue treatment or withdraw from the study during Treatment Period and who continue into the Observation Period, the observation phase data (collected bi-weekly) will be mapped to the nearest visit for primary analysis where treatment windows will be utilized for the mapping. |
| Treatment policy strategy | The data in the Treatment Period from Baseline to Day 43 will be used regardless of whether any intercurrent events occurred. |
| Composite strategy | The occurrence of any intercurrent events above will be handled by evaluating the corresponding study participants as treatment failures and imputed with a worst score (continuous) or non-responder (binary). |
| COVID-19 Hypothetical strategy | If participant experience ICE1 and/or ICE2, then data at and after the point of the intercurrent event for the purpose of analysis will be treated as missing. |
| strategy | Additionally, participant experience ICE3, ICE4 or those that have visits in treatment period affected (e.g. visit performed by video call) will be completely removed from analysis. |

# 8.2 Statistical analysis of the primary efficacy endpoint

The primary efficacy endpoint is the change from Baseline in MG-ADL score to Day 43 (Visit 10) and will be evaluated under the 'hypothetical & treatment policy' estimand based on RS using Hypothetical & Treatment Policy strategy.

Missing data in the primary analysis will be handled under a missing at random (MAR) assumption.

To check the assumptions around the estimand in the (primary) analysis of the primary endpoint, the following sensitivity and supplemental analyses will be performed:

- A sensitivity analysis using:
  - Hypothetical & treatment policy strategy on FAS:
  - Hypothetical & treatment policy strategy with a J2R approach on missing data will be used to verify the robustness of the MAR approach;
  - Hypothetical & treatment policy strategy based on the subgroup of the RS who received all doses.
  - Hypothetical & treatment policy strategy based on the subgroup of the FAS excluding confirmed COVID-19 cases.
- A supplemental analysis using:
  - Composite strategy to handle the occurrence of an intercurrent event as treatment failures. A trimmed mean approach will be implemented to impute missing data;
  - Treatment policy strategy to allow intercurrent events to be included in the treatment paradigm.

An additional analysis will be performed using COVID-19 Hypothetical strategy on RS.

The methods to handle the missing data caused by occurrence of ICEs in each analysis are detailed in Section 4.2.1.

Please see below for details about the estimands attributes for the evaluation of the primary endpoint (primary, sensitivity and supplemental analyses).

| <b>Study Treatment Name:</b> | Rozanolixizumab<br>(Treatment Arm 1) | Rozanolixizumab<br>(Treatment Arm 2) | Placebo<br>(Treatment Arm 3) |
|---|---|---|---|
| Dosage formulation: | Solution for infusion | Solution for infusion | Aqueous solution |
| Unit dose<br>strength(s)/Dosage<br>level(s): | | | 0.9% sodium chloride aqueous solution (physiological saline, preservative free) |
| Route of Administration | | Subcutaneous (sc) | 20. 4. |
| Dosing instructions: | doses of rozanolixizumab at (equivalent to approximately): Bodyweight <50kg: dose to be administered Bodyweight ≥50kg and <70kg: dose to be administered Bodyweight ≥70kg and <100kg: dose to be administered Bodyweight ≥100kg: dose to be administered | doses of rozanolixizumab at (equivalent to approximately): Bodyweight <50kg: dose to be administered Bodyweight ≥50kg and <70kg: dose to be administered Bodyweight ≥70kg and <100kg: dose to be administered Bodyweight ≥100kg: dose to be administered | doses of placebo at |
| Packaging and Labeling | Rozanolixizumab and matching placebo are manufactured, packaged, and labeled according to Good Manufacturing Practice guidelines and applicable laws or regulations. | | |

- 2. **Population**: study participants with generalized MG who comply with the inclusion/exclusion criteria specified in Section 5 in the study protocol
- 3. Endpoint: please refer to Section 2.2.1.1 for details.
- 4. Intercurrent Events (ICEs): See Section 4.2.1.
- 5. Population Level Summary (PLS): See table below.

Table 8-2: Intercurrent Events and Population Level Summary by Statistical Category

| Statistical<br>Category | Intercurrent Event Strategy | Population Level Summary |
|---|---|---|
| Primary | The ICEs are detailed in Section 8.1. A hypothetical & treatment policy strategy will be used to handle the ICEs. | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the MG-ADL score for study participants receiving rozanolixizumab versus placebo, using the RS. |
| Sensitivity | Hypothetical & treatment policy strategy, same as for the primary analysis | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the MG-ADL score for study participants receiving rozanolixizumab versus placebo, using the FAS. |
| Sensitivity | Hypothetical & treatment policy strategy, same as for the primary analysis Hypothetical & treatment policy strategy, same as for the primary | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the MG-ADL score for study participants receiving rozanolixizumab versus placebo, using the RS. A Jump-to-reference multiple imputation approach will be utilised to assess the validity of the MAR assumption. Missing data across all treatment groups will be imputed using the placebo distribution. |
| Sensitivity | Hypothetical & treatment policy strategy, same as for the primary analysis. | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the MG-ADL score for study participants receiving all doses of rozanolixizumab versus placebo. |
| Sensitivity | Hypothetical & treatment policy strategy, same as for the primary analysis. | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the MG-ADL score on the subgroup of the FAS excluding confirmed COVID-19 cases. |

| Statistical | Intercurrent Event Strategy | Population Level Summary |
|---|---|---|
| Category | | |
| Supplemental | The ICEs are detailed in Section 8.1. A composite strategy will be used to handle the ICEs. | Difference in mean change from Baseline (LSMD from ANCOVA) to Day 43 (Visit 10) in the MG-ADL score for study participants receiving rozanolixizumab versus placebo. A trimmed mean approach will be used where all missing data (including the main intercurrent events) will be imputed with the worst score of its respected questionnaire. A permutation-based test will be carried out, with the % trimming applied adaptively. The mean treatment difference of the trimmed population will be calculated on covariate-adjusted scores which are derived from an ANCOVA analysis of completers data. |
| Supplemental | The ICEs are detailed in Section 8.1. A treatment policy strategy will be used to handle the ICEs. | Difference in mean change from Baseline (LSMD from MMRM) to Day 43 (Visit 10) in the MG-ADL score for study participants receiving rozanolixizumab versus placebo. |

Note: CfB=Change from Baseline; LSMD=Least Squares Mean Difference; MMRM=mixed model for repeated measures; ANCOVA= analysis of covariance; MAR=Missing at Random

### 8.2.1 Derivation of primary efficacy endpoint

The complete list of MG-ADL items and scores are provided in Table 13–3. The total score will be calculated according to the rules set down in Section 13.3. The total score calculated after single item imputation will be used to calculate change from Baseline, in summaries and for efficacy analyses.

### 8.2.2 Primary analysis of the primary efficacy endpoint

The primary analysis is based on the RS under the hypothetical & treatment policy strategy (see details in Section 8.1). Any missing MG-ADL scores (including missing data after the intercurrent events) will be handled based on maximum likelihood estimation method under MAR assumption.

A stage-wise MMRM with treatment group, Baseline MG-ADL score, region, stratification factor(s) including MuSK(+/-) and /or AChR(+/-), and treatment group by day (interaction term) as fixed factors and study participant as a random effect. The MMRM will include Days 8, 15, 22, 29, 36 and 43.

The model will utilize an unstructured covariance pattern for the repeated measures. If the model does not converge using the unstructured pattern, then an autoregressive covariance structure

will be used. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom.

For each stage, the least squares means (LSMs) of each treatment group, and the least squares mean differences (LSMDs) between each dose group and placebo will be reported for Day 43 (Visit 10), along with the corresponding 2-sided 97.5% Cis and p-values.

The study follows a 2-stage group sequential adaptive design using combination test (Lehmacher and Wassmer, 1999) based on the inverse-normal method of combining independent stagewise p-values (Hedges and Olkin, 1985)

The analysis takes into account that the study is a 2-stage group sequential adaptive design assuming equal weighting of each stage, with weights =  $1/\sqrt{2}$ :

- Stage 1 Cohort up to the formal IA
- Stage 2 Cohort post-IA

The following sequential test statistic will be used to test the global null hypothesis at the end of stage 2:

$$T = \sum_{i=1}^{2} w_i \, \phi^{-1} (1 - p_i)$$

Where subscript i=1,2 represents the stage,  $p_i$  represents the appropriate multiplicity adjusted p-value at stage i (for example at stage 1,  $p_1 = \min(2 * p_{\min}, 1)$  where  $p_{\min}$  is the minimum of the two nominal p-values), the weights  $w_{ki} = 1/\sqrt{2}$  satisfy  $\sum_{i=1}^2 w_{ki}^2 = 1$  and  $\phi^{-1}$  is the inverse cumulative standard normal distribution function. The test statistic T and  $z = \phi^{-1}(1-p_i)$  have a standard normal distribution, (Lehmacher and Wassmer, 1999).

The combined p-value (2-sided) for the 2 stages, which tests the global null hypothesis, can be calculated by:

$$p = 2 * \{1 - \phi \left[ \frac{1}{\sqrt{2}} \{ \phi^{-1} (1 - p_1) + \phi^{-1} (1 - p_2) \} \right] \}$$

At the IA one p-value will be computed for each pairwise comparison. Assuming that the trial is not stopped for futility at IA, at the end of the trial the t-test statistics computed at each stage will be used following the p-value combination test method to derive the combined p-value for evaluation of primary efficacy endpoint. Overall statistical significance will be concluded if the combined p-value (2-sided) described above is less than 0.05. For each dose group, statistical significance will be determined in a similar way but using a closed test procedure. Formally, this will be computed as the p-value corresponding to the minimum adjusted Z-statistic of all hypotheses involving the particular dose group being considered. However, if one treatment arm with the largest test statistic is selected for the second stage, the rejection of the global hypothesis implies the rejection of the hypothesis related to the selected hypothesis. The predetermined alpha value for secondary endpoint testing is specified in Section 4.6.

The analysis will be conducted using SAS and RPACT which also produces the combined effect estimates together with multiplicity adjusted 95% CIs. The stagewise inputs for Rpact will be the model Least squares means, standard errors, sample size per group and degrees of freedom (for estimation of the common standard deviation).

The overall confidence intervals at stage 2 are computed separately for each treatment arm that was selected for stage 2. By use of the Inverse-Normal combination function together with the critical value Z<sub>alpha/2</sub>, the lower bound of the 2-sided 95% repeated confidence interval for a given treatment arm is found as the smallest value for which the multiplicity-adjusted combination test yields non-rejection at two-sided alpha=5%. The upper bound of the confidence interval will be found analogously.

8.2.3 Sensitivity analyses of the primary efficacy endpoint

8.2.3.1 Sensitivity Analysis #1

#### 8.2.3.1 Sensitivity Analysis #1

The first sensitivity analysis will be performed based on the FAS using the hypothetical & treatment policy strategy. The method to handle missing MG-ADL scores (including missing data after the intercurrent events) is specified in Section 4.2.1.

The same stage-wise analysis approach as primary analysis (Section 8.2.2) will be repeated.

#### Sensitivity Analysis #2 8.2.3.2

The second sensitivity analysis will be performed based on the RS under the hypothetical & treatment policy strategy. A J2R approach using Multiple Imputation (MI) method under missing not at random (MNAR) assumption will be used to handle any missing MG-ADL scores (including missing data after the intercurrent events). Missing data will be imputed based on the placebo group distribution, irrespective of individual treatment assignment.

The following is a summary of the imputation method.

100 imputed datasets (m) will be created using monotone linear regression imputation methods which will impute the study participants' missing post-baseline scores at each of the scheduled visits in the study (i.e., Days 1, 8, 15, 22, 29, 36 and 43). If the missing data does not follow a monotonic pattern, a sequential approach to imputing the data to produce a monotone missing data pattern will be applied using the MCMC impute=monotone option in PROC MI (SAS System). Then the monotone linear regression imputation methods will be applied.

The MI method allows for a pattern-mixture model approach assuming the data are MNAR. The MNAR option in PROC MI (SAS system) will be used to impute the placebo distribution as described in Yuan (2014).

Each of the imputed datasets will be analyzed via the specified MMRM model (see Section 8.2.2). The treatment effects and standard errors from LSMs and LSMDs will be combined across the 100 imputed datasets to produce an overall LSMs and LSMDs with associated p-value and 97.5 % CI using SAS PROC MIANALYZE.

The following variables will be included in the imputation model:

- o Baseline MG-ADL Score (continuous variable)
- MG-ADL Score at Days 8, 15, 22, 29, 36 and 43 (continuous variable)

Note: if the MI model does not converge or produce estimates (e.g., due to over-specification) the set of imputation variables may be modified.

#### 8.2.3.3 Sensitivity Analysis #3

The third sensitivity analysis will be performed based on the subgroup of the RS who received all 6 (sc) doses of IMP in the treatment period, using the hypothetical & treatment policy strategy and same missing data handling method as mentioned in Section 4.2.1.

The same stage-wise analysis approach as primary analysis (Section 8.2.2) will be repeated.

#### 8.2.3.4 Sensitivity Analysis #4

The fourth sensitivity analysis will be performed for the primary endpoint on the FAS excluding confirmed COVID-19 cases under the treatment policy strategy.

The method to handle missing MG-ADL scores (including missing data after the intercurrent events) is specified in Section 4.2.1.

The same stage-wise analysis approach as primary analysis (Section 8.2.2) will be repeated.

#### 8.2.4 Supplementary analyses of the primary efficacy endpoint

#### 8.2.4.1 Supplementary Analysis #1

The first supplementary analysis will be performed based on the RS, using the composite strategy (see details in Section 8.1). A trimmed mean approach, where missing data are assumed to be missing not at random (MNAR), will be used to impute missing MG-ADL scores (including the intercurrent events) with the worst score of the MG-ADL questionnaire.

The trimmed mean approach will be applied for each stage separately as follows:

- 1. Perform an analysis using ANCOVA model with treatment group, Baseline MG-ADL score, region, stratification factors (MuSK+/- and AChR+/-) as fixed effects excluding any study participants with missing data at Day 43 or who experienced an intercurrent event by Day 43.
- 2. Retain the coefficients from the model for Baseline MG-ADL score, region, and stratification factors (MuSK+/- and AChR+/-).
- 3. Calculate the adjusted endpoint for each study participant as based on the raw CfB and coefficients calculated from the ANCOVA in Step 1: Adjusted CfB = Raw CfB Stratification Coefficient\*Stratification (AChR/ MuSK) Baseline Score Coefficient\*Baseline MG-ADL score Region Coefficient\*Region.
- 4. Identify any study participants with missing data at Day 43 and any study participants who experienced any intercurrent event by Day 43. A worst score (i.e., 24) will be imputed for these study participants at Day 43 in order to flag them as worse responders than any subject who completes.
- 5. Determine the trim fraction to be used. This will be the maximum of dropout and intercurrent event rate in each of the three treatment groups. For example, if the rate of dropout/IE in the three groups is 10, 15 and 20% then the worst 20% of each group will be the trimmed.
- 6. Sort each treatment group in ascending order by adjusted endpoint Day 43 MG-ADL score and trim equal fractions from each treatment group that was calculated in Step 5 from the bottom.

- 7. Calculate the mean adjusted CfB score of the trimmed sample for each treatment group and the difference between trimmed means of each rozanolixizumab group and placebo.
- 8. Repeat Steps 5-7 (above) 10,000 times but each time with a new treatment group assignment (which is a permutation of the original treatment labels, i.e. take a 100% random sample of the original treatment variable without replacement) and a new trimming fraction appropriate to the current permutation.
- 9. Order the 10,000 permuted trimmed mean differences and count the number of those mean differences that exceed the observed trimmed mean difference calculated in Step 7 as  $n_1$ .
- 10. Then the 1-sided empirical p-value of the original trimmed mean difference =  $n_1/10000$ .

The one-sided p-values will be presented for each rozanolixizumab dose compared to placebo.

The p-values from Stage 1 and Stage 2 will be combined in the same manner as the primary analysis. Specifically, the final one-sided p-value is  $p = 1 - \phi \left[ \frac{1}{\sqrt{2}} \left\{ \phi^{-1} (1 - p_1) + \phi^{-1} (1 - p_2) \right\} \right]$ .

#### 8.2.4.2 Supplementary Analysis #2

The second supplementary analysis of the primary endpoint will be performed using a treatment policy strategy (see details in Section 8.1) based on the RS. Any missing MG-ADL scores will be handled based on maximum likelihood estimation method under MAR assumption.

The same stage-wise analysis approach as primary analysis (Section 8.2.2) will be repeated.

#### 8.2.5 Additional Analysis

An additional analysis of primary endpoint will be performed on RS under the COVID-19 hypothetical strategy (see details in Section 8.1). The same stage-wise analysis approach as primary analysis (Section 8.2.2) will be repeated.

### 8.2.6 Exploratory Analysis

An exploratory analysis of primary endpoint using historical MG-specific auto-antibodies as a covariate instead of Baseline MG-specific auto-antibodies. This analysis will be performed on RS under the hypothetical & treatment policy strategy (see details in Section 8.1). The same stage-wise analysis approach as primary analysis (Section 8.2.2) will be repeated.

## 8.3 Statistical analysis of the secondary efficacy endpoints

All secondary efficacy endpoints will be tested according to the testing strategy defined in Section 4.6.

Please see below for details about the estimands attributes for the evaluation of the secondary endpoints (secondary and sensitivity analyses).

- 1. **Treatment Conditions**: same as described in the estimand for the primary endpoint (Table 8-1).
- 2. **Population**: same as described in the estimand for the primary endpoint (Section 8.2).
- 3. Endpoints, ICEs and PLS: Please see Table 8-3 below.

Table 8-3: Secondary Efficacy Endpoints: Intercurrent Events and Population Level Summary by Statistical Category

| Statistical<br>Category | Endpoint | Intercurrent Event Strategy | Population Level Summary |
|---|---|---|---|
| Secondary | MG-ADL responder (≥2.0 points improvement from Baseline) at Day 43 (Visit 10) | The ICEs are detailed in Section 8.1. A composite strategy will be used to handle the ICEs. | Odds ratio at Day 43 (Visit 10) analyzed using a logistic regression model adjusting for covariates for study participants receiving rozanolixizumab versus placebo, using the RS. |
| Secondary | Change from<br>Baseline to<br>Day 43 (Visit<br>10) in MG-C<br>score | The ICEs are detailed in Section 8.1. A hypothetical & treatment policy strategy will be used to handle the ICEs. | Difference in mean change from Baseline (LSMD from MMRM) to Day 43 (Visit 10) in the MG-C sco for study participants receiving rozanolixizumab versus placebo. |
| Sensitivity | Change from<br>Baseline to<br>Day 43 (Visit<br>10) in MG-C<br>score | The ICEs are detailed in Section 8.1. A hypothetical & treatment policy strategy will be used to handle the ICEs. | Difference in mean change from Baseline (LSMD from CfB MMR) to Day 43 (Visit 10) in the MG-C score for study participants received rozanolixizumab versus placebo, using the RS. A J2R multiple imputation approach will be utilised to assess the validity of the MAR assumption. Missing data across at treatment groups will be imputed using the placebo distribution. |


| Statistical<br>Category | Endpoint | Intercurrent Event Strategy | Population Level Summary |
|---|---|---|---|
| Supplemental | Change from Baseline to Day 43 (Visit 10) in MG-C score | The ICEs are detailed in Section 8.1. A composite strategy will be used to handle the ICEs. | Difference in mean change from Baseline (LSMD from ANCOVA) to Day 43 (Visit 10) in the MG-C score for study participants receiving rozanolixizumab versus placebo. A trimmed mean approach will be used where all missing data (including the main intercurrent events) will be imputed with the worst score of its respected questionnaire. A permutation-based test will be carried out, with the % trimming applied adaptively. The mean treatment difference of the trimmed population will be calculated on covariate-adjusted scores which are derived from an ANCOVA analysis of completers data, using the RS. |
| Secondary | Change from<br>Baseline to<br>Day 43 (Visit<br>10) in QMG<br>score | Hypothetical & treatment policy strategy, same as for the MG-C secondary analysis | Difference in mean change from<br>Baseline (LSMD from MMRM) to<br>Day 43 (Visit 10) in the QMG score<br>for study participants receiving<br>rozanolixizumab versus placebo. |
| Sensitivity | Change from<br>Baseline to<br>Day 43 (Visit<br>10) in QMG<br>score | Hypothetical & treatment policy strategy, same as for the MG-C sensitivity analysis | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the QMG score for study participants receiving rozanolixizumab versus placebo, using the RS. A J2R multiple imputation approach will be utilised, same as the MG-C sensitivity analysis |
| Supplemental | Change from<br>Baseline to<br>Day 43 (Visit<br>10) in QMG<br>score | Composite strategy, same as for the MG-C supplemental analysis | Difference in mean change from Baseline (LSMD from ANCOVA) to Day 43 (Visit 10) in the QMG score for study participants receiving rozanolixizumab versus placebo. A trimmed mean approach will be used, as the MG-C supplemental analysis |


| Statistical<br>Category | Endpoint | Intercurrent Event Strategy | Population Level Summary |
|---|---|---|---|
| Secondary | Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Muscle Weakness Fatigability' score | Hypothetical & treatment policy strategy, same as for the MG-C secondary analysis | Difference in mean change from Baseline (LSMD from MMRM) to Day 43 (Visit 10) in the MG Symptoms PRO 'Muscle Weakness Fatigability' score for study participants receiving rozanolixizumab versus placebo. |
| Sensitivity | Change from Baseline to Day 43 (Visit 10) in MG Symptoms PRO 'Muscle Weakness Fatigability' score | Hypothetical & treatment policy strategy, same as for the MG-C sensitivity analysis | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the QMG score for study participants receiving rozanolixizumab versus placebo, using the RS. A J2R multiple imputation approach will be utilised, same as the MG-C sensitivity analysis |
| Supplemental | Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Muscle Weakness Fatigability' score | Composite strategy, same as for the MG-C supplemental analysis | Difference in mean change from Baseline (LSMD from ANCOVA) to Day 43 (Visit 10) in the MG Symptoms PRO 'Muscle Weakness Fatigability' score for study participants receiving rozanolixizumab versus placebo. A trimmed mean approach will be used, as the MG-C supplemental analysis |
| Secondary | Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Physical Fatigue' score | Hypothetical & treatment policy strategy, same as for the MG-C secondary analysis | Difference in mean change from<br>Baseline (LSMD from MMRM) to<br>Day 43 (Visit 10) in the MG<br>Symptoms PRO 'Physical Fatigue'<br>score for study participants receiving<br>rozanolixizumab versus placebo. |

| Statistical<br>Category | Endpoint | Intercurrent Event Strategy | Population Level Summary |
|---|---|---|---|
| Sensitivity | Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Physical Fatigue' score | Hypothetical & treatment policy strategy, same as for the MG-C sensitivity analysis | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the MG Symptoms PRO 'Physical Fatigue' score for study participants receiving rozanolixizumab versus placebo, using the RS. A J2R multiple imputation approach will be utilised, same as the MG-C sensitivity analysis |
| Supplemental | Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Physical Fatigue' score | Composite strategy, same as for the MG-C supplemental analysis | Difference in mean change from Baseline (LSMD from ANCOVA) to Day 43 (Visit 10) in the MG Symptoms PRO 'Physical Fatigue' score for study participants receiving rozanolixizumab versus placebo. A trimmed mean approach will be used, as the MG-C supplemental analysis |
| Secondary | Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Bulbar Symptoms' score | Hypothetical & treatment policy strategy, same as for the MG-C secondary analysis | Difference in mean change from Baseline (LSMD from MMRM) to Day 43 (Visit 10) in the MG Symptoms PRO 'Bulbar Symptoms' score for study participants receiving rozanolixizumab versus placebo. |
| Sensitivity | Change from<br>Baseline to<br>Day 43 (Visit<br>10) in the<br>MG<br>Symptoms<br>PRO 'Bulbar<br>Symptoms'<br>score | Hypothetical & treatment policy strategy, same as for the MG-C sensitivity analysis | Difference in mean change from Baseline (LSMD from CfB MMRM) to Day 43 (Visit 10) in the MG Symptoms PRO 'Bulbar Symptoms' score for study participants receiving rozanolixizumab versus placebo, using the RS. A J2R multiple imputation approach will be utilised, same as the MG-C sensitivity analysis |

| Statistical<br>Category | Endpoint | Intercurrent Event Strategy | Population Level Summary |
|---|---|---|---|
| Supplemental | Change from Baseline to Day 43 (Visit 10) in the MG Symptoms PRO 'Bulbar Symptoms' score | Composite strategy, same as for the MG-C supplemental analysis | Difference in mean change from Baseline (LSMD from ANCOVA) to Day 43 (Visit 10) in the MG Symptoms PRO 'Bulbar Symptoms' score for study participants receiving rozanolixizumab versus placebo. A trimmed mean approach will be used, as the MG-C supplemental analysis |

Note: CfB=Change from Baseline; LSMD=Least Squares Mean Difference; MMRM=mixed model for repeated measures; ANCOVA= analysis of covariance; MAR=Missing at Random

### 8.3.1 MG-ADL Responder Rate at Visit 10 (Day 43)

See Section 8.2.1 for the derivation of MG-ADL total score.

Study participants will be classified as responders at Visit 10 if the value is at least a 2-point improvement (decrease) from Baseline at Visit 10 (Day 43).

Analysis will be based on the RS under the composite strategy (see details in Section 8.1). Any missing data scores (including missing data due to the intercurrent events) will also be imputed as non-responders. Note that this endpoint is not part of the formal secondary endpoint testing strategy.

The number and percentage of study participants who are MG-ADL responders at Day 43 will be presented by treatment group and RLZ total for each stage. The odds ratio of the responder rates at Day 43 will be estimated and tested between treatment groups (each rozanolixizumab dose vs placebo) for each stage separately using logistic regression model with factors of treatment group, Baseline MG-ADL score and stratification factors (MuSK+/- and AChR+/-). The odds ratio with associated 95% CI and p-value based on the Wald test will be presented. Region may be added as an additional factor in the logistic regression model if significant in the primary analysis.

The odds ratios, 95% CIs, and p-values from each stage will be combined using the same inverse normal method used in the primary efficacy endpoint.

# 8.3.2 Change from Baseline to Day 43 (Visit 10) in MG-C score

The complete list of MG-C items and scores are provided in Table 13–2. The total score will be calculated according to the rules set down in Section 13.2. This total score will be used to calculate change from Baseline, in summaries and for efficacy analysis.

The following analyses will be performed:

- Secondary: The same approach as specified in Section 8.2.2 will be implemented.
- Sensitivity: The same approach as Section 8.2.3.2 will be applied.
- Supplemental: The same approach as Section 8.2.4.1 will be applied. The worst MG-C total score is 50.

- Additional: The same approach as Section 8.2.5 will be applied.
- Exploratory: The same approach as Section 8.2.6 will be applied.

#### 8.3.3 Change from Baseline to Day 43 (Visit 10) in QMC score

The complete list of QMG items and scores are provided in Table 13–1. Partially missing total scores will be imputed according to the rules set down in Section 13.1. This total score after single item imputation will be used to calculate change from Baseline, in summaries and for efficacy analysis.

The following analyses will be performed:

- Secondary: The same approach as specified in Section 8.2.2 will be implemented.
- Sensitivity: The same approach as Section 8.2.3.2 will be applied.
- Supplemental: The same approach as Section 8.2.4.1 will be applied. The worst QMG total score is 39.
- Additional: The same approach as Section 8.2.5 will be applied.
- Exploratory: The same approach as Section 8.2.6 will be applied.

#### 8.3.4 Change from Baseline in PRO Muscle Weakness Fatigability score

The PRO Muscle Weakness Fatigability score is based on the MG symptoms PRO instrument items 34-42. See Section 13.4 for the complete list of MG symptoms PRO items and scoring details.

The following analyses will be performed:

- Secondary: The same approach as specified in Section 8.2.2 will be implemented.
- Sensitivity: The same approach as Section 8.2.3.2 will be applied.
- Supplemental: The same approach as Section 8.2.4.1 will be applied. The worst PRO Muscle Weakness Fatigability score is 100.
- Additional: The same approach as Section 8.2.5 will be applied.
- Exploratory: The same approach as Section 8.2.6 will be applied.

#### 8.3.5 Change from Baseline in PRO Physical Fatigue score

The PRO Physical Fatigue score is based on the MG symptoms PRO instrument items 19-33.

The same stage-wise MMRM model and analysis approach as specified in Section 8.2.2 will be implemented to test for superiority.

The following analyses will be performed:

- Secondary: The same approach as specified in Section 8.2.2 will be implemented.
- Sensitivity: The same approach as Section 8.2.3.2 will be applied.
- Supplemental: The same approach as Section 8.2.4.1 will be applied. The worst PRO Physical Fatigue score is 100.

- Additional: The same approach as Section 8.2.5 will be applied.
- Exploratory: The same approach as Section 8.2.6 will be applied.

#### 8.3.6 Change from Baseline in PRO Bulbar Symptoms score

The PRO Bulbar Symptoms score is based on the MG symptoms PRO instrument items 6-15. The following analyses will be performed:

- Secondary: The same approach as specified in Section 8.2.2 will be implemented.
- Sensitivity: The same approach as Section 8.2.3.2 will be applied.
- Supplemental: The same approach as Section 8.2.4.1 will be applied. The worst PRO Bulbar Symptoms score is 100.
- Additional: The same approach as Section 8.2.5 will be applied.
- Exploratory: The same approach as Section 8.2.6 will be applied.

#### 8.4 Analysis of other efficacy endpoints

All other efficacy variables will be summarized overall using descriptive statistics, unless specified otherwise. No stage-wise summary will be performed, except for time to MG-ADL response. Missing data will be handled as described in Section 4.2.1.

#### 8.4.1 Use of rescue therapy due to worsening (IVIg, PEX)

The use of rescue therapy will be identified by a 'yes' response to the "Rescue Medication?" question on the concomitant medication CRF, or plasma exchange as collected on concomitant medical procedure CRF".

The number of study participants in each treatment group that use rescue therapy due to worsening (IVIg, PEX) will be summarized by treatment group and RLZ total.

The nominal p-value (calculated using a Pearson's Chi-Squared test for independence) will be presented for the difference between each rozanolixizumab dose and placebo in the percent of study participants using rescue therapy at a 2-sided 0.05 alpha level.

#### 8.4.2 Time to first rescue therapy

Time to first rescue therapy (in days) is defined as: Date of first rescue therapy use—Date of first IMP + 1.

Time to first rescue therapy will be estimated and presented using the Kaplan-Meier product-limit method for each treatment. Study participants who do not take rescue therapy will be censored at the date of withdrawal/study completion. Where there are several AEs which led to drop out, consider the earliest starting AE.

The number of study participants with first rescue therapy and number of censored study participants up to 8, 12, 24, 32, 43, 57, 71, 85, 99 days will be summarized using descriptive statistics.

The median time to first rescue therapy, including the two-sided 95% CI, will be calculated for each treatment.

#### 8.4.3 Time to MG-ADL response (≥2.0 points improvement from Baseline)

Time to MG-ADL response (in days) is defined as Date of First MG-ADL Response—Date of MG-ADL Baseline + 1.

Study participants who use rescue therapy prior to Day 43 or who are withdrawn from the treatment/study due to TEAEs before achieving first MG-ADL response will be censored at time of event. Study participants who never achieve a response by Day 43 will be censored at the date of their last MG-ADL assessment.

The number of study participants with 8, 12, 24, 32, 43 days to first MG-ADL response and number of censored study participants will be summarized descriptively.

Time to first MG-ADL response will be analyzed using a Cox Proportional Hazards model including fixed terms for treatment and stratification factors (MuSK+/- or AChR+/-). This model will be performed separately for study participants included in the interim analysis and for all study participants overall. Region may be added as an additional factor in the Cox Proportional Hazards model if it is significant in the primary analysis.

The Hazard Ratio (test/reference), 95% CI and p-values for each treatment comparison of interest will be presented for the Stage 1 (interim analysis), Stage 2 and overall (all data combined).

The log-hazard ratio, standard error estimates and (1-sided) p-values from the separate stagewise Cox Proportional Hazards models for the relevant treatment group will be used to create overall p-values and repeated confidence intervals using the same methodology as the primary efficacy analysis.

The time to first MG-ADL response will be presented graphically using a Kaplan-Meier curve by treatment group, RLZ total. See details in Section 9.3.2.

#### 8.4.4 QMG score

The QMG scores and change from Baseline will be summarized by treatment group, RLZ total and visit using descriptive statistics. The subgroup summaries will also be performed by MG-specific autoantibody (MuSK+ or AChR+) and by administered dose for each weight subgroup as specified in Section 4.9.1 and Section 4.9.3.

The QMG score (excluding ocular items) change from Baseline will be calculated the same as the change from Baseline in the QMG score. The QMG scores (excluding ocular items) and change from Baseline will be summarized by treatment group, RLZ total and visit using descriptive statistics.

Above QMG summaries will be repeated for COVID-19 free participants, where COVID-19 free participants exclude:

- Participants who discontinue treatment due to suspected/confirmed COVID-19 infection ("Confirmed COVID-19" or "Suspected COVID-19" as the relationship to COVID-19 in the COVID-19 Impact eCRF);
- Participants who discontinue treatment due to non-infection related COVID-19 issues ("General circumstances around COVID-19 without infection" or "other" as the relationship to COVID-19 in the COVID-19 Impact eCRF);

• Participants have visits affected in treatment period (e.g. visit performed by video call) due to COVID-19.

A boxplot of change from Baseline at Day 43 and a time plot of mean change and percentage change from Baseline for QMG will also be plotted by the following dose groups: placebo,

By-participant listings of QMG scores will be provided.

#### 8.4.5 QMG responder rate (≥3.0 points improvement from Baseline)

Study participants will be classified as responders at a visit if the value is at least a 3-point improvement (decrease) from Baseline. Missing data will be imputed using NRI per Section 4.2.1.

The number and percentage of observed and imputed responders will be summarized separately by treatment group, RLZ total and visit. In addition, QMG responders will be summarized by MG-specific autoantibody (MuSK+ or AChR+) and by administered dose for each weight subgroup as specified in Section 4.9.1 and Section 4.9.3. Same summaries will be repeated for COVID-19 free participants as defined in Section 8.4.4.

#### 8.4.6 MG-C score

The total scores and total score (excluding ocular items) with associated change from Baseline will be summarized by treatment group and RLZ total at scheduled visit using descriptive statistics. The subgroup summaries will also be performed by MG-specific autoantibody (MuSK+ or AChR+) and by administered dose for each weight subgroup as specified in Section 4.9.1 and Section 4.9.3. Same summaries will be repeated for COVID-19 free participants as defined in Section 8.4.4.

A boxplot of change from Baseline at Day 43 and a time plot of mean change and percentage change from Baseline for MG-C will also be plotted by the following dose groups: placebo,

By-participant listings of MG-C scores will be provided.

### 8.4.7 MG-C responder rate (≥3.0 points improvement from Baseline)

Participants will be classified as responders at a visit if the value is at least a 3-point improvement (decrease) from Baseline (Burns, Ted M et al [2010]). Missing data will be imputed using NRI per Section 4.2.1.

The number and percentage of observed and imputed responders will be summarized separately by treatment group, RLZ total and visit. In addition, MG-C responders will be summarized by MG-specific autoantibody (MuSK+ or AChR+) and by administered dose for each weight subgroup as specified in Section 4.9.1 and Section 4.9.3. Same summaries will be repeated for COVID-19 free participants as defined in Section 8.4.4.

#### 8.4.8 MG-ADL score

See Section 8.2.1 for the derivation of MG-ADL total score.

The MG-ADL scores and change from Baseline will be summarized by treatment group, RLZ total and visit using descriptive statistics. The subgroup summaries will also be performed by

subgroups in Section 4.9.1 and by administered dose for each weight subgroup as specified in Section 4.9.3.

The MG-ADL score (excluding ocular items) change from Baseline will be calculated the same as the change from Baseline in the MG-ADL score. The MG-ADL scores (excluding ocular items) and change from Baseline will be summarized by treatment group, RLZ total and visit using descriptive statistics.

The mean change from Baseline with 95% CI in MG-ADL total score over time with cumulative ADA or NAb status will be plotted by treatment group and RLZ total. See details in Section .

A boxplot of change from Baseline at Day 43 and a time plot of mean change and percentage change from Baseline for MG-ADL will also be plotted by the following dose groups: placebo,

The study participants with missing MG-ADL assessment and associated reasons at each scheduled visit will be summarized by treatment group and RLZ total. Same summaries will be repeated for COVID-19 free participants as defined in Section 8.4.4.

By-participant listings of MG-ADL values will be provided.

### 8.4.9 MG-ADL responder rate (≥2.0 points improvement from Baseline)

Derivation of the responder is detailed in Section 8.3.1.

The number and percentage of observed and imputed responders will be summarized separately by treatment group, RLZ total and visit. In addition, MG-ADL responders will be summarized by subgroups in Section 4.9.1 and by administered dose for each weight subgroup as specified in Section 4.9.3. Same summaries will be repeated for COVID-19 free participants as defined in Section 8.4.4.

#### 8.4.10 MG Symptoms PRO 'Physical Fatigue' score

See Section 8.3.5 for the derivation of MG Symptoms PRO 'Physical Fatigue' score.

The PRO Physical Fatigue scores and change from Baseline will be summarized by treatment group, RLZ total and visit using descriptive statistics. The subgroup summaries will also be performed by MG-specific autoantibody (MuSK+ or AChR+) and by administered dose for each weight subgroup as specified in Section 4.9.1 and Section 4.9.3.

In addition, empirical cumulative distribution functions of the change in score from Baseline to Day 43 will be plotted by treatment group and RLZ total.

By-participant listings of all MG Symptoms PRO values will be provided.

### 8.4.11 MG Symptoms PRO 'Muscle Weakness Fatigability'

See Section 8.3.4 for the derivation of MG Symptoms PRO 'Muscle Weakness Fatigability' score.

The PRO Muscle Weakness Fatigability scores and change from Baseline will be summarized by treatment group, RLZ total and visit using descriptive statistics. The subgroup summaries will also be performed by MG-specific autoantibody (MuSK+ or AChR+) and by administered dose for each weight subgroup as specified in Section 4.9.1 and Section 4.9.3.

In addition, empirical cumulative distribution functions of the change in score from Baseline to Day 43 will be plotted by treatment group and RLZ total.

#### 8.4.12 MG Symptoms PRO 'Bulbar Symptoms'

See Section 8.3.6 for the derivation of MG Symptoms PRO 'Bulbar Symptoms' score.

The PRO Bulbar Symptoms scores and change from Baseline will be summarized by treatment group, RLZ total and visit using descriptive statistics. The subgroup summaries will also be performed by MG-specific autoantibody (MuSK+ or AChR+) and by administered dose for each weight subgroup as specified in Section 4.9.1 and Section 4.9.3.

In addition, empirical cumulative distribution functions of the change in score from Baseline to Day 43 will be plotted by treatment group and RLZ total.

#### 8.4.13 Patient Global Impressions of Severity

A frequency table will be produced to summarize answers provided to the PGI-S ("none," "mild," "moderate," "severe," "very severe,") for each visit by treatment group and RLZ total.

A by-participant listing of PGI-S will be provided.

### 8.4.14 Patient Global Impressions of Change

A frequency table will be produced to summarize answers provided to the PGI-C ("very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse") for each visit by treatment group and RLZ total.

A by-participant listing of PGI-C will be provided.

# 8.4.15 MGII overall scores, ocular sub-scores, and generalized domain scores

The complete list of MGII items and scores are provided in Table 13-8. The total score will be calculated according to the rules set down in Section 13.5.

Summary statistics of the actual values and change from Baseline values will be used to summarize the MGII overall score and sub-scores separately by treatment group and RLZ total for each visit during Treatment period.

A by-participant listing of MGII scores will be provided.

#### 8.4.16 MG-QOL15r

The total score is calculated by summing all the individual items. See Section 13.6 for scoring details.

Summary statistics of the actual values and change from Baseline values will be used to summarize MG-QOL15r scores by treatment group and RLZ total for each visit.

A by-participant listing of MG-QOL15r scores will be provided.

#### 8.4.17 EQ-5D-5L

The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).

A frequency table will be produced to summarize answers provided to each of the 5 dimensions of the EQ-5D descriptive system at each scheduled visit by treatment group. The observed values of EQ VAS scores and change from Baseline will be summarized by treatment group and RLZ total at each scheduled visit. No imputation will be applied on missing item in EQ-5D descriptive system and EQ VAS.

A by-participant listings of EQ-5D-5L will be provided.

#### 8.4.18 Minimal symptom expression

Minimum Symptom Expression (MSE) is designed to assess how many study participants become free or virtually free of MG symptoms as measured by achieving an MG-ADL total score of 0 or 1 (Vissing et al. 2020). See Section 8.2.1 for the derivation of MG-ADL total score.

The number and percentage of study participants achieving MSE at any time during the treatment and observation phases will be summarized by treatment group and RLZ total.

#### 9 PHARMACOKINETICS AND PHARMACODYNAMICS

All analyses described in Section 9.1 will be performed on the PK-PPS, and all other analysis will be performed on Safety Set.

#### 9.1 Pharmacokinetics

Individual plasma concentrations of rozanolixizumab will be summarized by treatment group and overall for administered RLZ dose and RLZ total and scheduled sampling day for the PK-PPS using n, arithmetic mean, median, SD, minimum, maximum, geometric mean (geomean) with associated 95% CI, and geometric coefficient of variation (geoCV) (assuming log-normally distributed data).

A scatter plot of combined individual concentration versus time profiles will be presented in linear scale by treatment group with all study participants overlaid on the same plot, including day 3, 6, 24, 38, 41. The same plot will also be presented by administered RLZ dose ( ) and RLZ total.

Furthermore, a plot time course plot of geometric mean concentrations by administered RLZ dose will be presented by treatment group and RLZ total. See details in Section 4.9.3.

All figures will include the lower limit of quantification (LLOQ) on the semi-logarithmic plots.

The following rules will apply for PK data listings and summaries:

- Values below the LLOO will be reported as below the limit of quantification (BLO)
- Descriptive statistics of concentrations will be calculated if at most 1/3 of the individual data points at a timepoint are missing or are not quantifiable (<LLOQ). Values that are BLQ will be replaced by the numerical value of the LLOQ/2 in this instance. If more than 1/3 of the individual data points at a timepoint are missing or are not quantifiable, then only n, minimum, median and maximum will be presented. The other descriptive statistics will be left blank.
- If n<3, then only the n, minimum and maximum will be presented. If no study participants have data at a given timepoint, then only n=0 will be presented.

• The 95% CI lower and 95% CI upper should be left blank if the SD (or equivalently, the geoCV) is 0

The geoCV will be calculated using the following formula where SD is the standard deviation from the log-transformed data  $geoCV(\%) = \sqrt{exp(SD^2) - 1} \times 100$ .

Individual concentrations of rozanolixizumab will be listed by treatment group and RLZ total for the PK-PPS and will include the actual sampling time in days relative to the previous dose, the IgG observed at the same visit, the ADA titer observed for the binding assay and the NAb titer for the same visit, and change from Baseline in total IgG and IgG subclasses for the corresponding visit.

#### 9.2 Pharmacodynamics

#### 9.2.1 MG-specific autoantibodies

MG-specific autoantibodies (anti-MuSK/anti-AChR) Baseline values will be based on the last available assessment value prior to first IMP (excluding historical data collected on CRF since the assays were not from the same vendor as specified in this study).

MG-specific autoantibodies (anti-MuSK/anti-AChR) will be summarized by treatment group and RLZ total at scheduled visit for observed values, absolute and percentage changes from Baseline. Additional summary of absolute and percentage changes from Baseline in MG-specific autoantibodies (anti-MuSK/anti-AChR) will be performed by weight subgroup and total for administered dose and RLZ total at scheduled visit (reference Section 4.9.3). The maximum decrease from Baseline in MG-specific autoantibodies (change and percentage change) will be reported in the listing and summarized for each treatment.

Mean and mean percentage change from Baseline values in MG-Specific autoantibodies will be plotted over time by treatment, RLZ total and period with all treatments overlaid on the same plot and the plot will be repeated for the following dose groups: placebo,

Mean percent change from baseline of anti-MuSK and Total IgG, and mean change from baseline of MG-ADL, QMG, MG-C will be plotted over time by treatment and RLZ total for only participants who are anti-MuSK positive at baseline; Additionally, data from individual study participant will be plotted representing percentage change from Baseline in anti-MuSK and Total IgG, and MG-ADL, QMG, MG-C change from Baseline for only participants who are anti-MuSK positive at baseline. The same plots will be repeated for percentage change from Baseline values in anti-AChR for only participants who are anti-AChR positive at baseline.

A boxplot of maximum percentage change from Baseline for MG-specific autoantibodies will be plotted by the following dose groups: placebo,

MG-specific autoantibodies will be listed, together with total IgG, IgG subclasses, MG-ADL, QMG, MG-C change from Baseline.

The correlation between screening and Baseline assay (positive, negative) will be presented based on the Pearson correlation test.

#### 9.2.2 Total serum IgG and IgG subclasses

Total serum IgG concentrations and IgG subclasses will be summarized by treatment group, RLZ total and time point for observed values, change from Baseline, and percentage change from Baseline. Additional summary of absolute and percentage changes from Baseline in total IgG will be performed by weight subgroup and total for administered dose and RLZ total at scheduled visit (reference section 4.9).

The maximum change and percent change from Baseline in total serum IgG and IgG subclasses will be reported in the listing and summarized for each treatment. In the event that a decrease from Baseline in total serum IgG or IgG subclass is not observed in a given study participant, the maximum change will be reported as the smallest increase from Baseline.

Mean change and percent change from Baseline values in total serum IgG will be plotted over time by treatment and RLZ total with all treatments overlaid on the same plot, and the plot will be repeated by the following dose groups: placebo,

Spaghetti plots will be provided for total IgG and percentage change from baseline in total IgG over time stratified by treatment group, RLZ total and Baseline bodyweight group (<50kg, 50kg-<70 kg, 70-<100kg, ≥100kg) where the Baseline bodyweight group is multipaneled or overlaying with different colors within each treatment group.

For correlation analysis between clinical endpoints and PD data, scatterplots including regression lines and correlation coefficients will be provided for:

- Maximum change from baseline through to and including day 43 in total IgG versus change from baseline at day 43 in MG-ADL, QMG, and MG-C scores;
- Maximum percent change from baseline through to and including day 43 in total IgG versus change from baseline to day 43 in MG-ADL, QMG, and MG-C scores;
- Minimum total IgG through to and including day 43 versus change from baseline to day 43 in MG-ADL, QMG, and MG-C scores.

A boxplot of maximum percentage change from Baseline for total IgG will also be plotted by the following dose groups: placebo,

Serum concentration of change from Baseline in total IgG and IgG subclass will be listed together with concentrations of rozanolixizumab , ADA status and MG-ADL change from Baseline, as specified in Section 9.3.2. In addition, it will be listed with IgG subclasses and MG-specific autoantibodies as described in Section 9.2.1.

## 9.3 Anti-drug antibody status

Evaluation of rozanolixizumab immunogenicity will be performed using data from all evaluable study participants in the SS, defined as all study participants treated with rozanolixizumab who have an evaluable pretreatment (baseline) sample (negative or positive ADA sample status), and at least 1 evaluable post-baseline value.

Study participants with an evaluable pretreatment (baseline) sample but without a single evaluable sample taken post-baseline will be included in the reporting of pre-existing ADA but excluded from all other immunogenicity analyses.

The ADA of rozanolixizumab will be measured using a three-tiered assay approach: screening assay, confirmatory assay and titration assay. Any sample confirmed positive for ADA will be assayed to determine whether there is neutralizing potential. Samples that are neutralizing antibody (NAb) positive will be evaluated in a titration assay to quantify the NAb level and will be reported as titer. Samples from study participants on placebo will not be tested for anti-drug antibodies.

#### 9.3.1 ADA Data Consideration

#### **ADA Sample Status**

The ADA sample status will be determined for each pre-treatment (Baseline) and post-treatment (post-Baseline) visit where samples are taken for ADA analysis.

- Sample values that are either 'negative screen' or the combination of 'positive screen' and 'negative immunodepletion' will be defined as **ADA negative** if corresponding rozanolixizumab concentrations are equal or below the validated drug tolerance limit of the ADA assay (200µg/mL rozanolixizumab) allowing detection of 100ng/mL ADA
- Sample values that are either 'negative screen' or the combination of 'positive screen' and 'negative immune-depletion', but with corresponding rozanolixizumab concentrations above the validated drug tolerance limit of the ADA assay, will be defined as **ADA inconclusive**
- Sample values that are 'positive screen' and 'positive immunodepletion' will be defined as **ADA positive**
- Samples that could not be tested for ADA status due to inadequate sample volume, mishandling, or errors in sample collection, processing, storage, etc., will be defined as Missing.

NAb sample status (positive/negative/missing) will be determined for ADA positive samples.

#### ADA Baseline

By default, the Day 1 will be the Baseline value if the ADA sample status at screening is ADA negative or missing. If the ADA sample status at screening is ADA positive and ADA status at Day 1 is ADA negative or missing, the screening will be the Baseline value. If the ADA sample status at screening and Day 1 are the same, Day 1 will be the Baseline value.

#### ADA /NAb Participant Status

The ADA participant status will be classified on study participant and group level as outlined below (Shankar et al. 2014; Rup et al, 2015). A description of how study participants will be categorized for the immunogenicity assessment is provided in Table 9–1.

Individual study participants will be assessed for ADA participant status, composed of 6 categories: ADA negative, inconclusive, and ADA positive, whereby a positive participant's status is determined as originating from a treatment-induced, boosted, reduced or unaffected ADA response.

Study participants who are identified as being treatment-induced or treatment-boosted ADApositive will be grouped as treatment-emergent (TE)-ADA positive participants. Study participants who are identified as being treatment-reduced or treatment-unaffected ADA-positive will be grouped as non-TE-ADA positive participants. Both TE-ADA positive and non-TE-ADA positive participants will be further classified as NAb negative or NAb positive.

The individual and combined ADA participant categories will be summarized through the end of the 8-week observation week (Day 99), unless specified otherwise.

Terms and Definitions for ADA Evaluation in Study Participants Table 9–1:

| Classification | Classification Label | Definition |
|---|---|---|
| Individual par | ticipant categories | |
| 1 | Pre-ADA negative – treatment induced ADA negative (ADA-NEG) | Study participants who have an ADA negative sample at Baseline and all sampling points post-Baseline up to the timepoint of interest. |
| 2 | Inconclusive | Study participants who have an ADA positive or negative Baseline sample and some post-Baseline samples are missing or inconclusive, while other post-Baseline samples are ADA negative up to the timepoint of interest. |
| 3 | Pre-ADA negative – treatment induced ADA positive (TI-POS) | Study participants who have an ADA negative sample at Baseline and have least one ADA positive sample at any sampling point post-Baseline up to the timepoint of interest. |
| 4 | Pre-ADA positive – treatment boosted ADA positive (TB-POS) | Study participants who have an ADA positive sample at Baseline and at least one ADA positive sample at any sampling point post-Baseline up to the timepoint of interest, with increased titer values compared to Baseline (greater than a predefined fold difference increase from Baseline value which will be defined within the validation of the assay i.e. MSR of the assay <sup>a</sup> ). |
| 5 | Pre-ADA positive – treatment<br>reduced ADA positive (TR-<br>POS)<br>Pre-ADA positive – treatment | Study participants with an ADA positive sample at Baseline, and ADA negative samples at all sampling points post-Baseline up to the timepoint of interest. Study participants with an ADA positive at Baseline |
| | unaffected ADA positive (TU-POS) | and an ADA positive sample at any sampling point post-Baseline up to timepoint of interest with titer values of the same magnitude as Baseline (less than a predefined fold difference from the Baseline value which will be defined within the validation of the assay, i.e. MSR of the assay <sup>a</sup> ). |
| Combined par | ticipant categories | |


| 7 | Treatment emergent ADA | Includes study participants who are treatment |
|---|---|---|
| | positive (TE-POS) | induced ADA positive (category 3) or treatment |
| | | boosted ADA positive (category 4). |
| 8 | Non-treatment emergent ADA | Includes study participants who are treatment |
| | positive (Non-TE-POS) | reduced ADA positive (category 5) or treatment |
| | | unaffected ADA positive (category 6). |
| 9 | Treatment emergent ADA | Includes study participants who are treatment |
| | positive – NAb positive (TE- | emergent positive (category 7) and have at least one |
| | POS, Nab-POS) | NAb positive sample |
| 10 | Treatment emergent ADA | Includes study participants who are treatment |
| | positive – NAb negative (TE- | emergent positive (category 7) and have no NAb |
| | POS, Nab-NEG) | positive samples |
| 11 | Non-treatment emergent ADA | Includes study participants who are non-treatment |
| | positive NAb positive (Non- | emergent positive (category 8) and have at least one |
| | TE-POS, NAb-POS) | NAb positive sample |
| 12 | Non-treatment emergent ADA | Includes study participants who are non-treatment |
| | positive NAb negative | emergent positive (category 8) and have no NAb |
| | (Non-TE-POS, NAb-NEG) | positive samples |

<sup>&</sup>lt;sup>a</sup> The fold difference increase from baseline value, i.e. the minimum significant ratio (MSR) determined during assay validation, will be reported in the relevant tables, listings and figures. It reflects the fold difference in titer level that considered higher than the assay variation in titer determination

#### 9.3.2 ADA summaries

The following outputs will be presented on the SS

#### Tables:

- Number and percentage of study participants with positive, negative, inconclusive or missing ADA sample status at the time of each visit will be summarized by treatment group and RLZ total. Denominator is the number of study participants having a non-missing result at that visit. The same table will be repeated for NAb sample status (positive, negative, missing).
- Number and percentage of study participants in each of the individual and combined ADA
  participant status categories presented in will be
  summarized by treatment group and RLZ total.
- Total prevalence of pre-existing ADA and NAb, defined as number and percentage of participants having an ADA positive sample status at baseline, with the denominator being the total number of study participants having an evaluable sample result at Baseline. Missing samples will not be included in the denominator. The same will be repeated for NAb.
- The first occurrence of treatment-emergent ADA positivity: cumulative number and percentage of TE-ADA positive participants (category 7) who are ADA positive for the first time at each visit.
- Summary table of mean maximum percentage CFB in total IgG and mean CFB in MG-ADL total score at Day 43, summarized by ADA participant categories 1, 2, 9, 10, 11 and 12 for the corresponding time period of interest (up to Day 43) and by treatment group and RLZ total.

- Overall summary table of TEAEs within each of the ADA participant categories 1, 2, 7 and 8.
- Summary table of incidence of TEAEs by ADA participant category 1, 2, 7 and 8.
- Summary table of AEOF hypersensitivity reactions, anaphylactic reactions and infusion reactions by ADA participant category 1, 2, 7 and 8.

#### Figures:

- Individual time course plots for study participants with at least one ADA positive sample, representing ADA and NAb titers (on log-scale), rozanolixizumab plasma concentrations, percentage CFB for total IgG and MG-specific autoantibodies, and CFB for MG-ADL total score. The sub-title of the graph will include the study participant number, bodyweight category, treatment group, ADA participant category (2, 3,4,5,6). The dosing will be represented in the x axis with bars/arrows at the time of dose.
- Spaghetti plots of individual time course of ADA titer for ADA positive participants in categories 9, 10, 11 and 12, whereby all categories are overlaid on the same plot and visualized using different symbols and colors. The ADA titer results will be presented on a log-scale. Dosing time points should be indicated below the x-axis. The same plot will be repeated for NAb titer for NAb positive participants in categories 9 and 11.
- A box-and-whisker plot of maximum post-dose ADA titer (on log-scale) through the end of the observation period versus ADA participant category for categories 9, 10, 11 and 12. The same plot will be repeated for NAb titer for ADA participant categories 9 and 11.
- Scatter dot plot of individual rozanolixizumab post-dose plasma concentrations categorized by Day (i.e. Days 3, 6, 24, 38, 41) and for each Day by ADA participant categories 1, 2, 9, 10, 11 and 12. Individual samples that tested positive for ADA will be visualized using a symbol and/or color.
- Time course plot of mean change from Baseline in MG-ADL total, summarized by ADA participant category 1, 2, 7, and 8. Categories will be determined for the time period from baseline up to Day 43. Separate plots for each treatment group and RLZ total. The sample plot will be repeated for NAb related categories 9, 10, 11, 12.
- Spaghetti plots of individual time course of percentage CFB for total IgG, for each of the ADA participant categories 1, 2, 9, 10, 11 and 12, whereby the ADA participant categories are multipaneled. Separate plots for each treatment group and RLZ total (combined). Individual samples that tested positive for ADA will be visualized using a symbol and/or color. Dosing time points should be indicated below the x-axis.
- Scatter dot plot of individual CFB in MG-ADL total score categorized by ADA titer tertile (including category ADA not present) over time. The same plot will be repeated for NAb titer.
- Scatter dot plot of individual percentage CFB for total IgG categorized by ADA titer tertile (including category ADA not present) over time. The same plot will be repeated for NAb titer.

#### Listings:

- By-subject listing by treatment group, individual ADA participant category, screening and confirmatory assay results, ADA titer, fold change compared to baseline, and whether or not sample contains RLZ concentration above drug tolerance. In addition, the time since administration of IMP will be reported (in days).
- By-subject listing by treatment group, administered RLZ dose and timepoint, of ADA and NAb sample status, ADA titer, NAb titer, rozanolixizumab plasma concentration, CFB for total IgG, CFB for MG-specific autoantibodies, CFB for MG-ADL total score, QMG and MG-C, and individual ADA participant classifications. In addition, the time since administration of IMP will be reported (in days).
- By-subject listing of abovementioned TEAEs, the time of onset, the ADA and NAb sample status and ADA and NAb titers at the closest sampling time point prior to and subsequent to the TEAE, and time since last administration of IMP (in days).

#### 9.4 Immunology

All analyses described in this section will be based on the SS.

#### 9.4.1 Serum complement levels and plasma complement levels

Serum (C3 and C4) and plasma (C3a and C5a) complement variables will be listed by treatment group and RLZ total, visit and time point including changes from Baseline. Descriptive summaries will be presented for both absolute values and changes from Baseline for all study participants, and separately for study participants who experience an infusion reaction or hypersensitivity reaction or anaphylactic reaction. The selection criteria of infusion reaction or hypersensitivity reaction are described in Section 13.8.

Measurements BLQ will be imputed with half of the LLOQ for the purpose of calculating change from Baseline. Measurements above the limit of quantification (ALQ), if applicable, will be imputed to the upper limit of quantification.

Serum (C3 and C4) and plasma (C3a and C5a) complements results will be listed.

#### 9.4.2 Serum cytokines

Serum cytokines will be summarized by treatment group and RLZ total, visit and time point for both absolute values and changes from Baseline, for all study participants, and separately for study participants experiencing with serious or severe headache and/or infusion reactions or hypersensitivity reaction. The selection criteria of those events are described in Section 13.8.

Measurements BLQ will be imputed with half of the LLOQ for the purpose of calculating change from Baseline. Measurements ALQ, if applicable, will be imputed to the upper limit of quantification.

Cytokines results will be listed.

#### 9.4.3 Serum immunoglobulin concentrations

Immunoglobulins (IgE, IgA and IgM) will be summarized by treatment group, RLZ total and visit for absolute values, change from Baseline, and percent change from Baseline.

Individual figures over time (absolute value) will be presented by study participant, with all variables overlaid on the same plot and separate plots each study participant.

Measurements BLQ will be imputed with half of the LLOQ for the purpose of calculating change from Baseline. Measurements ALQ, if applicable, will be imputed to the upper limit of quantification.

Immunoglobulins (IgE, IgA, and IgM) will be listed.

#### 9.4.4 Anti-tetanus toxoid serum titers

Anti-tetanus toxoid serum titers will be summarized by treatment group, RLZ total and visit for both absolute values, change from Baseline, and percent change from Baseline.

The geometric mean change from Baseline with 95% CL in anti-tetanus toxoid serum titers.

The geometric mean change from Baseline with 95% CI in anti-tetanus toxoid serum titers versus time at each scheduled timepoint will be plotted by treatment group excluding all participants with undetectable Baseline titers. IgG values will be overlaid on the same plot.

Measurements BLQ will be imputed with half of the LLOQ for the purpose of calculating change from Baseline. Measurements, if applicable, will be imputed to the upper limit of quantification.

Anti-tetanus toxoid serum titers will be listed.

#### 10 SAFETY ANALYSES

All safety analyses will be presented using the SS. Listings will be presented by treatment group and study participant; tabulations will be presented by treatment group and RLZ total.

Unless otherwise specified, safety analyses will be presented by treatment group as defined in Section 3.6.

#### 10.1 Extent of exposure

The number of weeks on IMP will be summarized by treatment group and RLZ total. The number of days on IMP will be calculated as follows:

Number of weeks on IMP = 
$$\frac{[(Date \text{ of Last Dose Received}) - (Date \text{ of First Dose Received}) + 1]}{7}$$

The total number of infusions will be summarized using descriptive statistics by treatment group and RLZ total. Categorical summaries of the number of infusions (1-6) will also be summarized.

The summaries above will be repeated excluding the mock infusions.

All drug administration details will be listed.

#### 10.2 Adverse events

#### 10.2.1 Data considerations

Adverse events will be recorded from the time of informed consent until study completion. All AEs will be coded (Section 3.8).

In addition, AEs will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5 or later for severity. For any AEs where it is not possible to provide a CTCAE grading, the events will be assessed using a standard intensity classification (mild,


moderate and severe). For the purpose of the tabulations all CTCAE severity classifications will be mapped to a mild/moderate/severe grade as described below:

- Grade 1-- Mild

These will be tabulated together with the AEs that were not classified according to CTCAE criteria i.e., all Grade 1 AEs as per CTCAE criteria will be included in the 'mild' cottogether with those AEs classified as mild as per the 'criteria and 'criteria and case a mapped standard intensity classification per above rule is different from the standard. intensity classification on CRF, the worst case will be used as the standard intensity classification (i.e. an AE with Grade 1 and moderate as intensity classification will be classified into moderate).

A TEAE is defined as an AE starting on or after the time of first administration of IMP up to and including 8 weeks (56 days) after the final dose. Adverse events starting before the date of the first administration of IMP or after 8 weeks following the final dose of IMP will not be considered TEAEs. Thus AEs before first dosing and AEs after 8 weeks following the final dose will be combined in one category. Such events will be listed only.

Where dates are missing or partially missing. AEs will be assumed to be treatment-emergent unless evidence exists that does not allow the AE to be treatment-emergent. Handling of missing dates for classification of AEs as TEAEs is described in Section 4.2.2.

The following rules will be used to assign a TEAE to a study period:

- **Treatment Period:** a TEAE will be assigned to the Treatment Period for the tabulations if the start date of the event is on or after the date of the first administration of IMP on Day 1, up to 7 days following the final dose of IMP
- **Observation Period:** a TEAE will be assigned to the Observation Period for the tabulations if the start date of the event is greater than 7 days after the date of the final dose of IMP until 8 weeks following the final dose; events starting later than 8 weeks following the final dose of IMP are not considered TEAEs

In the case of early withdrawal in the Treatment Period, a TEAE will be assigned to the Treatment Period based on the last received IMP plus 168 hours (7 days). Subsequent TEAEs (up to 8 weeks post-last dose) will be assigned to the Observation Period.

A TEAE will be counted as a TEAE related to IMP if the response to the question "Relationship to Study Medication" is "Related". Severe TEAEs are those with CTCAE Grade 3 or above, or those without a CTCAE grading classified as 'severe' by the Investigator.

Es will be presented as "number of study participants (percentage of study participants) [number of events]". In this style of output, "[number of events]" will include all cases of an AE including repeat occurrences in individual study participants, while "number of study participants" will count each study participant only once.

#### 10.2.2 AE summaries

Summary tables with the number, percentage of study participants and frequency of TEAEs will be provided by treatment group and RLZ total. Additional details are as follows:

- 1. Overview of TEAEs will include following categories: any TEAEs, serious TEAEs, Any TEAEs by relationship

  Any TEAEs relative to ADA status

  Any TEAE by Risk Difference ≥5% (by decreasing frequency

  Non-serious TEAEs above reporting threshold

  Patal TEAEs

  atal TEAEs

  atal TEAEs participant discontinuation due to TEAEs, permanent withdrawal of IMP due to TEAEs, temporary withdrawal of IMP due to TEAEs, treatment-related TEAEs, severe TEAEs, TEAEs leading to death, all deaths (AEs leading to death).
- 2. Incidence of TEAEs will be summarized by SOC, HLT and PT for:
  - Any TEAEs

  - Any TEAEs by relationship
  - Any TEAEs relative to ADA status
  - Any TEAE by Risk Difference ≥5% (by decreasing frequency of Risk Difference)
  - Non-serious TEAEs above reporting threshold of 5% of study participants

  - Fatal TEAEs by relationship
  - Serious TEAEs
  - Serious TEAEs by relationship
  - Participant discontinuation due to TEAEs
  - TEAEs leading to permanent withdrawal of IMP
  - TEAEs leading to temporary withdrawal of IMP
  - Treatment-emergent AESM
  - Treatment-emergent AESI
- 3. Incidence of TEAEs will be summarized by PT for:
  - Any TEAEs by decreasing frequency of PT

AESMs include severe headache, severe GI disorders (i.e., abdominal pain, diarrhea, vomiting), and opportunistic infection.

AESIs are the cases of potential Hy's Law (see Section 10.3.1).

AESMs and AESIs will be identified based on the assessment by the Investigator as recorded in the CRF. An AE will be counted as an AESM if there is a 'yes' response to the question "Adverse event of Special Monitoring?" and 'no' otherwise. An AE will be counted as an AESI if there is a 'yes' response to the question "Adverse Event of Special Interest?" and 'no' otherwise.

When applicable adverse event summaries will be ordered by alphabetical SOC, alphabetical HLT within SOC and decreasing frequency of PT in the rozanolixizumab total column for tables.

Listings of all TEAEs, all non-serious TEAEs, serious TEAEs, permanent withdrawal of IMP due to AEs, study participant discontinuation from study due to AEs, AEs leading to death, AESIs, AESMs will be presented by treatment group and study participants.

#### 10.2.3 **Adverse Events of Focus**

Rozanolixizumab treatment-emergent adverse events of Focus (TEAEOF) include the following categories:

reaction

Juston reaction

Opportunistic infections

Reductions in albumin and plasma proteins

Effects on the kidney

Drug related hepatic disorders
subject listing of all treatment-emergented. The number and percentage of the number and percentage of treatment grown the treatment grown reatment grown. A by-subject listing of all treatment-emergent AEOF by category (as listed above) will be provided. The number and percentage of study participants who experience each treatmentemergent AEOF will be summarized by most recent dose level prior to onset of AEOFs and total Rozimab treatment group. The following summaries will be presented by SOC, HLT, and PT:

- Treatment-emergent AEOF
- Serious Treatment-emergent AEOFs
- Treatment-emergent AEOFs by relationship
- Treatment-emergent AEOFs by maximum intensity (mild, moderate and severe)
  - Treatment-emergent AEOF hypersensitivity reactions, anaphylactic reactions and infusion reactions by ADA
- Treatment-emergent AEOF headache and GI disturbances in Treatment period by intensity
- Treatment-emergent AEOFs by Risk Difference (by decreasing frequency of Risk Difference)

Graphs for treatment-emergent AEOF headache by time of onset (relative to infusion), severity, causality and duration for each study participant will also be provided.

#### 10.2.4 Safety analysis by weight subgroup and administered dose

To support the goal of a fixed dosing strategy for Rozanolixizumab, additional summary tables with the number, percentage of study participants and frequency of TEAEs (when applicable) will be provided by weight subgroup and administered dose and by SOC, HLT and PT for:

- Overview of TEAEs
- Incidence of TEAEs
- Incidence of Serious TEAEs
- Incidence of Severe TEAEs
- Incidence of AEOF of headache and GI disturbances
- Incidence of AEOF of headache and GI disturbances by maximum intensity (mild, moderate and severe)

### 10.3 Clinical laboratory evaluations

The following table (Table 10-1) lists safety laboratory assessments that are collected throughout the study:

Table 10-1: Clinical Laboratory Parameters

| Laboratory<br>Assessments | Parameters | | | | |
|---|---|---|---|---|---|
| Hematology | Platelet Count Red Blood Cell (RBC) Count Hemoglobin Hematocrit | | RBC Indices: Mean corpuscular volume Mean corpuscular hemoglobin %Reticulocytes | | WBC Count with Differential: Neutrophils Lymphocytes Monocytes Eosinophils Basophils |
| Clinical Chemistry | Blood Urea<br>Nitrogen<br>(BUN) | Potassi | um | Aspartate Aminotransferase (AST)/Serum Glutamic- Oxaloacetic Transaminase (SGOT) | Total and direct bilirubin |
| | Creatinine<br>Estimated<br>Glomerular | Sodiun | n | Alanine<br>Aminotransferase<br>(ALT)/ Serum<br>Glutamic-Pyruvic | Total Protein Albumin |

| Laboratory<br>Assessments | Parameters | | | |
|---|---|---|---|---|
| | Filtration Rate (eGFR) <sup>a</sup> | | Transaminase (SGPT) | |
| | Glucose<br>(fasting state,<br>preferred) | Calcium <sup>b</sup> | Alkaline<br>phosphatase | C-reactive protein (CRP) |
| | Lactate<br>dehydrogenase<br>(LDH) | High-<br>density<br>lipoprotein<br>(HDL) <sup>c</sup> | Total Cholesterol (TC) | Triglycerides (TRIG) |
| Routine Urinalysis | <ul> <li>Specific gravity</li> <li>Albumin, albumin/creatinine, creatinine</li> <li>pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase, hemoglobin by dipstick</li> <li>Microscopic examination (if blood or protein is abnormal)</li> </ul> | | | |
| Other Screening Tests | <ul> <li>Serum or urine human chorionic gonadotropin (hCG) pregnancy test (as needed for women of childbearing potential)<sup>d</sup></li> <li>PTT, INR, and HbA1c tests</li> <li>Serology testing (for Hepatitis B, Hepatitis C, and HIV) All study-required laboratory assessments will be performed by a central laboratory.</li> <li>The results of each test must be entered into the CRF.</li> </ul> | | | |

#### NOTES:

All study-required laboratory assessments will be performed by a central laboratory.

The results of each test must be entered into the CRF.

<sup>&</sup>lt;sup>a</sup> eGFR is calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula which is eGFR =  $141 * min(Scr/κ,1)\alpha * max(Scr/κ,1)^{-1.209} * 0.993^{Age} * 1.018$  [if female] \* 1.159 [if black]; where Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1. If race is not captured, participant will be assumed not Black in the calculation.

<sup>&</sup>lt;sup>b</sup> Corrected Calcium (mmol/L) =0.02 \* (40 – Albumin (g/L)) + Calcium (mmol/L).

<sup>&</sup>lt;sup>c</sup> Calculation of Low-density lipoprotein (LDL) will follow Friedewald equation, where LDL in mmol/L= TC - HDL - TRIG/2.22; LDL in mg/dL= LDL=TC-HDL-TRIG/5 (if all values are in mg/dL). This formula is applicable only if Triglycerides is less than or equal to 400 mg/dL (4.52 mmol/L).

<sup>&</sup>lt;sup>d</sup> Local urine testing will be standard for the protocol unless serum testing is required by local regulation or Institutional Review Board (IRB)/ Independent Ethics Committee (IEC).
Chemistry, hematology and quantitative urinalysis (observed value, absolute change from Baseline) will be summarized in standard unit using descriptive statistics by treatment group and RLZ total at each scheduled visit.

The central data will be used for the summary tables. Measurements BLQ will be imputed with half of the lower limit of quantification LLOQ, and measurements ALQ will be imputed to the upper quantification limit for the purpose of quantitative summaries.

The number and percentage of study participants who meet each of the markedly abnormal (MA) criteria outlined in Section 13.7 will be summarized by treatment group at any visit (including unscheduled visit).

The laboratory variables that are categorized as normal, high or low based on the reference range supplied by the analytical laboratory will be presented in shift tables from Baseline to any post-Baseline visit (including unscheduled visit) by treatment group.

Mean values in albumin, C-reactive protein and White Blood Cell Count with absolute count and differential (neutrophils, lymphocytes, monocytes, eosinophils and basophils) plotted over time by treatment, RLZ total with all treatments overlaid on the same plot. Lipids including Highdensity Lipoprotein, Low-density lipoprotein, Total Cholesterol, Triglycerides will be plotted the same way if data are available.

All laboratory test results will be listed, including Baseline, scheduled and unscheduled visits with results in standard unit. Values outside the reference range for the continuous variables will be flagged in the listings. The reference ranges will also be reported in the listings. In addition, the listings will include a flag for values identified as MA. Additional lab test, including pregnancy testing, will also be listed.

### 10.3.1 Potential drug-induced liver injury

The number and percentage of study participants who meet one or more of the following potential drug-induced liver injury (pDILI) criteria will be summarized by treatment group and RLZ total:

- Participants with at least one post-Baseline liver laboratory assessment
- Incidence of potential hepatotoxicity with symptoms potentially associated with hepatitis or hypersensitivity
- Incidence of potential hepatotoxicity with no symptoms potentially associated with hepatitis
  or hypersensitivity
- Laboratory criteria for pDILI:
  - (AST or ALT > 3 x ULN) and TBL > 1.5 x ULN
  - (AST or ALT > 3 x ULN) and TBL > 2 x ULN
  - (AST or ALT  $\geq$  3 x ULN) and TBL  $\geq$  2 x ULN and ALP  $\leq$  2 x ULN (Hy's Law)

In order to meet the above criteria, a study participant must experience the elevation in bilirubin and ALT or AST (and the absence of the ALP elevation) at the same visit. For example, a study participant who experiences a > 2x ULN elevation of bilirubin at one visit and a> 3x ULN

elevation in ALT (or AST) at a subsequent visit has not fulfilled the Hy's law criteria. If participant meets part of one criterion but at least one parameter is unknown, then he/she should not be considered for meeting the criterion.

Additional analyses for liver function tests (LFTs) will be performed to assess the potential for liver toxicities in accordance with the United States Food and Drug Administration guidelines. Per guidelines, the following criteria will be used to define levels of LFT elevation:

- Aspartate aminotransferase (AST): >3 x ULN, >5 x ULN, >8 x ULN, >10 x ULN, >20 x ULN
- Alanine aminotransferase (ALT): >3 x ULN, >5 x ULN, >8 x ULN, >10 x ULN, >20 x ULN
- AST or ALT: >3 x ULN, >5 x ULN, >8 x ULN, >10 x ULN, >20 x ULN
- Total bilirubin (TBL): >1.5 x ULN, >2 x ULN
- Alkaline phosphatase (ALP) >1.5 x ULN

A listing will also be provided for study participants who meet at least one of the above criteria. All results obtained at that visit for the specified parameters will be displayed.

# 10.4 Vital signs, physical findings, and other observations related to safety

### 10.4.1 Vital signs

Observed values and changes from Baseline will be summarized by vital signs variables (pulse rate, systolic and diastolic blood pressure, and temperature) and timepoint by treatment group.

The number and percentage of study participants who meet each of the MA criteria outlined in Section 13.7 will be summarized by treatment group and RLZ total at any visit (including unscheduled visit).

A by-participant listing of all vital sign measurements and change from Baseline will be presented by treatment group and timepoint. The listing will include a flag for values identified as MA.

Repeated and unscheduled measurements will be handled as described in Section 4.2.3.

## 10.4.2 Electrocardiograms

The following variables will be reported:

- Heart rate
- PR interval
- RR interval
- QRS duration
- OT interval
- QT corrected for heart rate using Fridericia's formula (QTcF =  $QT/RR^{1/3}$ )

Observed values and changes from Baseline will be summarized by treatment group and RLZ total at scheduled visit and by ECG variable. The number and percentage of study participants

with normal, abnormal not clinically significant and abnormal clinically significant ECG results will be provided in a shift table from Baseline to worst post-Baseline interpretation during the study.

For the ECG data, all calculations of changes from Baseline and descriptive statistics will be based on the mean of the triplicate assessments at each timepoint. In the event that there are not 3 available measurements at a given timepoint, the mean will be calculated based on the number of measurements for which data are provided.

The number and percentage of study participants who meet each of the MA criteria outlined in Section 13.6 will be summarized by treatment group at any visit (including unscheduled visit).

A listing of electrocardiogram data will be presented, including repeated and unscheduled measurements.

## 10.4.3 Other safety endpoints

## 10.4.3.1 Physical examination

Results of physical examination abnormalities will be listed.

## 10.4.3.2 Suicidal risk monitoring

The C-SSRS include: (i) suicidal ideation, (iii) suicidal behavior, (iii) suicidal ideation or behavior, and (iv) self-injurious behavior without suicidal intent.

Suicidal ideation is defined as an event in any of the following 5 categories:

Suicidal behavior is defined as an event in any of the following 5 categories:

•

Suicidal behavior or ideation is defined as an event in any of the above 10 categories.

Self-injurious behavior without suicidal intent is corresponding to the response to "Has subject engaged in Non-Suicidal Self-Injurious Behavior?" in questionnaire.

A by-participant listing of the C-SSRS questionnaire data will be provided by treatment group.

## 10.4.3.3 Assessment and management of Tuberculosis (TB)

By-participant listings of interferon gamma release assay (IGRA) TB test, chest X-ray and TB signs and symptoms questionnaire for TB will be provided.

### 11 OTHER ANALYSES

# 11.1 Specific analyses for Pharmaceuticals and Medical Devices Agency (PMDA)

The following endpoints will be summarized for study participants in Japan only:

- Study participant characteristics (as specified in Section 5)
- Demographics and other Baseline characteristics (as specified in Section 6)
- Primary efficacy endpoint (as specified in Section 8.2.2)
  - Change from Baseline in MG-ADL to Day 43 (Visit 10)
- Secondary efficacy endpoints (as mentioned in Section 8.3):
  - MG-ADL responder (≥2.0 points improvement from Baseline) at Day 43 (Visit 10)
  - Change from Baseline to Day 43 (Visit 10) in MG-C score
  - Change from Baseline to Day 43 (Visit 10) in QMG score
- Other efficacy endpoints (as mentioned in Section 8.4):
  - Use of rescue therapy due to worsening (IVIg, PEX)
  - Change from Baseline in MG-ADL at each scheduled assessment during Treatment and Observation Periods
    - In addition to the overall summary, the MG-ADL scores and change from Baseline will be summarized by the subgroup (MuSK+ or AChR+).
  - MG-ADL responder (≥2.0 points improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
  - Change from Baseline in QMG at each scheduled assessment during Treatment and Observation Periods
  - QMG responder (≥3.0 points improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
  - Change from Baseline in MG-C score at each scheduled assessment during Treatment and Observation Periods
  - MG-C responder (≥3 .0 points improvement from Baseline) at each scheduled assessment during Treatment and Observation Periods
  - Change from Baseline in MG-QOL15r at each scheduled assessment during Treatment and Observation Periods
- ADA summaries (as mentioned in Section 9.3.2):

- Number and percentage of study participants with positive, negative or missing ADA status at the time of each visit and overall will be summarized by treatment group and RLZ total.
- Number and percentage of study participants in each of the ADA classifications will be summarized by treatment group and RLZ total.
- Number and percentage of study participants with first occurrence of treatment-emergent ADA positive at each visit will be summarized by treatment group and RLZ total.
- The cumulative number of study participants with treatment-emergent ADA positive will also be presented.
- The time to achieving treatment-emergent ADA positive, separated by treatment group and ADA category, will be analyzed based on Kaplan-Meier methods.
- The incidence of NAb, defined as (cumulative) proportion of study participants having NAb positive samples at any point up to and including that time point will be summarized by treatment group and RLZ total. Missing samples will not be included in the denominator. This will be also plotted graphically overlaying the treatment groups.
- A summary table of all immune related TEAEs by ADA status will be presented by treatment group. For this summary, study participants will be presented for TEAEs occurring prior to becoming treatment emergent ADA positive, TEAEs occurring after becoming TE ADA positive, and TEAEs for study participants who remained TE ADA negative.

## Safety endpoints

The number, percentage of study participants and frequency of TEAEs will be summarized by treatment group and RLZ total. Additional details are as follows:

- An TEAE overview table will be provided, include following categories: any TEAEs, serious TEAEs, participant discontinuation due to TEAEs, permanent withdrawal of IMP due to TEAEs, temporary withdrawal of IMP due to TEAEs, treatment-related TEAEs, severe TEAEs, TEAEs leading to death, all deaths (AEs leading to death).
- Incidence of TEAE will be summarized by SOC, HLT, and PT for:
  - Any TEAEs
  - Severe TEAEs
  - Any TEAEs by maximum intensity (mild, moderate and severe)
  - Any TEAEs by relationship
  - Fatal TEAEs
  - Serious TEAEs
  - Serious TEAEs by relationship
  - Participant discontinuation due to TEAEs
  - TEAEs leading to permanent withdrawal of IMP

10 Nov 2021 MG0003

ay participant ay participant and a property of the participant and a participan


## 12 REFERENCES

Burns, Ted M et al. "The MG Composite: A valid and reliable outcome measure for myasthenia gravis." *Neurology* vol. 74,18 (2010): 1434-40. doi:10.1212/WNL.0b013e3181dc1b1e

Wassmer G and Brannath W. (2016) Group Sequential and Confirmatory Adaptive Designs in Clinical Trials. DOI 10.1007/978-3-319-32562-0

Hedges, Larry V., and Ingram Olkin. Statistical methods for meta-analysis. 1985; 10.2307/116953.

Lehmacher W and Wassmer G. Adaptive Sample Size Calculations in Group Sequential Trials. Biometrics. 1999;55:1286-90.

Yuan, Y. Sensitivity Analysis in Multiple Imputation for Missing Data. Paper SAS270-2014. SAS Institute (2014).

Levey et al. A New Equation to Estimate Glomerular Filtration Rate. Ann Intern Med. 2009; 150: 604-612.

Nehring, S.M.; Goyal, A.; Patel, B.C. (2020). StatPearls Publishing, web link: <a href="https://www.ncbi.nlm.nih.gov/books/NBK441843/">https://www.ncbi.nlm.nih.gov/books/NBK441843/</a>.

Permutt T and Li F. Trimmed Means for Symptom Trials with Dropouts. Pharmaceutical Statistics. 2017; 16: 20-28.

Vissing, J., Jacob, S., Fujita, K. P., O'Brien, F., & Howard, J. F. (2020). 'Minimal symptom expression' in patients with acetylcholine receptor antibody-positive refractory generalized myasthenia gravis treated with eculizumab. *Journal of neurology*, 1-11.

United States Department of Health and Human Services, National Cancer Institute. Common Terminology for Adverse Events (CTCAE), Version 5.0, November 17, 2017.

## 13 APPENDICES

### 13.1 QMG Scale

The QMG scale comprises 13 items, including ocular and facial movement, swallowing, speech, limb strength and forced vital capacity. Scoring for each item ranges from no weakness (0) to severe weakness (3), with an overall score range from 0 to 39, i.e., a higher score indicates more severe disease. A 3-point change in the overall score is considered to be clinically relevant.

The QMG testing form is provided in Table 13–1. The total score is obtained by summing the responses to each individual item.

The score ranges from 0 to 33.

In the event of missing data, the following rules will be applied:

- If 1 or 2 items are not answered, the overall score will be obtained by imputing the missing items with the average score across the remaining items at the specific visit. The imputed value will be rounded to one decimal place
- If more than 2 items are missing the overall score will not be calculated at the specific visit

Table 13-1: Quantitative myasthenia gravis testing form





## 13.2 MG-C score

**UCB** 

The MG-C score items and associated scores are provided in Table 13-2.

The MG-C score comprises 10 items, each of which is weighted differently in the calculation of the overall score. The overall score ranges from 0 to 50, with a higher score indicating more severe disease.

The total score is obtained by summing the responses to each individual item.



In the event of missing data at a particular timepoint, the MG-C score will not be calculated. Due to the different weighting applied to each item it is not possible to impute the missing data with the average score across the remaining items.

Table 13-2: MG-C score items and scoring algorithm





<sup>&</sup>lt;sup>a</sup> Moderate weakness for head and neck items should be construed as weakness that equals roughly 50%+/-15% of expected normal strength. Any weakness milder than that would be mild and any weakness more severe than that would be classified as severe.

#### **MG-Activities of Daily Living** 13.3

The MG-ADL score comprises 8 items, each with a score of 0 to 3. The total score is obtained by summing the responses to each individual item. Thus, the score ranges from 0 to 24 with a higher score indicating more disability. The MG-ADL testing form is provided in Table 13–3.

In the event of missing data, the following rules will be applied:

- If 1 or 2 items are not answered, the overall score will be obtained by imputing the missing items with the average score across the remaining items at the specific visit. The imputed If more than 2 items are missing the overall score will not be calculated. value will be rounded to one decimal place.

10 Nov 2021 MG0003

Table 13–3: MG-Activities of Daily Living



## 13.4 MG Symptoms PRO

The MG Symptoms PRO includes two steps: 1) rescoring the item responses; and 2) calculation of the final scores. Details of the scoring is found in the Myasthenia Gravis Symptoms PRO Instrument Scoring Manual date 28 February 2019.

Step 1: Rescoring the item responses. The item responses should be rescored so as the lowest item-level score is 0. Rescoring rules are provided in Table 13-4, Table 13-5, and Table 13-6.

Step 2: Calculation of the MG Symptoms PRO Scores

The scores are calculated using the formula below, i.e. the sum of item scores is linearly transformed to have all domain scores ranging from 0 to 100:

$$MG$$
 Symptom PRO scale score
$$= \frac{Sum \ of \ item \ scores \ within \ the \ scale}{Raw \ score \ range} \times \frac{Total \ number \ of \ items \ in \ the \ scale}{Number \ of \ non \ missing \ items \ in \ the \ scale} imes 100$$

The score for each scale is calculated only when at least 70% of the items are completed. Details on the minimum number of items needed for score calculation and the range of raw score are provided in Table 13-7.

Table 13-4: MG Symptoms: Ocular, Bulbar, and Respiratory Symptoms Rescoring



Table 13-4: MG Symptoms: Ocular, Bulbar, and Respiratory Symptoms Rescoring



Table 13-5: MG Symptoms: Physical Fatigue Rescoring





Table 13-6: MG Symptoms: Muscle Weakness Fatigability





Table 13-7: Description of the MG Symptoms PRO Scale Scores

| Scale | Number of Items | Number of items needed for score | Raw score range | Listing of items<br>included (MG<br>Symptoms PRO<br>item number) |
|---|---|---|---|---|
| Ocular symptoms | 5 | 4 | 0-15 | 1-5 |
| Bulbar symptoms | 10 | 7 | 0-30 | 6-15 |
| Respiratory symptoms | 3 | 3 | 0-9 | 16-18 |
| Physical fatigue | 15 | 11- | 0-60 | 19-33 |
| Muscle weakness fatigability | 9 | in sulfions | 0-36 | 34-42 |

## 13.5 MG Impairment Index

The MG-II is provided in Table 13-8. The MGII can be summarized as a total score and also as 2 sub-scores reflecting an Ocular and a Generalized domain.

The total score is the raw sum of all the items, including the clinical examination and the patient-reported questionnaire.

The ocular score is calculated by summing 8 items reflecting ocular impairments. These items are patient questionnaire items 1 to 6 and examination items 1 and 2.

The generalized score is calculated by adding items 7 to 22 from the patient questionnaire and items 3 to 6 from the examination.

In the event of missing data, the following rules will be applied:

- In the case where at least 7 of the 8 items from the Ocular subscale are answered, the Ocular subscale score will be generated after imputing the missing response by the average of non-missing responses, by adding all item scores. If there are 2 or more missing data out of the 8 Ocular subscale items, then the Ocular subscale score will be missing.
- In the case where at least 18 of the 20 items from the Generalized subscale are answered, the Generalized subscale score will be generated after imputing the missing response(s) by the average of non-missing responses, by adding all item scores. If there are 3 or more missing

#### MG Impairment Index (MGII)™ - Patient Questionnaire ID: Date: INSTRUCTIONS: Please answer the following questions regarding your symptoms. Only consider those that you think are related to myasthenia. Check the answer that best describes your symptoms over the past 2 weeks. PROBLEMS WITH YOUR EYES: Please answer regarding the past 2 weeks. 1. Double vision throughout the day Have you experienced episodes of Episodes only in No Double Episodes starting in Constant or present double vision? If yes, at what time Vision the evenings the afternoons most of the day do they occur (on average)? 2. Double vision with activities Have you experienced double vision No Double After less than hour, Constant double vision After more than with activities such as reading, driving, but not immediately Vision or it starts immediately watching TV or using a computer? If yes, how long does it take (on average) before the double vision occurs? 3. Severity of double vision Have you experienced double vision? Mild: it doesn't It affects my activities I need to cover lo Double If yes, how severe has it been (at affect my daily but no need to cover one eye to be able Vision your worst)? activities to function one eye 4. Eyelld drooping throghout the day Have you experienced drooping of No evelid Only in the Drooping starts in the Constant drooping or your eyelid(s)? If yes, when does it drooping present most of the day evenings afternoons occur (on average)? 5. Eyelid drooping with activities Have you experienced drooping of your No eyelid After more than After less than 1 hour, Constant drooping or it eyelid(s) with activities such as reading, drooping 1 hour but not immediately starts immediately driving, watching TV or using a computer? If yes, how long does it take (on average) before the drooping occurs? 6 Severity of eyelld drooping Have you experienced drooping of I need to lift my eyelid Mild: it doesn't It affects my vision No eyelid your eyelids? If yes, how severe has it or tilt my head to be affect my vision but no need to lift my drooping been (at your worst)? eyelid able to see

MGII. V1.0. English- Canada

## MG Impairment Index (MGII)™ - Patient Questionnaire

| | | | | ID: | |
|---|---|---|---|---|---|
| PROBLEMS EATING: Please an | swer regar | ding the past 2 | weeks. | | |
| 7. Difficulty swallowing | | | | | , NO' |
| orialisting. | allowing of o | casional episodes<br>choking/coughing<br>th food or liquids | Liquids return<br>through my nose,<br>but no problems<br>with solid food | Difficulty<br>swallowing hard<br>food, requiring a<br>change in diet | Unable to<br>swallow or<br>using a feeding<br>tube |
| 8. Chewing different types of food | 0 | 1 | 2 | | |
| Have you experienced difficulty chewing? How severe has it been (at your worst)? 9. Chewing tiredness/fatigue | No difficulty chewing | Difficulty chewin<br>hard foods (e.g<br>steak, raw carrot | . foods (e.g. ha | ving soft Unable<br>rd boiled only li | to chew (eating quids or feeding tube) |
| At your worst, how long does it take to develop fatigue or tiredness in your jaw? | No difficulty chewing | Difficulty chewin at the end of the meal | | g of the only li | e to chew (eating<br>quids or feeding<br>tube) |
| PROBLEMS SPEAKING AND BI | REATHING: | Please answer | regarding the | past 2 weeks. | |
| 10. Voice changes through the day | 7 | , KOL | | | |
| Have you experienced episodes of nasal, hoarse or weak voice? When do they occur on average? | No voice<br>changes | Voice changes of in the evenings | | the chan | onstant voice<br>ages or present<br>ost of the day |
| How long can you talk (ou average), before developing voice changes, such as nasal, hourse or weak voice? (Normal conversation, with pauses for other speakers) | No voice changes | Voice changes<br>after more than 3<br>minutes | • | minutes, or they | nt voice changes<br>start immediately<br>than 1 minute) |
| 12. Severity of voice changes | | | | | |
| At your worst, how severe have<br>your voice changes been? (Nasal,<br>hoarse, weak voice) | No voice changes | Mild changes: m<br>voice is mostly<br>clear | | ard to it is | rere changes:<br>impossible to<br>derstand me |

MGII. V1.0. English- Canada

## MG Impairment Index (MGII)™ - Patient Questionnaire

PROBLEMS SPEAKING AND BREATHING (Cont.): Please answer regarding the past 2 weeks. 13. Speech clarity through the day Have you experienced difficulty Constant slurring, or Slurred speech Slurred speech No episodes of pronouncing words or slurred starting in the present most only in the slurred speech speech? When does it occur on of the day evenings afternoons average? 14. Speech clarity with prolonged conversation How long can you talk (on Slurred speech Slurred speech after Constant slurring, or No episodes of average), before developing less than 30 minutes, it starts immediately after 30 minutes slurred speech slurred speech? (Normal but not immediately (less than 1 minute) conversation, with pauses for other speakers) 15. Severity of speech changes Mild slurring: At your worst, how severe have Moderate slurring: There Severe slurring: No episodes of your speech changes been? (Slur-It is easy to are some difficulties it is impossible to slurred speed understand me understanding me understand me ring, difficulty pronouncing words) 16. Difficulty breathing Have you experienced shortness With moderate No shortness of With minimal of breath that is caused by At rest or when Requiring effort (e.g. walking effort (e.g. getting breath (except myasthenia? (i.e. not caused lying on my assisted several blocks at my dressed, walking for strenuous by asthma, or other lung/heart ventilation back inside the house) own pace) disease) If yes, when has it occurred (at your worst)? GENERALIZED SYMPTOMS: Please answer regarding the past 2 weeks. 17. Overall physical tiredness Have you experienced overall Overall physical Overall physical Constant physical physical tiredness caused by No physical tiredness in the tiredness starting in tiredness, or present myasthenia gravis? (i.e. not by tiredness the afternoons most of the day evenings sleeplessness, depression or other medical conditions)


MGII, V1.0, English- Canada

Table 13-8: MG Impairment Index

# MG Impairment Index (MGII)™ - Patient Questionnaire

| GENERALIZED SYMPTOMS: Ple | ase answer | regarding the pa | ast 2 weeks. | "100) |
|---|---|---|---|---|
| 18. Arm weakness severity | | | | olli, c |
| Have you experienced weakness in your arms? If yes, how severe has it been (at your worst)? | No arm<br>weakness | Mild weakness<br>(e.g. difficulty<br>lifting heavy<br>objects) | Moderate weakness<br>(e.g. difficulty lifting arms<br>above the shoulders, but<br>I can do it) | Severe weakness (unable to lift arms above the shoulders) |
| 19. Arm weakness with prolonged | use | 1 | 200 | 102, |
| Have you experienced weakness in your arms after prolonged use? When does it happen (on average)? | No arm<br>weakness | Weakness when<br>keeping arms up for<br>long (e.g. washing<br>or drying my hair) | Weakness with prolonged<br>activities at shoulder level<br>(organizing objects on a<br>shelf, holding a phone to<br>the ear) | Weakness with<br>minimal effort (e.g.<br>desk work, chopping<br>vegetables) |
| 20. Leg weakness severity | | C POL | 5 1 | 3 |
| Have you experienced weakness in your legs? If yes, how severe has it been (at your worst)? | No leg<br>weakness | Mild weakness [e.g.<br>difficulty standing<br>from a squat or from<br>tying my shoes) | (e.g difficulty standing | Severe weakness<br>(e.g unable to stand<br>from a chair without<br>assistance) |
| 21. Leg weakness with prolonged | use O | | 2 | 3 |
| Have you experienced weakness in your legs after prolonged use? When does it happen (on average)? | No leg<br>weakness | Weakness when<br>walking more than<br>10 blocks at my own<br>pace | Weakness when walking less than 10 blocks at my own pace | Constant weakness or with minimal effort (standing, walking inside the house) |
| 22. Neck weakness | 0 | 1 | 2 | 3 |
| Have you experienced weakness<br>in your neck? When does it happen<br>(on average)? | No neck<br>weakness | Weakness only in the evenings | Weakness starting in the afternoons | Constant weakness or present most of the day |

MGII. V1.0. English- Canada

## MG Impairment Index (MGII) - Examination

| ID: |
|-------|
| Date: |

| manual. You will nee | | nation. Detailed instr | | | |
|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3(0) | Score |
| E1. Diplopia | No Diplopia | Diplopia in only 1 direction. | Diplopia in 2 directions. | Diplopia irl ≥3 ditections OR in primary gaze. | 0 |
| E2. Ptosis | No ptosis | Ptosis between 10-60 seconds. | Spontaneous<br>ptosis or in less than<br>10 seconds. | ijaii | |
| E3. Lower Facial<br>Strength | Normal strength | Can resist with cheeks, but air escapes through lips. | Unable to seal lips<br>or provide resis-<br>tance with cheeks. | | |
| E4. Arm Endurance | Holds arms for 180 seconds. | Holds arms for 91<br>179 seconds | Holds arms for 30-<br>90 seconds. | Holds arms for < 30 seconds. | |
| E5. Leg Enduranoe | Holds leg for 90 seconds. | Holds leg for 40-89 seconds. | Holds leg for 16-39 seconds. | Holds leg for ≤ 15 seconds. | |
| E6. Neok Endurance | Holds head for 60 seconds. | Holds head for 35-59 seconds. | Holds head for 11-<br>34 seconds. | Holds head for ≤ 10 seconds. | |


The MG-QOL15r is a brief survey, completed by the study participant, that is designed to assess some aspects of "quality of life" related to MG. The total score is calculated by summing all 15 individual items.

In the event of missing data, the following rules will be applied:

- are missing, the total score are missing are In the case where at least 70% of the items (i.e. 11 items out of the 15) are answered, the total score will be generated after imputing the missing responses by the average of available (ie
  - In the case where more than 30% (i.e. 5 items or more) are missing, the total score will not be

### Table 13-9: MG-QOL15r

Please indicate how true each statement has been (over the past few weeks).

- 1. I am frustrated by my MG
- I have trouble using my eyes because of my MG (e.g. double vision)
- 3. I have trouble eating because of MG
- 4. I have limited my social activity because of my MG
- My MG limits my ability to enjoy hobbies and fun activities
- I have trouble meeting the needs of my family because of my MG
- 7. I have to make plans around my MG
- 8. I am bothered by limitations in performing my work (include work at home) because of my MG
- 9. I have difficulty speaking due to MG
- 10. I have lost some personal independence because of my MG (e.g driving, shopping, running errands)
- 11. I am depressed about my MG
- 12. I have trouble walking due to MG
- 13. I have trouble getting around public places because of my MG
- 14. I feel overwhelmed by my MG
- 15. I have trouble performing my personal grooming needs due to MG

| | Not at all | Somewhat | Very much |
|---|------------|----------|-----------|
| | 0 | 1 | 2 |
| | | | 2 |
| | | | illo) |
| ì | | ail | Very much |
| | 1 | 100 | 10/13 |
| | 07 | 17 18 | |
| | D. OK | 7.0 | |
| 1 | JIPO'S | 0, | |
| | SiOli | | |
| | 3/1 | | |

MG-QOL15r Muscle and Nerve 2016 Dec;54(6):1015-1022.

Total MG-QOL15r score

MG-QOL15r - United States/English. MG-QOL15r\_AU1.0\_eng-USorf.doc

## 13.7 Markedly abnormal criteria for Rozanolixizumab program

The following criteria will be applied in the determination of marked abnormalities for laboratory assessment values. They are based on Version 5 of the Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or higher criteria unless otherwise noted. If both high and low criteria are shown for a parameter, the criteria should be summarized separately in tabular or graphical data summaries.

Table 13-10: Hematology

| Parameter | Unit | Unit | Marked Abnormality |
|---|---|---|---|
| | (conventional) | (standard) | Criteria |
| Hemoglobin | g/dL | g/L | <8.0 g/d L ;<80 g/L |
| WBC (Leukocytes) <sup>1</sup> | $10^{9}/L$ | $10^{9}/L$ | Low: $< 2.0 \times 10^9 / L$ |
| | | | High: $>30 \times 10^9/L$ |
| Lymphocytes | $10^{9}/L$ | $10^{9}/L$ | Low: $< 0.5 \times 10^9 / L$ |
| Absolute | | | High: $> 20 \times 10^9 / L$ |
| Neutrophils Absolute | $10^{9}/L$ | $10^{9}/L$ | $<1.0 \times 10^9/L$ |
| Platelets <sup>2</sup> | $10^{9}/L$ | $10^{9}/L$ | $<50.0 \times 10^9/L$ |

<sup>&</sup>lt;sup>1</sup>WBC (Leukocytes) markedly abnormal high criterion is not based on Version 5 CTCAE Grade 3 or higher criteria. Due to the mechanism of action of RLZ, the safety alert is related to infection risk which would be identified by a lower cut-point than the standard which is related to acute leukemias. A markedly abnormal high cut-point >30 x 10<sup>9</sup>/L is applied to flag leukocytosis (George 2012).

Table 13-9: Chemistry

| | - () | 7 0 (1) | |
|---|---|---|---|
| Parameter | Unit | Unit | Marked Abnormality Criteria |
| | (conventional) | (standard) | |
| AST (SGOT) | U/L | U/L | >5.0 x ULN |
| ALT (SGPT) | U/L | U/L | >5.0 x ULN |
| ALP (Alkaline | U/L | U/L | >5.0 x ULN |
| Phosphatase) | 20 20 | | |
| GGT (Gamma | U/L | U/L | >5.0 x ULN |
| Glutamyl | 0. | | |
| Transferase) | ķίO' | | |
| Bilirubin (Total) | mg/dL | umol/L | >3.0 x ULN if Baseline value is normal; |
| 111 | ) | | >3.0 x Baseline value if Baseline is |
| <i>cn</i> , 26. | | | abnormal |
| Albumin | g/dL | g/L | <2 g/dL; <20 g/L |
| Creatinine | mg/dL | umol/L | >3.0 x ULN |
| Estimate | mL/min/1.73 | mL/min/1.73 | eGFR <29 mL/min/1.73 m <sup>2</sup> |
| glomerular | $m^2$ | $m^2$ | |
| filtrate rate | | | |
| (eGFR) <sup>1</sup> | | | |
| C reactive | mg/L | mg/L | >10 mg/dL; >100mg/L |
| protein (CRP) <sup>2</sup> | | | |

| Calcium <sup>3</sup> | mg/dL | mmol/L | Low: Corrected serum calcium of <7.0 |
|---|---|---|---|
| | | | mg/dL; <1.75 mmol/L |
| | | | High: Corrected serum calcium of >12.5 |
| | | | mg/dL; >3.1 mmol/L |
| Immunoglobulin | (g/L) | (g/L) | ≤1 g/L |
| $G^4$ | | | × |
| Potassium | mmol/L | mmol/L | Low: <2.5 mmol/L |
| | | | High: >6.0 mmol/L |
| Sodium | mmol/L | mmol/L | Low: <125 mmol/L |
| | | | High: >155 mmol/L |
| Glucose <sup>5</sup> | mg/dL | mmol/L | Low: <40 mg/dL; <2.2 mmol/L |
| | _ | | High: > 250 mg/dL; >13.9 mmol/L |
| Total | mg/dL | mmol/L | >400 /dl; >10.34 mmol/L |
| Cholesterol | | | 16 110 |
| Triglycerides | mg/dL | mmol/L | >500 mg/dl; >5.7 mmol/L |

Abbreviations: ALT= alanine aminotransferase; AST = aspartate aminotransferase; dL = deciliter; GGT: gamma-glutamyltransferase; L = liter; mg = milligram; mmol = millimoles; μg = microgram; U = unit; ULN = upper limit of normal

Note: Marked abnormality criteria are defined by Grade 3 or higher events according to the Common Terminology for Adverse Events (CTCAE), Version 5.0, November 17, 2017 unless otherwise noted.

<sup>1</sup>eGFR is calculated using the Chronic Kidney Disease Epidemiology Collaboration or CKD-EPI formula (https://qxmd.com/calculate/calculator\_251/egfr-using-ckd-epi) which is eGFR = 141 \* min(Scr/κ,1)<sup>α</sup> \* max(Scr/κ, 1)<sup>-1.209</sup> \* 0.993<sup>Age</sup> \* 1.018 [if female] \* 1.159 [if black]; where Scr is serum creatinine (mg/dL), κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1. For derivation from values in standard units (umol/L) the κ values are 61.88 for females and 79.56 for males.

Table 13-10: Vital Signs

| Parameter | Abnormality Criteria |
|---|---|
| Pulse Rate (beats/minute) | ≤50 and a decrease from Baseline of ≥15 |
| 100 ico | ≥120 and an increase from Baseline of ≥15 |
| Systolic Blood Pressure (mmHg) | ≤ 90 and a decrease from Baseline of ≥20 |
| 700 3/1 | $\geq$ 180 and an increase from Baseline of $\geq$ 20 |
| Diastolic Blood Pressure (mmHg) | ≤50 and a decrease from Baseline of ≥15 |
| , , | ≥105 and an increase from Baseline of ≥15 |
| Temperature | >101 °F (38.3 °C) |
| Body Weight | ≥ 10% decrease from Baseline |
| | ≥ 10% increase from Baseline |

<sup>&</sup>lt;sup>2</sup>Includes CRP and High Sensitivity (HS) CRP. Reference for marked abnormality criteria: Nehring, S.M.; Goyal, A.; Patel, B.C. (2020). StatPearls Publishing, web link: <a href="https://www.ncbi.nlm.nih.gov/books/NBK441843/">https://www.ncbi.nlm.nih.gov/books/NBK441843/</a>. <sup>3</sup>Corrected Calcium (mmol/L) =0.02 \* (40 – Albumin (g/L)) + Calcium (mmol/L).

<sup>&</sup>lt;sup>4</sup>Immunoglobulin G criterion based on immunodeficiency literature and noted in RLZ study protocols.

<sup>&</sup>lt;sup>5</sup>Glucose high criterion defined by Grade 3 and higher events according to CTCAE, Version 4.03, June 14, 2010.

## Table 13-11: Electrocardiogram

| Parameter | Abnormality Criteria |
|-------------------|---------------------------------|
| QT interval (ms) | ≥500ms |
| | ≥60ms increase from Baseline |
| QTc(F) (ms) | ≥500ms |
| | ≥60ms increase from Baseline |
| PR interval (ms) | Treatment-emergent value >200ms |
| QRS interval (ms) | Treatment-emergent value >100ms |
| Heart rate (bpm) | <50bpm |
| | >120bpm |

Abbreviations: bpm = beats per minute; ms = milliseconds; QTc(F) = Fridericia corrected QT interval;

Note: Treatment-emergent is defined as meeting the criteria at any post-Baseline visit after the first infusion of study medication and within 56-days of the last infusion and not meeting the same criteria during Baseline

## 13.8 AEs of focus for Rozanolixizumab program

The AEOF selection criteria is specified in the Rozimab Safety AEs of Focus document developed by UCB. The purpose of this document is to detail the approach to identifying TEAEs meeting criteria for AEOF for the Rozanolixizumab (also called Rozimab) program.

## Following Events are AEOFs for Rozimab for MG studies:

| No | Event (also included in | Selection criteria |
|---|---|---|
| 110 | | Selection triteria |
| | Title of TFL output) | 0 10 |
| 1 | Headache | TEAE with HLGT='Headaches' |
| | (Note: also included in | |
| | AESM if severe) | |
| 2 | Gastrointestinal disturbances | TEAE with |
| | (Note: also included in | HLT='Gastrointestinal and abdominal pains (excl oral and |
| | AESM if severe) | throat)' or |
| | 50.00 | HLT='Gastrointestinal signs and symptoms NEC' or |
| | | HLT='Nausea and vomiting symptoms' or |
| | 8 | HLT='Diarrhoea (excl infective)' or |
| | ill die | HLT='Gastritis (excl infective)' |
| 3 | Hypersensitivity reactions | SMQ='Hypersensitivity' |
| 20 | | |
| 4 | Anaphylactic reactions | SMQ='Anaphylactic reaction' and |
| | | TEAEs that either emerged on the <b>same day</b> as when a study |
| | | medication injection reaction was received, or that emerged <b>one</b> |
| | | day after a study medication injection was received, and which |
| | | fulfill <u>any</u> of the following 3 criteria should be included in the |
| | | summary table: |
| | | - |

| | | 1. If a subject reports any TEAE which codes to a PT included in Category A, then the event will be flagged as an anaphylactic reaction. |
|---|---|---|
| | | 2. If a subject reports any TEAE which codes to a PT included in Category B <b>AND</b> reports any TEAE which codes to a PT included in Category C, <b>and both TEAEs have the same start date</b> , then both events will be flagged as anaphylactic reactions. |
| | | 3. If a subject reports any TEAE which codes to a PT included in Category D <b>AND</b> reports (either a TEAE which codes to a PT included in Category B <b>OR</b> a TEAE which codes to a PT included in Category C), <b>and both TEAEs have the same start date</b> , then both events will be flagged as anaphylactic reactions. |
| 5 | Injection site reactions | TEAE with HLT='Injection site reactions' or HLT='Infusion site reactions' or HLT='Administration site reactions NEC' |
| 6 | Infusion Reactions | Infusion reaction marked on AE CRF page (based on the assessment by the Investigator) |
| 7 | Opportunistic infections (Note: also included in AESM) | <ul> <li>Opportunistic infections (including tuberculosis) will be summarized in a stand-alone table using UCB-defined search criteria. Opportunistic infections are identified in two steps using the attached spreadsheet for MedDRA v24.0 in UCB Rozimab Safety AEs of focus document.</li> <li>Step 1: Refer to column B of the spreadsheet which identifies the Preferred Terms (PTs) to be classified as opportunistic infections using either a single 'x' or a double 'xx'.</li> <li>TEAEs which code to a PT flagged with a single 'x' need to also be serious in order to be considered an opportunistic infection.</li> <li>All TEAEs which code to a PT flagged with a double 'xx' are considered to be an opportunistic infection, regardless of seriousness.</li> <li>All serious TEAEs in the study database which code to a PT flagged with a single 'x' and all TEAEs in the study database which code to a PT flagged with a double 'xx' will be</li> </ul> |
| | | summarized as an opportunistic infection in the stand-alone table. [CQ97NAM= 'Opportunistic Infection— Automatic'] Step 2: Refer to column C of the spreadsheet which identifies the PTs that need to be evaluated on a case-by-case basis by the |

study physician and safety physician in order to determine whether it is a true opportunistic infection or not. The process for physician review is as follows:

- 1. Study programming team creates a spreadsheet which lists all of the subjects with a TEAE present in the database which codes to a PT identified as case-by-case. [CQ98NAM= Opportunistic Infection— Manual Review Candidate] Information from the AE dataset to be included in the spreadsheet: Subject ID, AE verbatim term, System Organ Class (SOC), High Level Term (HLT), Lower Level Term (LLT), PT, AE start date, AE end date, seriousness, severity, relationship to study medication, action taken. Additionally, a column will be included where the study physician/safety physician can document their decision on the case.
- 2. Study physician/safety physician (SPs) reviews the cases in the spreadsheet separately and reconciles final decision, and indicates in the additional column which AEs are confirmed to be opportunistic infections via a single 'x'.
- Study programming team incorporates these decisions into the AE dataset by merging the SPs decisions for individual subjects / PTs and flagging both the automatic and the confirmed opportunistic infections as such in the dataset. [CO99NAM= 'Opportunistic Infection – Adjudicated']

The SPs reviews the context of all of a subject's data (AEs and possibly other) and concludes individually.

Indicators of relevant cases may be e.g. repetitive occurrences, conjunction of other events or findings considered relevant. All subjects with a case-by-case PT reported that has been confirmed by the SPs to be an OI will be summarized as such in the stand-alone table, along with all of the events identified in Step 1 of this process.

[CQ99NAM= 'Opportunistic Infection – Adjudicated'] The timing and frequency of Step 2 should be outlined and agreed to by the study team at the beginning of the study. It is suggested that this process be executed multiple times throughout the course of the study, more frequently in the weeks leading up to database lock, and one final time immediately prior to database lock.

Following the initial physician review of case-by-case events, subsequent reviews will be based on the cumulative set of case-

#### AMENDMENT(S) TO THE STATISTICAL ANALYSIS PLAN 14

#### 14.1 **Amendment 1**

### Rationale for the amendment

- Modifications introduced in Protocol Amendment 3,
- COVID-19 strategy on the analyses,
- Specific analyses requests for PMDA,
- Additional analyses requested by sponsor
- Other cosmetics changes.

## **Modifications and changes**

| 14.1 Amendmen | t 1 | |
|---|---|---|
| Rationale for the amendmen | nt | |
| Rationale for the amendment This amendment is to apply following changes: Modifications introduced in Protocol Amendment 3, COVID-19 strategy on the analyses, Specific analyses requests for PMDA, Additional analyses requested by sponsor Other cosmetics changes. Modifications and changes Section # and Name Description of Change Brief Rationale | | |
| Modifications introduced in Protocol Amendment 3, | | |
| COVID-19 strategy on the analyses, | | |
| Specific analyses requests for PMDA, | | |
| Additional analyses requested by sponsor | | |
| • Other cosmetics changes. | | KING CLO |
| Modifications and changes | | To the |
| Section # and Name | Description of Change | Brief Rationale |
| Global | Minor administrative, formatting, and typographical changes have been made. | Updated to provide clarity and be consistent with remainder of SAP. |
| Global | Re-organized the paragraphs in some sections and added some clarifications. | For better understand and avoid misunderstanding of the analyses. |
| Global | "study drug" has been changed to "IMP" | Keep consistent terminology |
| Global | Updated abbreviations | Ensure abbreviations are used in the appropriate way. |
| 1. Introduction | Protocol Amendment 2 has been replaced with Protocol Amendment 3 | Protocol Amendment 3 has been approved. |
| 2.1.3 Other objectives | The objective relating to anti-drug antibody (ADA) was updated to include the impact it has on pharmacokinetics (PK) and pharmacodynamics (PD). | Updated in Protocol<br>Amendment 3 |
| 2.1.3 Other objectives | Evaluation of the effects of rozanolixizumab on serum cytokines was added to the study objectives. | Updated in Protocol<br>Amendment 3 |
| 2.1.3 Other objectives | Evaluation of the effects of rozanolixizumab on the $\alpha$ - and $\beta$ - globulins was removed from the study objectives. | Removed from Protocol<br>Amendment 3 |
| 2.1.3 Other objectives | Assessment of the effect of rozanolixizumab on deoxyribonucleic acid (DNA) and ribonucleic acid | Removed from Protocol<br>Amendment 3 |

| | (RNA) was removed from the study objectives and associated endpoints | |
|---|---|---|
| 2.1.3 Other objectives | Genetics was removed from the study objective. | Removed from Protocol<br>Amendment 3 |
| 2.1.3 Other objectives | The objective for exploratory biomarkers was made more general. | Updated in Protocol<br>Amendment 3 |
| 2.2.1.3 Efficacy endpoints | Other efficacy endpoints related to MG Impairment Index (MGII) scores have been moved to the end of the list. | Updated in Protocol<br>Amendment 3 |
| 2.2.1.3 Efficacy endpoints | An additional other efficacy endpoint has been added: "Minimal Symptom Expression (MG-ADL score of 0 or 1) at Day 43 (Visit 10)" | Updated in Protocol<br>Amendment 3 |
| 2.2.2.2 Pharmacodynamic endpoints | The pharmacodynamic endpoint for neurofilament-light (NF-L) levels has been removed. | Removed from Protocol<br>Amendment 3 |
| 2.2.4 Anti-drug antibody endpoints | New section was created for ADA endpoints | Separated from immunology endpoints |
| 2.2.5 Immunological endpoints | 'Observation Period' was removed from the endpoint relating to serum cytokines. | Updated in Protocol<br>Amendment 3 |
| 2.2.6 Other and exploratory endpoints | Genetics was removed from the study endpoint. | Removed from Protocol<br>Amendment 3 |
| 2.2.6 Other and exploratory endpoints | The endpoints for exploratory biomarkers was made more general. | Updated in Protocol<br>Amendment 3 |
| 2.3 Study design and conduct | The number of sites has been changed from 125 to 135. In addition, Asia has been added as a region for the study to be performed. | Updated in Protocol<br>Amendment 3 |
| 2.3 Study design and conduct | All reference to the rollover OLE study, MG0004, has been replaced to introduce the new OLE study, MG0007. | Updated in Protocol<br>Amendment 3 |
| 2.4 Determination of sample Size | Specify the calculation of second stage sample size | Clarifications on the sample size calculation |
| Figure 1-1 | The study schematic was updated with new figure. | Updated in Protocol<br>Amendment 3 |
| 3.2.1 Analysis time points | Added "Mapping to analysis visit windows is not applied, except for premature end of treatment (PEOT) visits (specified in Section 3.2.3)" | Clarified the mapping rule at PEOT visit |
| 3.2.2 Study periods | In Treatment Period definition, "ends after Day 43 assessment" has been | Clarified the end point of Treatment Period |

| | changed to "ends after Day 43/PEOT assessments." | |
|---|---|---|
| 3.2.2 Study periods | Clarified both Treatment and Observation periods are completed when study participants have a completed status in the Study Termination CRF | Ensured to be consistent with CRF guideline. |
| 3.5 Analysis sets | Remove "Analysis of the Safety Set (SS) will be according to the treatment the study participants actually received. Analysis of the Full Analysis Set (FAS) and Randomized Set (RS) will be according to the treatment to which the study participants were randomized." And explain the randomized or actual treatment used in section 3.5.2. and 3.5.3 Clarified that FAS is based on RS. | Simplified the sections. |
| 3.6 Treatment assignment and treatment groups | Added PK/PD analyses in the case study participants will be analyzed per actual treatment group | PK/PD analyses are also based on actual treatment group. |
| 3.8 Coding dictionaries | Updated MedDRA version to 23.0 | Latest coding version will be used in the study. |
| 3.9 Changes to protocoldefined analyses | Removed some changes that have been already incorporated into Protocol Amendment 3 and added interaction term used in the model of primary analysis. | Consistent with Protocol<br>Amendment 3 |
| 4.1 Adjustments for covariates | Specified the region category—North<br>America, Europe, and Asia [excluding<br>Japan], Japan | Clarification |
| 4.1 Adjustments for covariates | Clarified randomized stratification factor will be adjusted in the analysis model | Actual baseline stratification<br>factor could be different<br>from randomized one if it<br>has been entered by error in<br>IRWS at randomization |
| 4.2.1 Efficacy data | Added MGII scores and MG-QOL15r in this section regarding the rules for handling missing data | Missing in last version |
| 4.2.1 Efficacy data | Added a table to clarify the imputation methods for primary and secondary efficacy endpoints. | Further clarification |
| 4.2.2 Dates and times | Clarified the reasons for imputation of missing dates and times | Further clarification |

| 4.2.2 Dates and times | Added imputation rule for complete missing end date | Used for the calculation of AE duration |
|---|---|---|
| 4.2.2 Dates and times | Updated the rules in Table 4-1 | Further clarification |
| 4.2.3 Missing data due to COVID-19 | Added the new section for the approaches and strategies used to handle missing data due to COVID-19 | To address the impact of COVID-19 on the study data |
| 4.4.1 Timing of and basis for periodic data reviews and interim analysis | Updated the description of periodic data reviews and re-organize the section | Updated in Protocol<br>Amendment 3 |
| 4.4.1 Timing of and basis for periodic data reviews and interim analysis | Clarified the futility stopping rule is non-blinding and correct p-value at each dose to 0.025 | Clarification and mistake correction |
| 4.4.2 Data required for periodic data reviews and interim analyses | Updated the section and sub-sections title. | Further clarification |
| 4.6 Multiple comparisons/multiplicity | Updated the step number proceeded to in Scenario 1 | Incorrect step numbers in last version |
| 4.6 Multiple comparisons/multiplicity | In Scenario 2 Step 5, clarified that "Both doses are significant if the larger 2-sided p-value lesser than 0.5(1+1)*0.05=0.05. If not, then one dose is significant if the smaller p-value less than 0.025." | Truncation fraction is 1 for family 6. |
| 4.9 Examination of subgroups | Clarified randomized stratification factor will be used in the subgroup analyses | Actual baseline stratification<br>factor could be different<br>from randomized one if it<br>has been entered by error in<br>IRWS at randomization |
| 4.9 Examination of subgroups | Added additional subgroups for MG-ADL and subgroup only derived in analysis datasets | Additional subgroups were requested for PMDA submission |
| 4.9.1 Examination of COVID-19 Subgroups | New section was added to specify additional summary on COVID-19 subgroups, pre-, during and post- the COVID-19 pandemic | To analyze the amount of data pre-, during and post-the COVID-19 pandemic. |
| 5.1 Participant disposition | Added additional summaries of screen failure and disposition by pre-, during and post- the COVID-19 pandemic | To analyze the amount of data pre-, during and post-the COVID-19 pandemic. |
| 5.2 Protocol deviations | Added PD relationship to COVID-19 in summary table and additional summaries by pre-, during and post-the COVID-19 pandemic | To analyze the amount of data pre-, during and post-the COVID-19 pandemic. |

| 6.1 Demographics | Added "Notes: Missing age will be calculated as year of informed consent signed – year of birth" | Handling of missing age. |
|---|---|---|
| 6.1 Demographics | Added "A by-participant listing of demographics will be provided using the RS. Childbearing potential and lifestyle will be listed using the ES separately." | Missing in last version |
| 6.1 Demographics | Added additional summaries by pre-, during and post- the COVID-19 pandemic | To analyze the amount of data pre-, during and post-the COVID-19 pandemic. |
| 6.2 Other Baseline characteristics | Specified where to locate those baseline characteristics | Further clarification |
| 6.2 Other Baseline characteristics | Added "Thymectomy (yes, no)", "MG-specific autoantibody (MuSK+ /aChR+)" and Baseline MG-ADL category | Additional Baseline characteristics were requested for PMDA submission |
| 6.2 Other Baseline characteristics | Added age at initial MG diagnosis | Missing in last version |
| 6.2 Other Baseline characteristics | Added additional summaries by pre-, during and post- the COVID-19 pandemic | To analyze the amount of data pre-, during and post-the COVID-19 pandemic. |
| 6.3 Medical history and concomitant diseases | Added additional summaries by pre-,<br>during and post- the COVID-19<br>pandemic | To analyze the amount of data pre-, during and post-the COVID-19 pandemic. |
| 6.4.1 Categories of prior and concomitant medications | Updated the definition in 5 categories and added table to clarify it | Further clarification |
| 6.4.2 Assignment of medications to study period | Clarified the assignment of mediation to Treatment and Observation Period | Further clarification |
| 8.1 Handling of intercurrent events | New section was added to specify the intercurrent events and 2 new intercurrent events related to COVID-19. Listed the strategies for the intercurrent events. | Further clarification |
| 8.2 Statistical analysis of the primary efficacy endpoint | Added the paragraph to briefly describe the analyses for primary endpoint and list the estimand attributes in Table 8-1 and 8-2 | Estimand attributes of primary endpoint were not clear in last version. |
| 8.2.2 Primary analysis of the primary efficacy endpoint | Updated sequential test formula and descriptions | Incorrect in last version |
| 8.2.3.2 Sensitivity Analysis #2 | New sensitivity analysis using jump-<br>to-reference approach is added | Updated in Protocol<br>Amendment 3 |

| 8.2.4.1 Supplementary<br>Analysis #1 | The analysis using trimmed mean approach is downgraded to supplementary analysis. Methodology updated. | Updated in Protocol<br>Amendment 3 |
|---|---|---|
| 8.2.5 Additional analysis | Additional analysis was added using study participant not affected by COVID-19 | To check the COVID-19 impact on primary endpoint |
| 8.3.1 MG-ADL Responder<br>Rate at Visit 10 (Day 43) | Added "Any missing data scores (including missing data due to the intercurrent events) due to other reasons will also be imputed as non-responders." | Further clarifications on how to handle missing MG-ADL responder |
| 8.4 Analysis of other efficacy endpoints | Clarified summary of other efficacy endpoints will be performed overall, except for time to MG-ADL response. | Further clarification |
| 8.4.1 Use of rescue therapy due to worsening (IVIg, PEX) | Specified the alpha level to be used in the statistical test | Missing in last version |
| 8.4.2 Time to first rescue therapy | Updated the censoring rule and added summary of study participants with 8, 12, 24, 32, 43, 57, 71, 85, 99 days to first rescue therapy and number of censored study participants | Missing in last version |
| 8.4.3 Time to MG-ADL response ( $\geq$ 2.0 points improvement from Baseline) | Updated the censoring rule and added summary of study participants with 8, 12, 24, 32, 43 days to first rescue therapy and number of censored study participants. | Missing in last version |
| 8.4.3 Time to MG-ADL response (≥2.0 points improvement from Baseline) | Clarified the censoring rule and the KM plot by treatment group and cumulative ADA/NAb positivity | Further clarification |
| 8.4.4 QMG score | Added "The subgroup summaries will also be performed as specified in Section 4.9." and "By-participant listings of QMG scores will be provided." | Missing in last version |
| 8.4.5 QMG responder rate (≥3.0 points improvement from Baseline) | Added "In addition, QMG responders will be summarized by the subgroup (MuSK+ or aChR+)." | Additional subgroups were requested for PMDA submission |
| 8.4.5 QMG responder rate (≥3.0 points improvement from Baseline) | Specified both observed and imputed responders will be summarized. | Further clarification |
| 8.4.6 MG-C score | Added "The subgroup summaries will also be performed as specified in Section 4.9." and "By-participant | Missing in last version |

| | listings of QMG scores will be provided." | |
|---|---|---|
| 8.4.7 MG-C responder rate (≥5.0 points improvement from Baseline) | Added "In addition, MG-C responders will be summarized by the subgroup (MuSK+ or aChR+)." | Additional subgroups were requested for PMDA submission |
| 8.4.7 MG-C responder rate (≥5.0 points improvement from Baseline) | Specified both observed and imputed responders will be summarized. | Further clarification |
| 8.4.8 MG-ADL score | Added "The subgroup summaries will also be performed as specified in Section 4.9." | Missing in last version |
| 8.4.8 MG-ADL score | Added "Additionally, a table will summarize missing MG-ADL assessment at each scheduled visit by treatment group." | Assess the COVID-19 impact on the efficacy data |
| 8.4.8 MG-ADL score | Clarified the KM plot by treatment group and cumulative ADA/NAb positivity | Clarification of the plot |
| 8.4.9 MG-ADL responder rate (≥2.0 points improvement from Baseline) | Added "In addition, MG-ADL responders will be summarized by the subgroup (MuSK+ or aChR+)." | Additional subgroups were requested for PMDA submission |
| 8.4.9 MG-ADL responder rate (≥2.0 points improvement from Baseline) | Specified both observed and imputed responders will be summarized. | Further clarification |
| 8.4.10 MG Symptoms PRO 'Physical Fatigue' score | Added "The subgroup summaries will also be performed as specified in Section 4.9." and "By-participant listings of all MG Symptoms PRO values will be provided." | Missing in last version |
| 8.4.11 MG Symptoms PRO 'Muscle Weakness Fatigability' | Added "The subgroup summaries will also be performed as specified in Section 4.9." | Missing in last version |
| 8.4.12 MG Symptoms PRO 'Bulbar Symptoms' | Added "The subgroup summaries will also be performed as specified in Section 4.9." | Missing in last version |
| 8.4.13 MG Symptoms PRO 'Respiratory Symptoms' score | Removed description of the score | Details of PRO items can be found in the protocol. |
| 8.4.14 MG Symptoms PRO 'Ocular Symptoms' score | Removed description of the score | Details of PRO items can be found in the protocol. |
| 8.4.15 Patient Global<br>Impressions of Severity | Removed description of the score | Details of PRO items can be found in the protocol. |
| 8.4.15 Patient Global<br>Impressions of Severity | Added "A by-participant listing of PGI-S will be provided." | Missing in last version |
|---|---|---|
| 8.4.16 Patient Global<br>Impressions of Change | Removed description of the score | Details of PRO items can be found in the protocol. |
| 8.4.16 Patient Global<br>Impressions of Change | Added "A by-participant listing of PGI-C will be provided." | Missing in last version |
| 8.4.17 MGII overall scores, ocular sub-scores, and generalized domain scores | Removed description of the score | Details of PRO items can be found in the protocol. |
| 8.4.17 MGII overall scores, ocular sub-scores, and generalized domain scores | Added "A by-participant listing of MGII scores will be provided. | Missing in last version |
| 8.4.18 MG-QOL15r | Removed description of the score | Details of PRO items can be found in the protocol. |
| 8.4.18 MG-QOL15r | Added "A by-participant listing of MG-QOL15r scores will be provided." | Missing in last version |
| 8.4.20 Minimal symptom expression | New efficacy endpoint was added. | Added in Protocol<br>Amendment 3 |
| 9.2 Pharmacodynamics | Removed NF-L | Removed in Protocol<br>Amendment 3 |
| 9.2.1 MG-specific autoantibodies | Added additional plots and correlation tables. Added efficacy data in listings. | Requested by sponsor |
| 9.3 Anti-drug antibody | Created separate section for ADA | Separated it with immunology endpoints. |
| 9.3 Anti-drug antibody | Clarified the ADA analyses | Requested by sponsor |
| 9.4.2 Cytokines | Added summary for study participants experiencing with serious or severe headache and/or infusion reactions or hypersensitivity reaction. | Updated in in Protocol<br>Amendment 3 |
| 10.2.2 AE summaries | Updated the AE summaries. | Requested by sponsor |
| 11.1 Specific analyses for<br>Pharmaceuticals and Medical<br>Devices Agency (PMDA) | Listed specific analyses for PMDA | Specific analyses were requested for patients in Japan only |
| 13.6 MG-QOL15r | Added scoring details of MG-QOL15r | Missing in last version |
| 13.7 Markedly abnormal criteria for Rozanolixizumab program | Updated the criteria per new MA document provided by UCB | Document is updated by sponsor |
| 13.8 AEs of focus of Rozanolixizumab | Updated the criteria per new UCB<br>Rozimab Safety AEs of Focus<br>document | Document is updated by sponsor |

#### 14.2 **Amendment 2**

#### Rationale for the amendment

- Update and/or Clarification on various wording, definition and cutoff values.
- Update to be consistent across MG studies and follow Protocol Amendment 4 edits.
- Incorporate regulatory feedback on ICE handling.
- Additional analyses requested by sponsor.
- Other cosmetics changes.

## **Modifications and changes**

| Nationale for the a | menument | |
|---|---|---|
| • Update and/or • | Clarification on various wording, defin | ition and cutoff values. |
| • Update to be co | Update to be consistent across MG studies and follow Protocol Amendment 4 edits. | |
| • Incorporate regu | ulatory feedback on ICE handling. | :120 |
| • Additional analy | yses requested by sponsor. | |
| • Other cosmetics | changes. | |
| Modifications and | changes | |
| Section # and<br>Name | Description of Change | Protocol Amendment 4 edits. Brief Rationale |
| | Add "(excluding ocular items)" to<br>Change from Baseline in MG-ADL at<br>each scheduled assessment during<br>Treatment and Observation Period | Updated as it was an omission from the previous protocol amendment. |
| | Add "at any time up to and including" to Minimal symptom expression (MG-ADL score of 0 or 1) at Day 43 (Visit 10) | Updated as it was an omission from the previous protocol amendment. |
| 2.2.1.3 Other efficacy endpoints | Remove "and Observation" in Change from Baseline in MG Impairment Index (MGII) scores at each scheduled assessment during Treatment and Observation Periods. Remove "and Observation" in Change from Baseline in MGII ocular subscores at each scheduled assessment during Treatment and Observation Periods. Remove "and Observation" in Change from Baseline in MGII generalized domain sub-scores at each scheduled assessment during Treatment Periods. | These PRO will not be assessed during the Observation Period. |
| 3.3 Definition of Baseline values | Baseline definition to include using of IMP date, if time is missing, but assessment date is on same date as first IMP | Updated to provide Clarification on baseline values. |

| 3.9 Changes to protocol-defined analysis | Add "estimand and ICE strategies to be based on regulatory feedback". Update Potential Hy's Law to Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) >3x Upper Limit of Normal (ULN) and total Bilirubin (TBL) >2xULN, and Alkaline Phosphatase (ALP) <2 x ULN. The Full Analysis Set (FAS) will consist of all study participants in the RS. Update MG specific autoantibodies stratification factor from a single two category factor to two binary | Update as PD to RA4 |
|---|---|---|
| | factors, MuSK (+/-) and aChR (+/-). Minimal Symptom Expression (MG-ADL score of 0 or 1) at any time up to and include both treatment and observation phase, where the protocol only states to include up to Day43 (Visit10). | on Valiatile |
| 4.1Adjustment for covariates | Change MG-specific autoantibody stratification factor in statical modeling to be based on values evaluated at Baseline instead of IWRS at randomization. Add explanation on handling of missing MG-specific autoantibody stratification factors. | Updated to provide further clarification on source of the baseline MG-specific autoantibody values as stratification factor. |
| 4.4.2.2 Data required for interim analysis | Remove MG Symptoms PRO tables from IA list | Updated to meet IA meeting decision, not necessary for IA and for DMC. |
| 4.9 Examination of subgroups | Change MG-specific autoantibody stratification factor in the subgroup analysis to be based on values evaluated at Baseline instead of IWRS at randomization. | Updated to provide further clarification. On source of the baseline MG-specific autoantibody values as stratification factor. |

| | For Baseline Characteristics table, MG-ADL cut off value was set to be <5, >=5 | Updated to set cutoff value for clarification. |
|---|---|---|
| 5.1 Participant<br>Disposition | Add primary reason for participants roll over from MG3 to MG4/7. "Mandatory withdrawal due to need for rescue therapy and roll over to extension study" to be under "Other". | Add explanation for participants that has completed the treatment in MG0003 and then needs rescue treatment and instead roll over to the MG0004/7 extension studies. |
| 5.1,<br>6.1, 6.2, 6.3<br>8.1, 8.3.1, 8.4.1,<br>8.4.3-8.4.20<br>9.1, 9.2, 9.2.1,<br>9.2.2, 9.3.2,<br>9.4.1-9.4.4<br>10.1 | Add "RLZ total" as a group for all summaries and plots | General update |
| 6.2 Other Baseline characteristics | Change and separate "Baseline" and "historical" MG-specific autoantibodies summary, and add comparison. | Updated to provide further clarification on data source of "Historical" and "Baseline" MG-specific antibodies. |
| 6.2 Other Baseline characteristics | Change Age at initial MG diagnosis = (Date of Initial MG Diagnosis—Date of Birth+1)/365.25 | Updated to correct error in formula. |
| 8.1 Handling of intercurrent events | Change ICE2 treatment discontinuation to permanent treatment discontinuation. Combine previously hypothetical strategy with new edits to Target treatment strategy as Hypothetical & Treatment Strategy to handle ICEs, | Update based on regulatory suggestions. |
| 8.1 Handling of intercurrent events | Clarified that study participants with visits in treatment period affected by COVID-19 will be removed for COVID-19 free analysis. | To clarify when to remove study participant, as it doesn't make sense to remove the study participant if COVID only affected visit (s) during the observation period of the study participant. |
| 8.2 Statistical analysis of the primary efficacy endpoint | Change "Treatment condition of interest" to "Treatment Conditions". Change "Population of interest(targeted)" to "Population". | Update in accordance to ICH GCP estimand attributes. |

| 8.3 Statistical analysis of the secondary efficacy endpoint | | |
|---|---|---|
| 8.2 Statistical analysis of the primary efficacy endpoint 8.2.4.1 | Define "worst score" for imputation to be from its respected questionnaire. | Updated to provide further clarification. |
| Supplementary analysis #1 | | clarification. |
| 8.2.3.4 Sensitivity<br>Analysis #4 | Add an additional sensitivity analysis of the primary endpoint (on the FAS), excluding confirmed COVID-19 cases | Update based on regulatory suggestions. |
| 8.4 Analysis of other efficacy endpoints | Add analyses for COVID-19 free patients for QMG and MG-C as well. | To check the impact of COVID-19. |
| 9.3 Anti-drug antibody status | ADA related modification | Updated to be consistent across the Phase 3 rozanolixizumab clinical program. |
| | Added AESM definition. | For better understanding and reminder to check the data. |
| 10.2.2 AE summaries | Added TEAEs leading to death by relationship | Required for final CSR. |
| | Define risk difference of > 5% to be displayed. | Further clarity on % risk difference for display. |
| 10.3 Clinical laboratory evaluations | Remove "If multiple central lab data were captured at scheduled visits, the average would be used for continuous values, or the worst will be used for categorical values" | Updated to be consistent across the Phase 3 rozanolixizumab clinical program. |
| 10.21.20 | Remove HDL, total cholesterol, and<br>Triglycerides from Clinical Chemistry | |
| 10.3.1 Potential drug-induced liver injury | Update criteria for pDILI | Updated to be consistent across the Phase 3 rozanolixizumab clinical program. |
| 11.1 Specific<br>analysis for<br>Pharmaceuticals<br>and Medical | Remove MG Symptoms PRO related secondary efficacy endpoints Remove Time to first rescue, EQ-5D-5L from other efficacy | Update to align with Japanese table review. |
| Devices Agency | endpoints | |

| | | Remove AESM, AEOFs, lab, vital signs and ECG from safety endpoints. | |
|---|---|---|---|
| | 11.2 Headache<br>Questionnaire | Change each study participant to each applicable study participant using ES | Update to provide further clarification |
| | 13.1 QMG Scale | Update table 13-1 with new scale values based on updates in QMG CRF. | Updated to be consistent across the Phase 3 rozanolixizumab clinical program. |
| | 13.8 AEs of focus | Update to include MedDRA 23.1 | Update to current version of MedDRA |
| Kils | 90ch sibbilit | Update table 13-1 with new scale values based on updates in QMG CRF. Update to include MedDRA 23.1 | any marketing the street of th |


### 14.3 Amendment 3

#### **Rationale for the amendment**

- Update PK/PD related sections
- Update to be consistent across MG studies and follow Protocol Amendment 4 edits.
- Update to add additional exploratory analysis and figures for display
- Clarification on various definitions.

# **Modifications and changes**

| Section # and Name | <b>Description of Change</b> | Brief Rationale |
|---|---|---|
| Throughout | Update to MedDRA v24.0 | General update |
| | MG-C responder rate from ≥ 5 points improvement from Baseline to ≥ 3 points | General update |
| | Correction to typos and abbreviations. | cialio. |
| 2.2.1.3 Other efficacy endpoints | Patient Global Impressions of<br>Severity (PGI-S) at each<br>scheduled assessment during the<br>Treatment and Observation | Correction. |
| | Periods instead of change from Baseline of PGI-S. | |
| 3.3 Definition of Baseline | Add "and time if time is collected for the individual assessment)" Add "MG-specific autoantibodies MuSK and aChR Baseline is detailed in Section 9.2.1" | Clarification and to be consistent with all MG studies. |
| 3.5.4 Pharmacokinetic Per-<br>Protocol Set | Change to "at least 1 dose of rozanolixizumab, had at least 1 quanifiable concentration"; Add "Post-Baseline deviations will not necessarily lead to total exclusion of a study participant from the PK-PPS but may lead to exclusion of specific data." | Clarification |
| 3.7 Center Pooling Strategy | Add region categorization. | Clarification |

| 3.8 Coding Dictionaries | Update version and date. | General update and to be consistent with all MG studies. |
|---|---|---|
| 3.9 Changes to protocol-defined analysis | MG-C responder definition will<br>be 3-point improvement instead<br>of 5-point.<br>PGI-S instead of change from<br>Baseline of PGI-S | Update as PD to PA4 |
| | LDL calculation | |
| 4.1 Adjustments for covariate | Add "a post-Baseline measurement may be used. If this is not available, then" | Clarification O |
| 4.2.1 Efficacy data | Apply NRI imputation to include timepoints after use of rescue medication. | Clarification |
| 4.2.2 Dates and Time | Remove duplication in calculation rules in Table 4-1 | Correction to typo |
| 4.9.1 General subgroups | Add "using the same algorithm for missing values as specified in Section 4.1". Add "Historical MuSK (+/non +) and historical AChR (+/non +) will also be examined in the subgroup analysis, in this case, Baseline MuSK(+/-) and Baseline AChR(+/-) will replaced by Historical MuSK (+/non +) and historical AChR(+/non +). " | Clarification |
| 4.9.1 General subgroups | Add "Forest plot will be provided"; Remove MG Baseline medication definition and add to section 6.4.3 | General summary |
| 5.1 Participant Disposition | Add summary table to show count of participant by visit. | General summary |

| 6.1 Demographic | Add "The same summary will also be presented by stages". | General summary |
|---|---|---|
| 6.2 Other Baseline characteristics | Add reference to 6.4.3 | Clarification |
| Characteristics | Add "The same summary will also be presented by stages". | .10 |
| | Add "Procedure History CRF" to Thymectomy | Clarification |
| 6.3 Medical History and<br>Concomitant Diseases | Add "history of headache" | Clarification |
| 6.4.3 Baseline MG medication definition | Add new section to define MG Baseline medication definition. | Clarification |
| 8.2.6 Exploratory Analysis | Repeat section 8.2.2 using historical MG-specific autoantibodies status. | Add exploratory analysis |
| 8.3.2 -8.3.6 | Add "Exploratory: The same approach as Section 8.2.6 will be applied" | Add exploratory analysis |
| 8.4.3 Time to MG-ADL | Update for clarification. | Clarification |
| Response | Remove KP plot by "overall ADA or neutralizing antibody (NAb) status" | Remove plots to be consistent with PK section. |
| 9 PHARMACOKINETICS | Ò | |
| AND<br>PHARMACODYNAMICS | Add "all other analysis will be performed on Safety Set" | Clarification |
| 9.1 Pharmacokinetics | Remove paragraph on plots for ADA titer and ADA status | Remove duplication |
| 90cs 361 | Explain spaghetti plot to be plotted "by treatment group" and "administered RLZ dose | |
| | total" | Clarification |

| | Remove geometric mean plot by cumulative ADA status | Remove plots |
|---|---|---|
| | Replace arithmetic mean plot by geometric time course plot | Remove plots |
| | Adding guidelines on data to be presented "If more than 1/3 of the individual data points at a timepoint are missing or are not quantifiable, then only n, minimum, median and maximum will be presented. The other descriptive statistics will be left blank. • If n<3, then only the n, minimum and maximum will be presented. If no study participants have data at a given timepoint, then only n=0 will be presented." | Clarification |
| | Add "Change from baseline" for IgG and IgG subclass, and remove "MG-ADL change from Baseline" from graph. | Further Clarification |
| 9.2.1 MG-specific autoantibodies | Add MG-specific autoantibodies<br>Baseline definition | Further clarification |
| 9.2.1 MG-specific autoantibodies | Adding reference | General update |
| 9.2.1 MG-specific autoantibodies | Add "The maximum decrease from Baseline in MG-specific autoantibodies (change absolute and percentage change decrease) will be reported in the listing and summarized for each treatment." For MG-specific auto antibodies summaries. | Clarification |
| | Add "and the plot will be repeated for the following dose groups: placebo, | Clarification |

| | *** | |
|---|---|---|
| | Add "Mean percent change from baseline of anti-MuSK and Total IgG, and mean change from baseline of MG-ADL, QMG, MG-C will be plotted over time by treatment and RLZ total for only participants who are anti-MuSK positive at baseline" | Add plots Change plot style |
| | Change time course plots to "boxplot of maximum percent change" for MG-Specific autoantibodies | Change plot style |
| 9.2.2 Total serum IgG and IgG subclasses | Replace "decrease" and "absolute change "as "change and percent change " | Clarification |
| | Clarify "mean change" instead<br>of "mean" plot will be plotted,<br>also add dose group plots to IgG<br>mean change and percentage<br>graph | Clarification |
| ~e | Remove "absolute", add "Total" to IgG | Clarification |
| 90chusus calious al | Remove "Individual plots per study participant will be plotted representing total IgG, MG-specific autoantibodies, NAb titer, MG-ADL total score. See details in Section 9.3.2." and "A plot of geometric mean of total IgG (absolute) and arithmetic mean of percentage change from Baseline by cumulative ADA status will be presented by treatment group and RLZ total. See details in Section 9.3.2." | Remove plots |

| | - | |
|---|---|---|
| | Change "Absolute reduction" to "Change"; "to" day 43 to "at" day 43; "relative reduction " to "Percent change" | Clarification |
| | Remove "up to day 43 and time plot of mean change and percent change " | Remove plots and Clarification |
| | Add "change from baseline concentration of total IgG and IgG subclass" to listing | General update |
| | Add "Samples that are NAb positive will be evaluated in a titration assay to quantify the NAb level and will be reported as titer. Samples from study participants on placebo will not | Remove plots and Clarification General update |
| 9.3 Anti-drug antibody status | be tested for anti-drug antibodies." | Clarification |
| 9.3.1 ADA Data Consideration | add "if corresponding rozanolixizumab concentrations are equal or below the validated drug tolerance limit of the ADA assay (200µg/mL rozanolixizumab) allowing detection of 100ng/mL ADA" to ADA negative definition; Add definition of ADA inconclusive "Sample values that are either 'negative screen' or the combination of 'positive screen' and 'negative immune-depletion', but with corresponding rozanolixizumab concentrations above the validated drug tolerance limit of the ADA assay, will be defined as ADA inconclusive " | Update ADA sample status definition |
| | change "ADA Classification"<br>to "ADA/NAb participant<br>Status" | Update ADA sample status definition |

| | Update Table 9-1 for participant ADA/NAb classification | Update ADA sample status definition |
|---|---|---|
| | Remove Cumulative ADA status and Overall ADA status | Update ADA sample status definition |
| 9.3.2 ADA Summaries | Update tables, figures and listings based on new definition of ADA participant category. Also add scatter plots, and remove geometrics mean plots | Clarification Remove plots |
| | Remove Time to MG-ADL KP plots by ADA/NAb status | Remove plots |
| 10.2.3 AE of Focus | Add Treatment-emergent to<br>all tables; Add AEOF table by<br>Risk Difference ≥5% (by<br>decreasing frequency of Risk<br>Difference) | Clarification |
| 10.3 Clinical laboratory evaluations | Replace "Change from<br>Baseline" with "Mean" value for<br>plotting. Update Table 10-1. | Clarification and update per PA4 |
| | Add plots for lipids if data available. | Clarification |
| 12 Reference | Add reference for "The MG<br>Composite" by Burns, Ted M et<br>al. | Add reference |
| 13.7 Markedly abnormal criteria for Rozanolixizumab program | Added corrected calcium algorithm and updated the marked abnormality criteria for corrected calcium and eGFR formula parameters. | Clarification to align with literature values |
| 13.8 AEs of focus | Updated definitions of AEOF | To be consistent across MG studies |

acal an of the an of the an of the any make tind authorization of the any make tind authorization and any extensions of ratialitions thereof.

This document cannot be used any extensions of ratialitions and any extensions of ratialitions and any extensions of ratialitions and any extensions of ratialitions and any extensions of the contract of the

